# **Clinical Study Protocol**

# A Phase III Randomised, Double-blind, Multicentre Study to Compare the Efficacy, Safety, Pharmacokinetics, and Immunogenicity between SB12 (proposed eculizumab biosimilar) and Soliris® in Subjects with Paroxysmal Nocturnal Haemoglobinuria

| Product | SB12 (proposed eculizumab biosimilar) |
|----------------|---------------------------------------|
| FudwaCT Number | 2019 002957 21 |

EudraCT Number 2018-002857-31
US pre-IND Number PIND 135254
Protocol Number SB12-3003
Study Phase Phase III

**Version and Effective Date** Version 6.0 Nov 27, 2020

Version 5.0 Aug 21, 2020 Version 4.0 Nov 29, 2019

Version 3.0 Dec 12, 2018

Oct 08, 2018

Version 1.0 Jul 31, 2018

**Sponsor** Samsung Bioepis Co., Ltd.

107, Cheomdan-daero, Yeonsu-gu,

Incheon, 21987 Republic of Korea

Version 2.0

This document contains confidential information belonging to Samsung Bioepis Co., Ltd. Your acceptance or review of this document constitutes agreement that you will not copy or disclose the information contained herein to others or use it for unauthorised purposes without written authorisation from the Sponsor.

# **SYNOPSIS**

| Name of Sponsor/Company: | Samsung Bioepis Co., Ltd. |
|----------------------------|---------------------------------------|
| Name of Finished Product: | SB12 (proposed eculizumab biosimilar) |
| Name of Active Ingredient: | Eculizumab |

**Title of Study:** A Phase III Randomised, Double-blind, Multicentre Study to Compare the Efficacy, Safety, Pharmacokinetics, and Immunogenicity between SB12 (proposed eculizumab biosimilar) and Soliris<sup>®</sup> in Subjects with Paroxysmal Nocturnal Haemoglobinuria

Protocol No: SB12-3003 Phase: III

**Planned Study Period:** After Screening, the duration of study participation will be 58 weeks per subject including 50 weeks of treatment and 8 weeks of post-treatment follow-up. After completion of study treatment, subjects may be entered into an extended supply of up to 2 years.

#### **Objectives:**

#### Primary objective

The primary objective of this study is to demonstrate comparable clinical efficacy of SB12 and Soliris<sup>®</sup>, by evaluating the lactate dehydrogenase (LDH) in subjects with paroxysmal nocturnal haemoglobinuria (PNH).

#### Secondary objectives

The secondary objectives are:

- To evaluate the efficacy of SB12 compared to Soliris® by
  - LDH profile over time
  - Number of units of packed red blood cells (pRBCs) transfused
- To evaluate the safety and tolerability of SB12 compared to Soliris®
- To evaluate the pharmacokinetic (PK) of SB12 compared to Soliris®
- To evaluate the immunogenicity of SB12 compared to Soliris®
- To evaluate the pharmacodynamic (PD) of SB12 compared to Soliris®

# **Study Design:**

This is a randomised, Phase III, double-blind, multicentre, cross-over study to compare the efficacy, safety, pharmacokinetics, and immunogenicity between SB12 and Soliris® in subjects with PNH.

Subjects will be randomised in a 1:1 ratio to treatment sequence I (SB12 to Soliris®) or treatment sequence II (Soliris® to SB12). Subjects who are randomised to initially receive SB12 will be switched to receive Soliris® and subjects who are randomised to initially receive Soliris® will be switched to receive SB12 at Week 26.

In special circumstances of a shortage of the comparator, to ensure continuity of study treatment for the duration of study, the Sponsor will provide SB12 instead of Soliris<sup>®</sup> in a blinded manner.

After completion of activities at Week 52, an open-label extended supply of SB12 will be provided for up to 2 calendar years to subjects who have benefited from study treatment and opt to participate in extended supply under an ethical basis.

#### **Number of Subjects:**

A total of approximately 50 subjects (25 subjects per treatment sequence) will be randomised in this study.

| Name of Sponsor/Compar | y: Samsung Bioepis Co. | Samsung Bioepis Co., Ltd. |
|---|---|---|
| Name of Finished Product | SB12 (proposed eculi | SB12 (proposed eculizumab biosimilar) |
| Name of Active Ingredient | t: Eculizumab | |
| Treatment Sequence | Period 1 | Period 2 |
| I (n = 25) | SB12 | Soliris <sup>®</sup> |
| II (n = 25) | Soliris <sup>®</sup> | SB12 |

# Target Population:

Eculizumab-naïve patients with PNH

#### **Eligibility Criteria:**

#### Inclusion criteria

Subjects must meet all of the following criteria to be eligible for the study:

- 1. Male or female aged 18 or older at the time of signing the informed consent form (ICF), if local regulations are different in this regard, follow the local regulations.
- 2. Documented diagnosis of PNH.
- 3. Presence of the PNH white blood cell (WBC) clone, with a granulocyte or monocyte clone size of ≥ 10% by high-sensitivity flow cytometry at Screening.
- 4. Documented LDH level  $\geq 1.5 \times$  upper limit of normal (ULN) at Screening.
- 5. History of transfusion for anaemia within 12 months prior to Screening or having PNH-related symptoms (e.g., fatigue, haemoglobinuria, abdominal pain, chest pain, shortness of breath [dyspnoea], dysphagia, erectile dysfunction) at Screening.
- 6. All subjects must be vaccinated against *Neisseria meningitidis* within 3 years prior to or on Day 1 in accordance with current local guidelines or Soliris® Summary of Product Characteristics (SmPC) to reduce the risk of meningococcal infection.
- 7. Female subjects who are not pregnant or nursing at Screening and on initiation of study drug (Day 1) and who are not planning to become pregnant from Screening until 5 months after the last dose of study drug.
- 8. Subjects and their partners of childbearing potential (female or male) who agree to use of a highly effective contraceptive method (e.g., established use of oral, injected or implanted hormonal contraceptive, placement of an intrauterine device or intrauterine system, male sterilisation, or true abstinence [see Section 8.4.1]) from Screening until 5 months after the last dose of study drug.
- 9. Subjects must be able to understand the implications of taking part in the study and be willing to follow the study instructions and requirements fully.
- 10. Subjects must be able to provide informed consent, which must be obtained prior to any study related procedures.

#### Exclusion criteria

Subjects meeting any of the following criteria are not eligible for the study:

1. Previous treatment with a complement pathway inhibitor (including eculizumab).

| Name of Sponsor/Company: | Samsung Bioepis Co., Ltd. |
|----------------------------|---------------------------------------|
| Name of Finished Product: | SB12 (proposed eculizumab biosimilar) |
| Name of Active Ingredient: | Eculizumab |

- 2. Known hypersensitivity to the investigational product (IP) or any of the ingredients or excipients of the IP.
- 3. Known contraindication/hypersensitivity for meningococcal vaccine or the antibiotic to be used in the study.
- 4. Abnormal haematological parameters at Screening defined as the following:
  - a. Absolute neutrophil count (ANC)  $\leq 0.5 \times 10^3/\mu L$
  - b. Platelet count  $< 70 \times 10^3/\mu L$
- 5. History of meningococcal disease.
- 6. History of haematopoietic stem cell transplantation.
- 7. History of serious thrombotic event (e.g., stroke, myocardial infarction, pulmonary embolism, etc.).
- 8. Known or suspected active bacterial, virus, fungal infection within 30 days prior to initiation of study drug (Day 1).
- 9. Known history of human immunodeficiency virus (HIV) infection or have positive results at Screening.
- 10. Concomitant use of any of the following medications is prohibited if the following conditions apply.
  - a. Erythropoietin, systemic corticosteroids, low-molecular-weight heparins, iron supplements, and androgen therapy that have not been on a stable dose for at least 4 weeks prior to initiation of study drug (Day 1).
  - b. Warfarin with an unstable international normalised ratio (INR) for at least 4 weeks prior to initiation of study drug (Day 1) at the discretion of the Investigator.
  - c. Cyclosporine that has not been on a stable dose for at least 8 weeks prior to initiation of study drug (Day 1).
- 11. Subjects who have received or participated in another investigational drug, device, or procedures within 30 days or within 5 half-lives of that IP prior to Screening, whichever is greater.
- 12. History of malignancy within 5 years prior to Screening, except for curatively treated carcinoma in situ of uterine cervix, basal cell carcinoma of the skin, or squamous cell carcinoma of the skin.
- 13. Any other cardiac, hepatic, immunologic, pulmonary, rheumatoid disease, other conditions causing rise in LDH (e.g., tumours, muscular dystrophies, liver and bile disease, etc.), or the disorder which, at the discretion of the Investigator, will put the subjects at risk if they are enrolled.
- 14. Other unspecified reasons that, at the discretion of the Investigator or Sponsor, make the subjects unsuitable for enrolment.

# **Investigational Products:**

- Name: SB12 (proposed eculizumab biosimilar) or Soliris®
- Formulation: A vial of 30 mL contains 300 mg of eculizumab (10 mg/mL)
- Route of administration: Intravenous (IV) infusion  $35 \pm 10$  minutes

| Name of Sponsor/Company: | Samsung Bioepis Co., Ltd. |
|----------------------------|---------------------------------------|
| Name of Finished Product: | SB12 (proposed eculizumab biosimilar) |
| Name of Active Ingredient: | Eculizumab |

• Dose regimen: 600 mg every 7 days for the first 4 weeks (initial phase) and 900 mg for the fifth week, followed by 900 mg every  $14 \pm 2$  days until Week 50 (maintenance phase).

#### **Main Criteria for Evaluation**

#### **Primary endpoints**

- LDH level (U/L) at Week 26
- Time-adjusted area under the effect curve (AUEC) of LDH from Week 14 to Week 26 and from Week 40 to Week 52

#### **Secondary endpoints**

#### Efficacy endpoints

- LDH profile over time
- Number of units of pRBCs transfused throughout the study period

#### Safety endpoints

- Incidence of adverse events (AEs)
- Incidence of serious AEs (SAEs)
- Incidence of infection-related AEs
  - Meningococcal infection
  - Other systemic infections
- Incidence of infusion-related reactions (IRRs)

Safety of subjects will be monitored by 12-lead electrocardiogram (ECG), vital sign assessment, and physical examination. Haematological, biochemical, and urinalysis laboratory parameters will be also measured.

#### PK endpoint

• Concentration prior to infusion (trough serum concentration [C<sub>trough</sub>]) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, and 52

#### Immunogenicity endpoints

- Incidence of anti-drug antibodies (ADAs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and early termination (ET) visit
- Incidence of neutralising antibodies (NAbs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and ET visit

# PD endpoint

Terminal complement activity at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 26, 28, 30, 32, 36, 40, and 52

#### **Statistical Methods**

# Analysis sets for efficacy analyses

Modified Full Analysis Set (M-FAS) consists of all randomised subjects who do not have positive result of pharmacogenetic analysis (C5 gene polymorphism). However, subjects who do not have any efficacy assessment result after randomisation and do not receive IP during the study period will be excluded from this analysis set. Following the intent-to-treat principle, subjects will be analysed according to the treatment sequence they are assigned to at randomisation.

Per-Protocol Set for AUEC of LDH (PPS-AUEC) consists of all M-FAS subjects who have sufficient LDH assessments for AUEC calculation without any major protocol deviations (PDs) that have impact on efficacy assessment. Subjects excluded from the primary analysis will be pre-defined on a case-by-case basis prior to unblinding the treatment sequence assignment for analyses. In addition, subjects who received different treatment from the randomised treatment sequence due to a shortage of the comparator will be excluded from this analysis set.

Per-Protocol Set for LDH at a single time point (PPS-single) consists of all M-FAS subjects who have LDH assessment at Week 26 without any major PDs that have impact on efficacy assessment. Subjects excluded from the primary analysis will be pre-defined on a case-by-case basis prior to unblinding the treatment sequence assignment for analyses. In addition, subjects who received different treatment in Period 1 from the randomised treatment sequence due to a shortage of the comparator will be excluded from this analysis set.

#### Efficacy analyses

for those who are in favour of the time-adjusted AUEC of LDH, the primary efficacy analysis will be performed for the PPS-AUEC using a linear mixed model with treatment, sequence, period, and gender as fixed effects, and subject nested within sequence as a random effect. The analysis will be performed with loge-transformed time-adjusted AUEC of LDH estimating the difference in least squares means and its 90% confidence interval (CI), and back transformation of those values will provide the ratio of geometric means and 90% CI. The equivalence will be declared if the two-sided 90% CI of the ratio of geometric means in time-adjusted AUEC of LDH between SB12 and Soliris® lies within the pre-defined equivalence margin of [0.77, 1.29].

for those who are in favour of the LDH level at a single time point, the primary efficacy analysis will be performed for the PPS-single using a linear mixed model with treatment, and gender as a fixed effect. The analysis will be performed with log<sub>e</sub>-transformed LDH at Week 26 estimating the difference in least squares means and its 95% CI, and the delta method will be used to provide the mean difference and 95% CI in original scale. The equivalence will be declared if the two-sided 95% CI of the mean difference in LDH level at Week 26 between SB12 and Soliris<sup>®</sup> lies within the pre-defined equivalence margin of [-1.2 × ULN, 1.2 × ULN] where ULN of LDH to be specified in the central laboratory specification for this study. If normal range of LDH is gender specific, the smaller/smallest ULN will be used for the equivalence margin; otherwise ULN is not gender specific, unified ULN will be used for the equivalence margin.

For sensitivity analysis, the primary efficacy analysis will be repeated for the M-FAS. Missing data will be imputed using multiple imputation method for subjects who drop out for the study prior to the primary analysis time point. Complete case analysis will also be performed.

As a secondary efficacy endpoint, the number of units of pRBCs transfused will be summarised descriptively by treatment sequence and treatment sequence within period and will be analysed using Wilcoxon rank-sum test. And mean LDH profile will be presented over time.

#### Safety analyses

Safety analyses will be performed in the Safety Set (SAF).

| Name of Sponsor/Company: | Samsung Bioepis Co., Ltd. |
|----------------------------|---------------------------------------|
| Name of Finished Product: | SB12 (proposed eculizumab biosimilar) |
| Name of Active Ingredient: | Eculizumab |

All reported terms for AEs will be coded using Medical Dictionary for Regulatory Activities (MedDRA®). AEs will be collected and classified according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0.

All AE data will be summarised by count and percentage of subjects experiencing events by system organ class, preferred term. TEAEs leading to IP discontinuation and treatment-emergent AEs (TEAEs) by causality and severity will be summarised similarly. Infection-related AEs including meningococcal infection and other systemic infection, and IRRs will also be summarised.

Changes in vital signs and clinical laboratory parameters will be summarised descriptively by treatment sequence and visit. Other safety variables will be summarised unless otherwise specified.

Additional analyses will be performed for the subjects who received different treatment from the randomised treatment sequence due to a shortage of the comparator if needed. For example, AEs and concomitant medications will be analysed based on the actual switched treatment.

#### PK analyses

PK analysis will be performed for the PK Analysis Set (PKS). C<sub>trough</sub> will be summarised descriptively by treatment sequence and visit.

## Immunogenicity analyses

The immunogenicity analyses will be performed for the SAF. ADA and NAb results will be summarised with count and percentage by treatment sequence and visit. The incidence of overall ADA will be summarised by treatment sequence and period.

#### PD analyses

PD analysis will be performed for the PD Analysis Set (PDS). The absolute value and change from baseline in terminal complement activities will be summarised by treatment sequence and visit.

#### Sample size

The equivalence margin for the mean difference of LDH at Week 26 is derived from two historical studies with Soliris<sup>®</sup>. In TRIUMPH study, the mean (standard deviation [SD]) of LDH at Week 26 is 327.3 (432.9) U/L and 2,418.9 (930.6) U/L for eculizumab and non-eculizumab arms, respectively. PNH registry study reported the mean of LDH at 6 months is 352.1 (224.0) U/L and 1,201.0 (815.6) U/L for eculizumab and non-eculizumab arms, respectively.

A meta-analysis with fixed-effect model estimates –1,152.5 U/L of LDH mean at Week 26 with a 95% CI [–1,303.4, –1,001.7]. The of upper limit of 95% CI was approximately U/L, which implies that at least treatment effect is obtained to preserve the treatment effect over placebo if the U/L was statistically chosen as the equivalence limit.

In the clinical study, LDH detection level or normal range of LDH would depend on the specification of laboratory parameters chosen for the study. Therefore, it is not likely to be clinically meaningful to propose any specific LDH level as the equivalence margin without the consideration of normal range of LDH level.

| Name of Sponsor/Company: | Samsung Bioepis Co., Ltd. |
|----------------------------|---------------------------------------|
| Name of Finished Product: | SB12 (proposed eculizumab biosimilar) |
| Name of Active Ingredient: | Eculizumab |

Therefore, the equivalence margin will be  $[-1.2 \times \text{ULN}, 1.2 \times \text{ULN}]$  for the comparison with the 95% CI of the mean difference in LDH at Week 26 where ULN of LDH to be specified in the central laboratory specification for this study. For sample size calculation, [-268 U/L, 268 U/L] is chosen to be 23 subjects per treatment sequence with the assumptions of no mean difference and common SD of 270 U/L at the overall 5% significance level. Assuming a 5% loss from randomised subjects after 26 weeks, a sample size of 25 subjects per treatment sequence (overall sample size of 50) will give 23 completers per treatment sequence after 26 weeks, which is estimated to give 80% power to detect the equivalence within the margin of 268 U/L.

For calculation of the equivalence margin for time-adjusted AUEC of LDH, mean and coefficient of variation (%CV) were referred from TRIUMPH study. The mean (%CV) of AUEC of LDH at Week 26 is 81,140.0 U/L × day (142.45%) and 429,874.1 U/L × day (33.49%) for eculizumab and non-eculizumab arms, respectively.

From the results in the reference study, mean ratio of AUEC of LDH is estimated to be 0.19 with a 90% CI [0.1308, 0.2724]. The upper limit of the equivalence margin is calculated as where it preserves at least of eculizumab treatment effect over the placebo, but the equivalence margin will be [0.77, 1.29] for the comparison with the 90% CI of mean ratio of time-adjusted AUEC of LDH.

With the given equivalence margin of [0.77, 1.29], 22 subjects per treatment sequence was calculated with the assumptions of the mean ratio of 1, common %CV of 42% at the overall 10% significance level. Assuming a 10% loss from randomised subjects after 52 weeks, a sample size of 25 subjects per treatment sequence (overall sample size of 50) will give 22 completers per treatment sequence after 52 weeks, which is estimated to give 80% power to detect the equivalence within the margin of [0.77, 1.29].

Therefore, the sample size of 50 allows enough power to detect the equivalence in both situations.

# GRAPHICAL STUDY DESIGN AND SCHEDULE OF ACTIVITIES



#### Figure 1. Graphical Study Design

- ® = Randomisation; AUEC = Area under the Effect Curve; EOS = End of Study; n = No. of Subjects; PNH = Paroxysmal Nocturnal Haemoglobinuria; W = Week
- a. Randomisation will trigger the shipping of study drugs to investigational site. The initiation of study drug should be done within 21 days of randomisation.
- b. Week 0 (Day 1) is defined as the day of the initiation of study drug. During Week 0 (Day 1) to Week 3, 600 mg of SB12 or Soliris® every 7 ± 2 days
- c. From Week 4, 900 mg of SB12 or Soliris<sup>®</sup> every  $14 \pm 2$  days up to Week 50.
- d. Primary endpoints: 1) LDH level (U/L) at Week 26 and 2) AUEC of LDH from Week 14 to Week 26 and from Week 40 to Week 52
- e. Cross-over from SB12 to Soliris® and Soliris® to SB12 at Week 26
- f. After completion of activities at Week 52, an open-label extended supply of SB12 will be provided for up to 2 calendar years to subjects who have benefited from study treatment and opt to participate in extended supply under an ethical basis.
- g. EOS is defined as either completion of safety follow-up at Week 58 or completion of ET visit (8 weeks after the last dose of SB12 or Soliris®), which may be up to Week 56.
- h. During the treatment period, in special circumstances of a shortage of the comparator, to ensure continuity of study treatment for the duration of study, the Sponsor will provide SB12 instead of Soliris® in a blinded manner.

Table 1. Schedule of Activities (Period 1, before Cross-over)

| Assessments | Study Period | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Visit | Scree | Randomi | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 |
| Week | -ning | -sation | 0 | 1 | 2 | 3 | 4 | 6 | 8 | 10 | 12 | 14 | 16 | 18 | 20 | 22 | 24 |
| Day (± Visit Window) | -63 to<br>-22 | -21 to -1 | 1 | 8<br>(±2) | 15<br>(±2) | 22<br>(±2) | 29<br>(±2) | 43<br>(±2) | 57<br>(±2) | 71<br>(±2) | 85<br>(±2) | 99<br>(±2) | 113<br>(±2) | 127<br>(±2) | 141<br>(±2) | 155<br>(±2) | 169<br>(±2) |
| Obtain informed consent <sup>1</sup> | ✓ | | | | | | | | | | | | | | | | |
| Demographic information | ✓ | | | | | | | | | | | | | | | | |
| Medical, transfusion, and thrombosis history | ✓ | | | | | | | | | | | | | | | | |
| Vaccination for Neisseria meningitidis <sup>2</sup> | ✓ | ✓ | ✓ | | | | | | | | | | | | | | |
| Serology (HIV-1 and HIV-2) | ✓ | | | | | | | | | | | | | | | | |
| FSH <sup>3</sup> | ✓ | | | | | | | | | | | | | | | | |
| Randomisation <sup>4</sup> | | ✓ | | | | | | | | | | | | | | | |
| Pharmacogenetic sampling <sup>5</sup> | | | ✓ | | | | | | | | | | | | | | |
| 12-lead ECG <sup>6</sup> | ✓ | | | | | | | | | | | ✓ | | | | | |
| Pregnancy test <sup>7</sup> | ✓ | | ✓ | | | | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | | ✓ |
| PNH clone size <sup>8</sup> | ✓ | | ✓ | | | | | | | | | ✓ | | | | | |
| Coagulation profile <sup>9</sup> | ✓ | | ✓ | | | | | | | | | ✓ | | | | | |
| Ferritin, vitamin B <sub>12</sub> , folate | ✓ | | ✓ | | | | | | | | | ✓ | | | | | |
| LDH <sup>10</sup> | ✓ | | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |
| Haematology and chemistry tests <sup>11</sup> | ✓ | | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |
| Reticulocyte count, haptoglobin, free haemoglobin | ✓ | | ✓ | | ✓ | | ✓ | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | |
| Urinalysis | ✓ | | ✓ | | ✓ | | ✓ | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | |
| Blood sampling for PK analysis <sup>12</sup> | | | ✓ | | ✓ | | ✓ | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | |
| Blood sampling for PD analysis <sup>13</sup> | | | ✓ | | ✓ | | ✓ | ✓ | | ✓ | | ✓ | | | | | <u> </u> |
| Blood sampling for immunogenicity assay <sup>14</sup> | | | ✓ | | ✓ | | ✓ | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | |
| PNH symptomatology <sup>15</sup> | ✓ | | ✓ | | | | ✓ | | | | | ✓ | | | | | |
| Physical examination <sup>16</sup> | ✓ | | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |
| Vital sign <sup>17</sup> | ✓ | | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |
| IP administration <sup>18</sup> | | | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |
| Adverse events <sup>19</sup> | Continuously | | | | | | | | | | | | | | | | |
| Previous and concomitant medications <sup>20</sup> | | | | | | | | Contin | uously | | | | | | | | |
| Thrombosis record (MAVEs) | | | | | | | | Contin | uously | | | | | | | | |
| Transfusion record (date and number of pRBCs) <sup>21</sup> | | | | | | | | Contin | uously | | | | | | | | |

HIV = Human Immunodeficiency Virus; FSH = Follicle Stimulating Hormone; ECG = Electrocardiogram; PNH = Paroxysmal Nocturnal Haemoglobinuria; LDH = Lactate Dehydrogenase; PK = Pharmacokinetic; PD = Pharmacodynamic; IP = Investigational Product; MAVEs = Major Adverse Vascular Events; pRBCs = Packed Red Blood Cells

Samsung Bioepis -  Information

- 1. Informed consent should be obtained prior to any study related procedures.
- 2. Neisseria meningitidis vaccination should be conducted prior to or on Day 1 according to current local guidelines or Soliris® SmPC. In case subjects were vaccinated against meningococcal infection within 3 years prior to Day 1, which is properly documented, vaccination could be omitted. Subject who initiates study drug administration less than 14 days after receiving a meningococcal vaccine must receive treatment with appropriate prophylactic antibiotics (e.g., ciprofloxacin) until 14 days after vaccination.
- 3. FSH levels will be measured at Screening and Week 26 in order to confirm postmenopausal status only for women who present natural (spontaneous) amenorrhea for at least 12 months prior to Screening regardless of the subjects' age.
- 4. All screening procedures must be completed and reviewed within 42 days prior to randomisation. All eligibility criteria not dependent on Day 1 must be reviewed and confirmed prior to randomisation. The initiation of study drug (Day 1) should be done within 21 days of randomisation. Eligibility criteria that are dependent on Day 1 should be checked at Day 1 and if found in violation then should be withdrawn according to discontinuation criteria.
- 5. Blood sample for pharmacogenetic analysis (C5 gene polymorphism) will be taken at Day 1. If missing, it would be taken at the next scheduled blood sampling time.
- 6. Twelve-lead ECG will be collected at Screening and pre-dose on Week 14, Week 26, Week 40, and Week 52.
- 7. Females of childbearing potential only. Serum pregnancy test at Screening and 8 weeks after the last dose of study drug in case of early termination (ET); urine pregnancy test at other applicable visits before study drug administration.
- 8. Both white blood cell (WBC) and red blood cell (RBC) clone size will be measured by flow cytometry at Screening and prior to dosing at Day 1 and Week 52. At other visits (Week 14, Week 26, and Week 40), only RBC clone size will be measured prior to dosing.
- 9. Parameters included in coagulation profile are prothrombin time, partial thromboplastin time, and international normalised ratio (INR).
- 10. LDH will be measured at pre-dose on each visit and will also be measured if the suspected sign or symptom of breakthrough haemolysis occurs.
- 11. Parameters included in haematology test are WBC count, RBC count, haemoglobin, haematocrit, platelet count, differential WBC count, nucleated RBC, mean corpuscular haemoglobin (MCH), mean corpuscular haemoglobin concentration (MCHC), mean corpuscular volume (MCV), mean platelet volume (MPV), and red cell distribution width (RDW). Parameters included in chemistry tests are sodium, potassium, creatinine, blood urea nitrogen (BUN), glucose, calcium, phosphorus, total bilirubin, direct/indirect bilirubin, albumin, total protein, alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), and gamma-glutamyl transpeptidase. All these parameters will be measured at pre-dose on each visit.
- 12. Blood sample for PK analysis will be taken prior to dosing at Weeks 0, 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, and 52. Blood samples should be collected at the same day of study drug administration. If the administration of IPs is delayed for any reasons after pre-dose blood sampling for PK analysis, blood sample should be re-collected on actual dosing day and be used for analysis. PK samples will also be collected if the suspected sign or symptom of breakthrough haemolysis occurs.
- 13. Blood sample for PD (terminal complement activity) analysis will be taken prior to dosing at Weeks 0, 2, 4, 6, 10, 14, 26, 28, 30, 32, 36, 40, and 52. Blood samples should be collected at the same day of study drug administration. If the administration of IPs is delayed for any reasons after pre-dose blood sampling for PD analysis, blood sample should be re-collected on actual dosing day and be used for analysis. PD samples will also be collected if the suspected sign or symptom of breakthrough haemolysis occurs.
- 14. Blood sample for immunogenicity assay will be taken prior to dosing at Weeks 0, 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and ET visit. Blood samples should be collected at the same day of study drug administration. If the administration of IPs is delayed for any reasons after pre-dose blood sampling for immunogenicity assay, blood sample should be recollected on actual dosing day and be used for analysis.
- 15. Investigator and/or designee will assess the PNH-related symptoms including fatigue, haemoglobinuria (discolouration of urine), chest pain, abdominal pain, dyspnoea, dysphagia, and erectile dysfunction.
- 16. Physical examination including height and weight at Screening; physical examination including weight at subsequent visits. Physical examination will be conducted before study drug administration.
- 17. Measured in a sitting position after remaining in a sitting or supine position for at least 5 minutes, including blood pressure, heart rate, and body temperature. On dosing days, vital signs will be taken before study drug administration.
- 18. Intravenous (IV) infusion will be performed for  $35 \pm 10$  minutes.

- 19. Adverse events (AEs) will be collected from the time of signing the informed consent until end of study (EOS).
- 20. Previous medications (within 4 weeks prior to Screening except immunosuppressant, 8 weeks prior to Screening for immunosuppressant) will be recorded and concomitant medications will be recorded until EOS.
- 21. Transfusion record will be collected from the time of signing the informed consent until EOS.

Table 2. Schedule of Activities (Period 2 and Safety Follow-up/ET, after Cross-over)

| Assessments | | | | | | | | | Stu | dy Per | iod | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Visit | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 23 | 24 | 25 | 26 | 27 | 28 | 29 | Safety<br>Follow-up <sup>21</sup> | ET <sup>22</sup> |
| Week | 26 <sup>1</sup> | 28 | 30 | 32 | 34 | 36 | 38 | 40 | 42 | 44 | 46 | 48 | 50 | 52 <sup>20</sup> | 58 | 8 (±1) weeks |
| Day (± Visit Window) | 183<br>(±2) | 197<br>(±2) | 211<br>(±2) | 225<br>(±2) | 239<br>(±2) | 253<br>(±2) | 267<br>(±2) | 281<br>(±2) | 295<br>(±2) | 309<br>(±2) | 323<br>(±2) | 337<br>(±2) | 351<br>(±2) | 365<br>(±2) | 407 (±7) | after the last<br>dose of study<br>drug |
| FSH <sup>2</sup> | ✓ | | | | | | | | | | | | | | | |
| 12-lead ECG <sup>3</sup> | ✓ | | | | | | | ✓ | | | | | | ✓ | | |
| Pregnancy test <sup>4</sup> | ✓ | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | | ✓ |
| PNH clone size <sup>5</sup> | ✓ | | | | | | | ✓ | | | | | | ✓ | | |
| Coagulation profile <sup>6</sup> | ✓ | | | | | | | ✓ | | | | | | ✓ | | |
| Ferritin, vitamin B <sub>12</sub> , folate | ✓ | | | | | | | ✓ | | | | | | ✓ | | |
| LDH <sup>7</sup> | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | | ✓ |
| Haematology and chemistry tests <sup>8</sup> | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | | ✓ |
| Reticulocyte count, haptoglobin, free haemoglobin | ✓ | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | | ✓ |
| Urinalysis | ✓ | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | | ✓ |
| Blood sampling for PK analysis <sup>9</sup> | ✓ | ✓ | ✓ | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | | |
| Blood sampling for PD analysis <sup>10</sup> | ✓ | ✓ | ✓ | ✓ | | ✓ | | ✓ | | | | | | ✓ | | |
| Blood sampling for immunogenicity assay <sup>11</sup> | ✓ | ✓ | ✓ | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | | ✓ | | ✓ |
| PNH symptomatology <sup>12</sup> | ✓ | | ✓ | | | | | ✓ | | | | | | ✓ | | |
| Physical examination <sup>13</sup> | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | | ✓ |
| Vital sign <sup>14</sup> | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | | ✓ |
| IP administration <sup>15</sup> | <b>√</b> 16 | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | | | |
| Adverse events <sup>17</sup> | | | | | | | | | | ntinuou | | | | | | |
| Previous and concomitant medications <sup>18</sup> | | | | | | | | | Coı | ntinuou | sly | | | | | |
| Thrombosis record (MAVEs) | | | | | | | | | | ntinuou | | | | | | |
| Transfusion record (date and number of pRBCs) <sup>19</sup> | | | | | | | | | Coı | ntinuou | sly | | | | | |

ET = Early Termination; FSH = Follicle Stimulating Hormone; ECG = Electrocardiogram; PNH = Paroxysmal Nocturnal Haemoglobinuria; LDH = Lactate Dehydrogenase; PK = Pharmacokinetic; PD = Pharmacodynamic; IP = Investigational Product; MAVEs = Major Adverse Vascular Events; pRBCs = Packed Red Blood Cells

- 1. All subjects who roll over into Period 2 will be switched to receive the other IP (SB12 or Soliris®) on Week 26 after all assessments have been performed.
- 2. FSH levels will be measured at Screening and Week 26 in order to confirm postmenopausal status only for women who present natural (spontaneous) amenorrhea for at least 12 months prior to Screening regardless of the subjects' age.
- 3. Twelve-lead ECG will be collected at Screening and pre-dose on Week 14, Week 26, Week 40, and Week 52.

Samsung Bioepis -  Information

- 4. Females of childbearing potential only. Serum pregnancy test at Screening and 8 weeks after the last dose of study drug in case of ET; urine pregnancy test at other applicable visits before study drug administration.
- 5. Both WBC and RBC clone size will be measured by flow cytometry at Screening and prior to dosing at Day 1 and Week 52. At other visits (Week 14, Week 26, and Week 40), only RBC clone size will be measured prior to dosing.
- 6. Parameters included in coagulation profile are prothrombin time, partial thromboplastin time, and INR.
- 7. LDH will be measured at pre-dose on each visit and will also be measured if the suspected sign or symptom of breakthrough haemolysis occurs.
- 8. Parameters included in haematology test are WBC count, RBC count, haemoglobin, haematocrit, platelet count, differential WBC count, nucleated RBC, MCH, MCHC, MCV, MPV and RDW. Parameters included in chemistry tests are sodium, potassium, creatinine, BUN, glucose, calcium, phosphorus, total bilirubin, direct/indirect bilirubin, albumin, total protein, ALT, AST, ALP, and gamma-glutamyl transpeptidase. All these parameters will be measured at pre-dose on each visit.
- 9. Blood sample for PK analysis will be taken prior to dosing at Weeks 0, 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, and 52. Blood samples should be collected at the same day of study drug administration. If the administration of IPs is delayed for any reasons after pre-dose blood sampling for PK analysis, blood sample should be re-collected on actual dosing day and be used for analysis. PK samples will also be collected if the suspected sign or symptom of breakthrough haemolysis occurs.
- 10. Blood sample for PD (terminal complement activity) analysis will be taken prior to dosing at Weeks 0, 2, 4, 6, 10, 14, 26, 28, 30, 32, 36, 40, and 52. Blood samples should be collected at the same day of study drug administration. If the administration of IPs is delayed for any reasons after pre-dose blood sampling for PD analysis, blood sample should be re-collected on actual dosing day and be used for analysis. PD samples will also be collected if the suspected sign or symptom of breakthrough haemolysis occurs.
- 11. Blood sample for immunogenicity assay will be taken prior to dosing at Weeks 0, 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and ET visit. Blood samples should be collected at the same day of study drug administration. If the administration of IPs is delayed for any reasons after pre-dose blood sampling for immunogenicity assay, blood sample should be recollected on actual dosing day and be used for analysis.
- 12. Investigator and/or designee will assess the PNH-related symptoms including fatigue, haemoglobinuria (discolouration of urine), chest pain, abdominal pain, dyspnoea, dysphagia, and erectile dysfunction.
- 13. Physical examination including height and weight at Screening; physical examination including weight at subsequent visits. Physical examination will be conducted before study drug administration.
- 14. Measured in a sitting position after remaining in a sitting or supine position for at least 5 minutes, including blood pressure, heart rate, and body temperature. On dosing days, vital signs will be taken before study drug administration.
- 15. IV infusion will be performed for  $35 \pm 10$  minutes.
- 16. The switched IP will be received on Week 26 and dosing on Week 26 is the start of Period 2.
- 17. AEs will be collected from the time of signing the informed consent until EOS.
- 18. Concomitant medications will be recorded until EOS.
- 19. Transfusion record will be collected from the time of signing the informed consent until EOS.
- 20. After completion of activities at Week 52, an open-label extended supply of SB12 will be provided for up to 2 calendar years to subjects who have benefited from study treatment and opt to participate in extended supply under an ethical basis. The Week 52 activities must be completed prior to initiation of extended supply. Subjects who are eligible to participate should provide separate informed consent prior to enter an extended supply of SB12.
- 21. Safety follow-up will be done at Week 58 for subjects who complete the study treatments until Week 50, regardless whether subject receives extended supply of SB12 or not. These activities will be conducted either by visit or by phone call on subjects' preference.
- 22. ET visit is defined as 8 weeks after the last dose of SB12 or Soliris®, which may be up to Week 56. Subjects who discontinue from the study at any time post-Day 1 (after the initiation of study drug) before completion of last study treatment at Week 50 will be required to have an ET visit.

# LIST OF ABBREVIATIONS

ADAs Anti-drug antibodies

ADL Activities of daily living

AEs Adverse events

aHUS Atypical haemolytic uremic syndrome

ALP Alkaline phosphatase

ALT Alanine aminotransferase

ANC Absolute neutrophil count

AST Aspartate aminotransferase

ATG Anti-thymocyte globulin

AUEC Area under the effect curve

BUN Blood urea nitrogen

CHO Chinese hamster ovary

CI Confidence interval

COVID-19 Coronavirus Disease 2019

CRO Contract research organisation

CSR Clinical study report

C<sub>trough</sub> Trough serum concentration

CV Coefficient of variation

DNA Deoxyribonucleic acid

DSMB Data and Safety Monitoring Board

DSUR Development Safety Update Report

ECG Electrocardiogram

eCRF Electronic case report form

EMA European Medicines Agency

EOS End of study

ESF Eligibility screening form

ET Early termination

EU European Union

FDA Food and Drug Administration

FSH Follicle stimulating hormone

GCP Good Clinical Practice

gMG Generalised myasthenia gravis

GMP Good Manufacturing Practice

GPI Glycosylphosphatidylinositol

HIV Human immunodeficiency virus

IB Investigator's Brochure

ICF Informed consent form

ICH International Council for Harmonisation

IEC Independent Ethics Committee

IgG Immunoglobulin G

INR International normalised ratio

IP Investigational product

IRB Institutional Review Board

IRRs Infusion-related reactions

IV Intravenous

IWRS Interactive web response system

LDH Lactate dehydrogenase

MAC Membrane attack complex

MAVE Major adverse vascular event

MCH Mean corpuscular haemoglobin

MCHC Mean corpuscular haemoglobin concentration

MCV Mean corpuscular volume

Medical Dictionary for Regulatory Activities

M-FAS Modified Full Analysis Set

MFDS Ministry of Food and Drug Safety

MPV Mean platelet volume

NAbs Neutralising antibodies

NCI-CTCAE

National Cancer Institute-Common Terminology Criteria for Adverse

**Events** 

NMOSD Neuromyelitis optica spectrum disorder

NO Nitric oxide

PC Product Complaints

PD Pharmacodynamic

PDs Protocol deviations

PDS PD Analysis Set

PIG-A Phosphatidylinositol glycan class-A

PK Pharmacokinetic
PKS PK Analysis Set

PNH Paroxysmal nocturnal haemoglobinuria

PPS-AUEC Per-Protocol Set for AUEC of LDH

PPS-single Per-Protocol Set for LDH at a single time point

pRBCs Packed red blood cells

PSUR Periodic Safety Update Report

RAN Randomised Set

RBC Red blood cell

RDW Red cell distribution width

RSI Reference safety information

SAEs Serious adverse events

SAF Safety Set

SAP Statistical analysis plan

SD Standard deviation

SmPC Summary of Product Characteristics

SOP Standard operating procedure

TEAEs Treatment-emergent adverse events

TOST Two one-sided test

ULN Upper limit of normal

US United States of America

WBC White blood cell

WHO-DDE World Health Organization-Drug Dictionary Enhanced

# **TABLE OF CONTENTS**

| SYNOPSIS | 2 |
|---------------------------------------------------|----|
| GRAPHICAL STUDY DESIGN AND SCHEDULE OF ACTIVITIES | 9 |
| LIST OF ABBREVIATIONS | 15 |
| TABLE OF CONTENTS | 18 |
| LIST OF TABLES | 23 |
| LIST OF FIGURES | 23 |
| LIST OF STUDY STAFF | 24 |
| 1. INTRODUCTION | |
| 1.1. Paroxysmal Nocturnal Haemoglobinuria | 25 |
| 1.2. Overview of SB12 | 25 |
| 1.2.1. Non-clinical Studies of SB12 | 26 |
| 1.2.2. Clinical Pharmacology of SB12 | 26 |
| 1.3. Comparator Investigational Product: Soliris® | 26 |
| 1.3.1. Non-clinical Data of Soliris® | 26 |
| 1.3.2. Clinical Data of Soliris <sup>®</sup> | 27 |
| 1.4. Study Rationale | 28 |
| 1.5. Risk and Benefit Assessment | 28 |
| 1.5.1. Known Potential Risks | 28 |
| 1.5.2. Known Potential Benefits | 29 |
| 1.5.3. Assessment of Potential Risks and Benefits | 29 |
| 2. STUDY OBJECTIVES AND ENDPOINTS | 29 |
| 2.1. Study Objectives | 29 |
| 2.1.1. Primary Objective | 29 |
| 2.1.2. Secondary Objectives | 29 |
| 2.2. Endpoints | 30 |
| 2.2.1. Primary Endpoints | 30 |
| 2.2.2. Secondary Endpoints | 30 |
| 3. STUDY DESIGN | 31 |
| 3.1. Overview of Study Design | |
| 3.2. Rationale for Study Design | |
| 3.2.1. Scientific Rationale for Study Design | |
| $\sim$ $\sim$ | |

| 3.2.2. Rationale for Dose Selection | 32 |
|------------------------------------------------------------------------|----|
| 3.2.3. Rationale for Pharmacokinetic Assessments | 32 |
| 3.2.4. Rationale for Immunogenicity Assessments | 32 |
| 3.3. Duration of Study Participation | 32 |
| 3.4. Number of Subjects | 33 |
| 3.5. End of Study Definition | 33 |
| 4. STUDY POPULATION | 33 |
| 4.1. Overview | 33 |
| 4.2. Inclusion Criteria | 33 |
| 4.3. Exclusion Criteria | 34 |
| 4.4. Screen Failures and Re-screening | 35 |
| 5. TREATMENT AND INVESTIGATIONAL PRODUCT | 35 |
| 5.1. Treatment of the Subjects | 35 |
| 5.1.1. Dosing and Treatment Schedule | 35 |
| 5.1.2. Assignment of Subjects to Treatment Sequence | 36 |
| 5.1.3. Blinding | 36 |
| 5.2. Investigational Product | 36 |
| 5.2.1. Identity of Investigational Product | 36 |
| 5.2.2. Formulation, Packaging, and Labelling | 37 |
| 5.2.3. Product Storage and Stability | 37 |
| 5.2.4. Preparation and Administration of Investigational Products | 37 |
| 5.2.5. Treatment Compliance and Investigational Product Accountability | 38 |
| 5.3. Concomitant Medication or Treatment | 39 |
| 5.3.1. Permitted Concomitant Medications or Treatment | 39 |
| 5.3.2. Prohibited Concomitant Medications or Treatment | 39 |
| 6. STUDY ASSESSMENT | 39 |
| 6.1. Efficacy Assessment | 39 |
| 6.1.1. Disease-related Laboratory Parameters | 39 |
| 6.1.2. Breakthrough Haemolysis | 40 |
| 6.1.3. Transfusions | 40 |
| 6.1.4. Major Adverse Vascular Events | 40 |
| 6.1.5. Paroxysmal Nocturnal Haemoglobinuria-related Symptoms | 40 |

| 6.2. Safety Assessment | 41 |
|-----------------------------------------------------|----|
| 6.2.1. Adverse Events | 41 |
| 6.2.2. Clinical Laboratory Evaluations | 41 |
| 6.2.3. Physical Examinations | 43 |
| 6.2.4. Twelve-lead Electrocardiograms | 43 |
| 6.2.5. Vital Signs | 43 |
| 6.3. Other Assessments | 43 |
| 6.3.1. Pharmacokinetic Assessments | 43 |
| 6.3.2. Immunogenicity Assessments | 43 |
| 6.3.3. Pharmacodynamic Assessments | 44 |
| 6.3.4. Pharmacogenetic Assessments | 44 |
| 7. STUDY PROCEDURES | 45 |
| 7.1. Study Flow and Visit Schedule | 45 |
| 7.1.1. Screening Period | 45 |
| 7.1.2. Randomisation | 47 |
| 7.1.3. Treatment Period | 47 |
| 7.1.4. Unscheduled Visits | 50 |
| 7.2. Discontinuation | 50 |
| 7.2.1. Subject Discontinuation from Study Treatment | 50 |
| 7.2.2. Investigational Site Discontinuation | 52 |
| 7.3. Early Termination of the Study | 52 |
| 8. SAFETY MONITORING AND REPORTING | 52 |
| 8.1. Adverse Events | 52 |
| 8.1.1. Definition of Adverse Event | 52 |
| 8.1.2. Period of Observation for Adverse Events | 53 |
| 8.1.3. Reporting Adverse Events | 53 |
| 8.1.4. Severity Assessment | 53 |
| 8.1.5. Causality Assessment. | 54 |
| 8.1.6. Expectedness Assessment | 54 |
| 8.1.7. Withdrawal due to Adverse Events | 54 |
| 8.2. Serious Adverse Events | 54 |
| 8.2.1. Definition of Serious Adverse Event | 54 |

| 8.2.2. Reporting Serious Adverse Events | 56 |
|---------------------------------------------------------------------|----|
| 8.3. Adverse Events of Special Interest | 56 |
| 8.3.1. Meningococcal Infection | 56 |
| 8.3.2. Other Systemic Infections | 57 |
| 8.3.3. Infusion-related Reactions | 57 |
| 8.4. Pregnancy | 58 |
| 8.4.1. Pregnancy Prevention | 58 |
| 8.5. Emergency Unblinding of Assigned Treatment | 59 |
| 8.6. Independent Data and Safety Monitoring Board | 59 |
| 9. STATISTICAL METHODS AND DATA ANALYSIS | 59 |
| 9.1. Statistical Hypotheses | 59 |
| 9.2. Analysis Sets | 60 |
| 9.3. Subject Demographic and Baseline Characteristics | 60 |
| 9.4. Analysis of the Primary Objectives | 61 |
| 9.5. Analysis of the Secondary Objectives | 61 |
| 9.5.1. Efficacy Variable Analyses | 61 |
| 9.5.2. Safety Analyses | 62 |
| 9.5.3. Pharmacokinetic Analyses | 62 |
| 9.5.4. Immunogenicity Analyses | 62 |
| 9.5.5. Pharmacodynamic Analyses | 62 |
| 9.6. Sample Size Calculations | 62 |
| 10. DATA COLLECTION AND MANAGEMENT | 64 |
| 10.1. Data Confidentiality | 64 |
| 10.2. Monitoring | 64 |
| 10.3. Data Handling and Record Keeping | 65 |
| 10.4. Future Use of Stored Specimens and Data | 65 |
| 10.5. Database Management and Coding | 65 |
| 10.6. Quality Control and Quality Assurance | 66 |
| 10.7. Protocol Deviation | 66 |
| 11. ETHICS CONSIDERATIONS AND ADMINISTRATIVE PROCEDURES | 66 |
| 11.1. Institutional Review Boards and Independent Ethics Committees | 66 |
| 11.2. Ethical Conduct of the Study | 67 |

# **SAMSUNG BIOEPIS**

| 11.3. Written Informed Consent | 67 |
|----------------------------------------------------|---------|
| 11.4. Investigator Information | 67 |
| 11.4.1. Investigator Obligations | 67 |
| 11.4.2. Training of Investigational Site Personnel | 67 |
| 11.4.3. Protocol Signatures | 67 |
| 11.4.4. Financing and Insurance | 68 |
| 12. PUBLICATION POLICY | 68 |
| 13. EXTENDED SUPPLY | 69 |
| 14. REFERENCES | 70 |
| APPENDIX A. PAROXYSMAL NOCTURNAL HAEMOGLOBINURIA S | YMPTOMS |
| SUBJECT QUESTIONNAIRE | 72 |
| PROTOCOL SIGNATURE PAGES | 73 |
| CHANGE HISTORY OF PROTOCOL AMENDMENT | 76 |
| Amendment 1: Version 2.0, Oct 08, 2018 | 76 |
| Amendment 2: Version 3.0, Dec 12, 2018 | 82 |
| Amendment 3: Version 4.0, Nov 29, 2019 | 91 |
| Amendment 4: Version 5.0, Aug 21, 2020 | 138 |
| Amendment 5: Version 6.0, Nov 27, 2020 | 166 |

# **LIST OF TABLES**

| Table 1. Schedule of Activities (Period 1, before Cross-over) | 10 |
|---|---|
| Table 2. Schedule of Activities (Period 2 and Safety Follow-up/ET, after Cross-over) | 13 |
| Table 3. Investigational Products Description | 36 |
| Table 4. Parameters for Clinical Laboratory Tests | 42 |
| Table 5. Severity Grade of NCI-CTCAE v5.0 | 53 |
| Table 6. LDH Level from Reference Studies | 63 |
| LIST OF FIGURES | |
| Figure 1. Graphical Study Design | 9 |

# LIST OF STUDY STAFF



#### 1. Introduction

# 1.1. Paroxysmal Nocturnal Haemoglobinuria

Paroxysmal nocturnal haemoglobinuria (PNH) is an acquired haematopoietic disorder characterised by intravascular haemolysis and manifested by haemoglobinuria, anaemia, and venous thrombosis, which in turn produces severe and even potentially fatal clinical consequences. PNH is a very rare disease with a prevalence of about 16 per million people, and it can present at any range but mainly occurs in young adults, with the usual age at diagnosis being early 30s [1; 2; 3].

PNH results from a somatic mutation in the phosphatidylinositol glycan class-A (PIG-A) gene which is necessary for the synthesis of glycosylphosphatidylinositol (GPI)-anchors. The mutation leads to a deficiency of the GPI-anchored terminal complement inhibitors (e.g., CD55, CD59) on the surface of clonal populations of haematopoietic stem cells. Normally CD59 forms a defensive shield for red blood cells (RBCs) against complement-mediated lysis and inhibits the assembly of the membrane attack complex (MAC). The CD55 prevents formation and augments instability of the C3 convertases, attenuating the complement cascade. Without these complement inhibitors on the surface of cells, the cells are subjected to complement-mediated haemolysis, which in turn produces the clinical manifestations of the disease. The clinical features of the PNH arise as a result of complement-mediated haemolysis in unprotected RBCs, leukocytes, and platelets as well as the release of free haemoglobin that occurs with RBCs destruction [4].

Haemolysis contributes significantly to the anaemia and treatment is indicated for the following reasons: (1) Patients with chronic haemolysis complain of lethargy, malaise, myalgia, and loss of sense of well-being that diminishes significantly quality of life; (2) there is evidence that chronic haemolysis has an untoward effect on renal function; (3) the dysphagia and male impotence of PNH appear related to haemolysis; (4) a correlation between thrombosis and haemolysis may exist [5].

Conventional treatment options such as corticosteroids were limited, and the outcome of treatment was often unsatisfactory. Bone marrow transplantation is a curative treatment for PNH, but the procedure has risks of transplant-related morbidity and mortality and most PNH patients lack a suitable donor [6].

Soliris® (eculizumab, Alexion Pharmaceuticals, Inc.) is a humanised monoclonal antibody that blocks terminal complement by binding to C5 and is the approved therapy for PNH. The drug is highly effective in stopping intravascular haemolysis, eliminating or decreasing the need for RBC transfusions, improving quality of life, and reducing the risk of thrombosis, the leading cause of mortality from PNH [7; 8; 9].

# 1.2. Overview of SB12

SB12 has been developed as a similar biological medicinal product to Soliris® (eculizumab, Alexion Pharmaceuticals, Inc.). Soliris® is currently indicated for the treatment of patients with PNH, atypical haemolytic uremic syndrome (aHUS), refractory generalised myasthenia gravis (gMG), and neuromyelitis optica spectrum disorder (NMOSD) [10; 21]. SB12 and Soliris® have identical primary structure and the active substance for both products is eculizumab, a humanised monoclonal antibody (immunoglobulin G[IgG]2/4 kappa) that binds to the human C5 complement protein with high affinity. Binding to this protein blocks its cleavage into C5a and C5b, thereby inhibiting terminal complement-mediated intravascular haemolysis.

SB12 is produced by recombinant deoxyribonucleic acid (DNA) technology in a chinese hamster ovary (CHO) mammalian cell expression system and purified by various affinity and ion exchange chromatography steps that include specific viral inactivation and removal procedures.

According to the guideline International Council for Harmonisation (ICH) Q6B, characterisation of a biological therapeutic must involve its physicochemical properties, biological activities, purity, impurities, and quantity. The characterisation study will employ the 'state-of-the-art' analytical methods in order to investigate the primary, secondary, higher-order structures, and the post-translational modifications associated the structural heterogeneity, the charge variants, the purity, and the biological activities. It was demonstrated that SB12 has similar structural, physicochemical, and biological characteristics with Soliris<sup>®</sup>.

#### 1.2.1. Non-clinical Studies of SB12

As outlined in the "Guideline on similar biological medicinal products containing monoclonal antibodies" [11], a risk-based approach was taken to the non-clinical evaluation of SB12. A series of *in vitro* biologic activity studies was performed in order to demonstrate similarity between SB12 and Soliris®. In addition, *in vivo* non-clinical study may not be necessary to provide non-clinical evidence of similarity between the two products, as eculizumab does not inhibit C5 in animal species. Therefore, no pharmacology or toxicology studies were conducted with eculizumab in normal rodents or non-human primates. Also, non-clinical safety pharmacology, reproductive and developmental toxicity, and carcinogenicity studies were not performed, as they are not required for non-clinical testing of biosimilars as outlined in the "Guideline on similar biological medicinal products containing monoclonal antibodies" [11]. There were no significantly different results observed in the *in vitro* studies between SB12 and Soliris®.

# 1.2.2. Clinical Pharmacology of SB12

Based on biosimilarity between SB12 and Soliris®, which was demonstrated through extensive quality and non-clinical similarity exercise, a Phase I study was conducted in healthy subjects to compare the pharmacokinetic (PK), safety, tolerability, immunogenicity, and pharmacodynamic (PD) profiles and a Phase III study will be conducted in subjects with PNH to compare the efficacy, safety, pharmacokinetics, and immunogenicity of SB12 to Soliris®. Information on the safety of SB12 based on the product information of Soliris®, non-clinical, and clinical exercise is presented in the Investigator's Brochure (IB).

# 1.3. Comparator Investigational Product: Soliris®

# 1.3.1. Non-clinical Data of Soliris®

The tissue cross-reactivity of eculizumab was evaluated by assessing binding to a panel of 38 human tissues. C5 expression in the human tissue panel examined in this study is consistent with published reports of C5 expression, as C5 has been reported in smooth muscle, striated muscle, and renal proximal tubular epithelium. No unexpected tissue cross-reactivity was observed.

Animal reproduction studies have not been conducted with eculizumab due to lack of pharmacologic activity in non-human species and no animal studies have been conducted to evaluate the genotoxic and carcinogenic potential of eculizumab.

In a 26-week toxicity study performed in mice with a surrogate antibody directed against murine C5, treatment did not affect any of the toxicity parameters examined. Haemolytic activity during the course of the study was effectively blocked in both female and male mice.

No clear treatment-related effects or adverse effects were observed in reproductive toxicology studies in mice with a surrogate terminal complement inhibitory antibody, which was utilised to assess the reproductive safety of C5 inhibitor. These studies included assessment of fertility and early embryonic development, developmental toxicity, and pre and post-natal development.

When maternal exposure to the antibody occurred during organogenesis, two cases of retinal dysplasia and one case of umbilical hernia were observed among 230 offspring born to mothers exposed to the higher antibody dose (approximately 4 times the maximum recommended human Soliris® dose, based on a body weight comparison); however, the exposure did not increase foetal loss or neonatal death.

Regarding *in vivo* non-clinical study, the publicly available information of Soliris® performed a species cross-reactivity of eculizumab to the functional complement C5 inhibition activity of eculizumab in human serum samples compared to primate and non-primate serum samples including eight-different species. The result concluded that there is no cross-reactivity of the eculizumab with non-primate species and primate species and that the result suggests that eculizumab effectively inhibits C5 only in human serum. In this context, the *in vivo* study in irrelevant non-primate animal species is unlikely to provide any additional meaningful non-clinical evidence.

# 1.3.2. Clinical Data of Soliris®

In 40 patients with PNH, a 1-compartmental model was used to estimate PK parameters after multiple doses. Mean clearance was  $0.31 \pm 0.12$  mL/h/kg, mean volume of distribution was  $110.3 \pm 17.9$  mL/kg, and mean elimination half-life was  $11.3 \pm 3.4$  days. The steady state is achieved by 4 weeks using the PNH adult dosing regimen.

In PNH patients, PD activity correlates directly with eculizumab serum concentrations and maintenance of trough levels above  $\geq$  35  $\mu g/mL$  results in essentially complete blockade of haemolytic activity in the majority of PNH patients.

The safety and efficacy of Soliris® in PNH patients were assessed in a randomised, double-blind, placebo-controlled 26-week study (C04-001). PNH patients were also treated with Soliris® in a single arm 52-week study (C04-002) and in a long term extension study (E05-001). Patients received meningococcal vaccination prior to receipt of Soliris®. In all studies, the dose of eculizumab was 600 mg every  $7 \pm 2$  days for 4 weeks, followed by 900 mg  $7 \pm 2$  days later, then 900 mg every  $14 \pm 2$  days for the study duration. Soliris® was administered as an intravenous (IV) infusion over 25-45 minutes. An observational non-interventional registry in patients with PNH (M07-001) was also initiated to characterise the natural history of PNH in untreated patients and the clinical outcomes during Soliris® treatment.

In study C04-001 (TRIUMPH), PNH patients with at least 4 transfusions in the prior 12 months, flow cytometric confirmation of at least 10% PNH cells, and platelet counts of at least 100,000/µL were randomised to either Soliris<sup>®</sup> (n = 43) or placebo (n = 44). Prior to randomisation, all patients underwent an initial observation period to confirm the need for RBC transfusion and to identify the haemoglobin concentration (the 'set-point') which would define each patient's haemoglobin stabilisation and transfusion outcomes. The haemoglobin set-point was less than or equal to 9 g/dL in patients with symptoms and was less than or equal to 7 g/dL in patients without symptoms. Primary efficacy endpoints were haemoglobin stabilisation (patients who maintained a haemoglobin concentration above the haemoglobin set-point and avoid any RBC transfusion for the entire 26-week period) and blood transfusion requirement. Fatigue and health-related quality of life were relevant secondary endpoints. Haemolysis was monitored mainly by the measurement of serum lactate dehydrogenase (LDH) levels, and the proportion of PNH RBCs was monitored by flow cytometry. Patients receiving anticoagulants and systemic corticosteroids at baseline continued these medications. Major baseline characteristics were balanced. Study patients treated with Soliris® had significantly reduced (p < 0.001) haemolysis resulting in improvements in anaemia as indicated by increased haemoglobin stabilisation and reduced need for RBC transfusions compared to placebo treated patients. These effects were seen among patients within each of the three pre-study RBC transfusion strata (4-14 units; 15-25 units; > 25 units). After 3 weeks of Soliris® treatment, patients reported less fatigue and improved health-related quality of life.

Because of the study sample size and duration, the effects of Soliris® on thrombotic events could not be determined.

In the non-controlled study C04-002 (SHEPHERD), PNH patients with at least one transfusion in the prior 24 months and at least 30,000 platelets/µL received Soliris® over 52-week period. Concomitant medications included anti-thrombotic agents in 63% of the patients and systemic corticosteroid in 40% of the patients. Ninety-six of the 97 enrolled patients completed the study (one patient died following a thrombotic event). A reduction in intravascular haemolysis as measured by serum LDH levels was sustained for the treatment period and resulted in increased transfusion avoidance, a reduced need for RBC transfusion and less fatigue.

## 1.4. Study Rationale

Patients with PNH suffer from severe impaired quality of life arising from haemolysis leading to anaemia, thrombosis, renal impairment, and fatigue, which are the most common morbidities for this disease, with a significant increase in free haemoglobin levels. Cell-free haemoglobin consumes the serum nitric oxide (NO) and reduction in serum NO causes smooth muscle dystonia including vasoconstriction and gastrointestinal contractions and these consequences induce abdominal pain, dysphagia, pulmonary hypertension, dyspnoea, or erectile dysfunction [12; 13; 14; 15; 16]. Low serum NO also results in platelet activation/aggregation and thrombosis which may lead arterial myocardial infarction or cerebral vascular accident [12].

Thrombosis and renal failure are the leading cause of death in PNH and PNH patients with haemolysis whose LDH level is equal to or greater than 1.5 × upper limit of normal (ULN) showed a 4.8-fold increase in mortality rate compared with the general population [16].

Currently there are no approved treatments for PNH except for Soliris<sup>®</sup> but several types of supportive care have no any impact on progression or risk of severe morbidities and mortality. Unfortunately eculizumab does not alter the underlying defect of the disease, thus, treatment needs to continue lifelong or until spontaneous remission, however Soliris<sup>®</sup> is barely affordable for the most of PNH patients as it costs 700,000 USD a year [1; 17].

Considering all the treatment options available, it is highly expected there are still patient needs for the right treatment with reasonable price. SB12 would meet this patient needs in extending the treatment opportunity by providing the medicine with lower price than the originator.

#### 1.5. Risk and Benefit Assessment

#### 1.5.1. Known Potential Risks

According to Soliris<sup>®</sup> Summary of Product Characteristics (SmPC) [10], supportive safety data were collected from 31 completed clinical studies that included 1,503 patients exposed to eculizumab in complement-mediated disease populations, including PNH, aHUS, refractory gMG and NMOSD. The most common adverse reaction was headache (occurred mostly in the initial phase) and the most frequently reported serious adverse reaction was meningococcal sepsis.

Considering the mechanism of action of eculizumab, C5 inhibition is known to increase the susceptibility to infection caused by encapsulated bacteria, especially by *Neisseria meningitidis*. In order to minimise the risk of meningococcal infection, all subjects participating in this study will receive meningococcal vaccines according to current local guidelines or Soliris® SmPC before investigational product (IP) administration. However, vaccination may not be sufficient to prevent meningococcal infection. Consideration will be given to current local guidelines and/or the discretion of the Investigator on the appropriate use of antibacterial agents. All subjects will be monitored for early signs of

meningococcal infection, evaluated immediately if infection is suspected, and treated with appropriate antibiotics if necessary.

According to the study design, the switch of IP (cross-over) occurs during the study. The potential negative impact from this IP switch is considered to be minimal given similarity and comparability of SB12 to Soliris<sup>®</sup> and low antibody responses in Soliris<sup>®</sup> (3.4%) similar to that of placebo (4.8%) in placebo controlled studies in subjects with PNH [10].

In order to ensure the safety of subjects who participate in the study, the followings will be performed during the study. This study will take place at multicentre with accessible medical facilities which will allow immediate treatment of medical emergencies. All study related procedures will be conducted by medical staff with appropriate level of training and expertise and an understanding of the IPs, its target and mechanism of action. Subjects will have a safety follow-up until 8 weeks after the last dose of study drug. An independent Data and Safety Monitoring Board (DSMB) will convene at pre-specified intervals to conduct interim monitoring of accumulating safety data. Following each data review, the DSMB will make recommendations regarding the conduct of the study, including continuation of the study without modifications, modification of the protocol, pausing of subject enrolment until the resolution of issues, or termination of the study for safety reasons.

#### 1.5.2. Known Potential Benefits

Soliris® is the approved therapy for PNH and is indicated for the treatment patients with aHUS, gMG, and NMOSD [10; 21]. The drug is highly effective in stopping intravascular haemolysis, eliminating or decreasing the need for RBC transfusions, improving quality of life, and reducing the risk of thrombosis, the leading cause of mortality from PNH [7; 8; 9].

Although clinical data is currently unavailable, SB12 is expected to have similar clinical outcome to Soliris® based on the physicochemical and biological similarity.

# 1.5.3. Assessment of Potential Risks and Benefits

The available data demonstrate a high degree of physicochemical and biological similarity of SB12 with the reference medicinal product (Soliris®). The suitability of the methodology employed to evaluate the similarity of SB12 and Soliris® in a pharmaceutical setting and these data were confirmed by the European Medicines Agency (EMA) and the United States of America (US) Food and Drug Administration (FDA). The known and potential risks of receiving SB12 are expected to be similar to those seen with Soliris®. In conclusion, sufficient evidence exists for the justification of the administration of SB12, as a similar biological medicinal product of Soliris®, to subjects with PNH.

The study protocol provides adequate instructions for the detection and treatment of adverse events (AEs) arising following the administration of the IP.

# 2. Study Objectives and Endpoints

# 2.1. Study Objectives

#### 2.1.1. Primary Objective

The primary objective of this study is to demonstrate comparable clinical efficacy of SB12 and Soliris<sup>®</sup>, by evaluating the LDH in subjects with PNH.

# 2.1.2. Secondary Objectives

The secondary objectives are:

- To evaluate the efficacy of SB12 compared to Soliris® by
  - LDH profile over time
  - Number of units of packed red blood cells (pRBCs) transfused
- To evaluate the safety and tolerability of SB12 compared to Soliris®
- To evaluate the PK of SB12 compared to Soliris<sup>®</sup>
- To evaluate the immunogenicity of SB12 compared to Soliris®
- To evaluate the PD of SB12 compared to Soliris®

# 2.2. Endpoints

# 2.2.1. Primary Endpoints

- LDH level (U/L) at Week 26
- Time-adjusted area under the effect curve (AUEC) of LDH from Week 14 to Week 26 and from Week 40 to Week 52

# 2.2.2. Secondary Endpoints

# **Efficacy endpoints**

- LDH profile over time
- Number of units of pRBCs transfused throughout the study period

## **Safety endpoints**

- Incidence of AEs
- Incidence of serious AEs (SAEs)
- Incidence of infection-related AEs
  - Meningococcal infection
  - Other systemic infection
- Incidence of infusion-related reactions (IRRs)

Safety of subjects will be monitored by 12-lead electrocardiogram (ECG), vital sign assessment, and physical examination. Haematological, biochemical, and urinalysis laboratory parameters will be also measured.

# PK endpoint

Concentration prior to infusion (trough serum concentration [C<sub>trough</sub>]) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, and 52

# **Immunogenicity endpoints**

- Incidence of anti-drug antibodies (ADAs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and early termination (ET) visit
- Incidence of neutralising antibodies (NAbs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, Samsung Bioepis * Information*

30, 32, 36, 40, 44, 48, 52, and ET visit

#### PD endpoint

• Terminal complement activity at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 26, 28, 30, 32, 36, 40, and 52

# 3. Study Design

# 3.1. Overview of Study Design

This is a randomised, Phase III, double-blind, multicentre, cross-over study to compare the efficacy, safety, pharmacokinetics, and immunogenicity between SB12 and Soliris® in subjects with PNH.

Subjects will be randomised in a 1:1 ratio to treatment sequence I (SB12 to Soliris®) or treatment sequence II (Soliris® to SB12). Subjects randomly assigned to treatment with SB12 or Soliris® will receive 600 mg of eculizumab IV every week for first 4 weeks (initial phase) and 900 mg for the fifth week, followed by 900 mg every 2 weeks thereafter. Subjects who are randomised to initially receive SB12 will be switched to receive Soliris® and subjects who are randomised to initially receive Soliris® will be switched to receive SB12 at Week 26. SB12 or Soliris® will be given until Week 50. However, in special circumtances of a shortage of the comparator, to ensure continuity of study treatment for the duration of study, the Sponsor will provide SB12 instead of Soliris® in a blinded manner.

Details of assessment that will be conducted and treatment that will be administered are presented in, Table 1 and Table 2. The last assessment will be performed at Week 58 or 8 weeks after the last dose of SB12 or Soliris<sup>®</sup> in case of ET.

After completion of activities at Week 52, an open-label extended supply of SB12 will be provided for up to 2 calendar years to subjects who have benefited from study treatment and opt to participate in extended supply under an ethical basis.

# 3.2. Rationale for Study Design

# 3.2.1. Scientific Rationale for Study Design

It is acknowledged that PNH is a rare disease with an estimated incidence of 0.1-0.2/100,000 persons/year [18] and executing an adequately powered comparative trial is therefore challenging. The guiding principle of a biosimilar development is, however to demonstrate similar clinical efficacy and safety compared to the reference medicinal product, not patient benefit per se, which has already been shown for the reference medicinal product [11]. In view of this, the two arms design with randomisation between SB12 and Soliris® is endorsed. And in view of the very limited sample size (approximately 50 subjects), the study will be conducted in treatment-naïve patients to allow proper evaluation of safety and immunogenicity of the compound, as it reduces heterogeneity of the population.

LDH has been considered an authentic and useful clinical marker and direct measure of intravascular haemolysis in patients with PNH, published data support. And also, LDH is useful in evaluating response to treatment, as its level decreases along with the reduction of the haemolytic rate, which has been described in PNH following treatment [19; 20]. Results from the eculizumab clinical study showed that serum LDH levels continued markedly elevated and unchanged in untreated patients, while eculizumab treated patients had an immediate reduction in serum LDH to normal or near normal level [10; 21]. The reduction of serum LDH level reflected a rapid, sustained reduction in haemolysis and improvement in fatigue as well [9].

This study has two different primary endpoints, depending on regulatory agency's requirements for

assessing equivalence in efficacy between SB12 and Soliris®.

for analysis of haemolysis reduction as measured by time-adjusted AUEC of LDH between two different time points in each period, the primary objective is to demonstrate comparable clinical efficacy of SB12 and Soliris® in terms of time-adjusted AUEC of LDH from Week 14 to Week 26 and from Week 40 to Week 52.

for analysis of haemolysis reduction as measured by the LDH level at single time point, the primary objective is to demonstrate comparable clinical efficacy of SB12 and Soliris<sup>®</sup> in terms of the LDH level (U/L) at Week 26.

#### 3.2.2. Rationale for Dose Selection

The dosing regimen for adult patients ( $\geq$  18 years of age) of Soliris<sup>®</sup> is approved for the treatment of PNH as 4-week initial phase followed by a maintenance phase as below:

- Initial phase: 600 mg of Soliris® administered via a 25-45 minutes IV infusion every 7 days for the first 4 weeks
- Maintenance phase: 900 mg of Soliris® administered via a 25-45 minutes IV infusion for the fifth week, followed by 900 mg of Soliris® administered via a 25-45 minutes IV infusion every  $14 \pm 2$  days

As SB12 is a proposed biosimilar of Soliris®, an identical dose is selected for both treatments.

#### 3.2.3. Rationale for Pharmacokinetic Assessments

A randomised, three-arm, parallel, single-dose Phase I PK study was conducted in healthy subjects to demonstrate similarity in PK profiles of SB12, European Union (EU) sourced Soliris<sup>®</sup>, and US sourced Soliris<sup>®</sup>. However, since target-mediated clearance of eculizumab can be more accurately investigated in patients, additional PK assessments will be performed in this Phase III study to provide supportive evidence to PK similarity.

# 3.2.4. Rationale for Immunogenicity Assessments

Biological/biotechnology-derived proteins can induce an unwanted immune response that is triggered by more than a single factor and the consequence of immunogenicity may vary considerably, ranging from irrelevant to therapy to serious and life-threatening. Immune responses may affect both safety and effectiveness such as altering PK, inducing anaphylaxis, or promoting development of NAbs that neutralise the product as well as its endogenous protein counterpart.

In all clinical studies of Soliris<sup>®</sup>, the frequency of ADAs has been reported as 0.0% to 4.8%. In PNH placebo controlled studies, low antibody responses have been reported with a frequency (3.4%) similar to that of placebo (4.8%). There has been no observed correlation of antibody development to clinical response or AEs.

For subject safety and for demonstrating biosimilarity, immunogenicity will be assessed in this study according to the recommended guideline.

# 3.3. Duration of Study Participation

After Screening, the duration of study participation will be 58 weeks per subject including 50 weeks of treatment and 8 weeks of post-treatment follow-up. After completion of study treatment, subjects may be entered into an extended supply of up to 2 years.

# 3.4. Number of Subjects

Approximately 50 subjects (25 subjects per treatment sequence) are planned to be randomised in this study over a planned recruitment period.

# 3.5. End of Study Definition

A subject is considered to have completed the study if he or she has completed all study treatment and the last visit or the last scheduled procedure shown in Table 2. The end of study (EOS) is defined as completion of safety follow-up at Week 58 or completion of ET visit (8 weeks after the last dose of SB12 or Soliris<sup>®</sup>). The end of this clinical study is defined as completion of the last subject's EOS.

# 4. Study Population

#### 4.1. Overview

The study population for this study is subjects with PNH.

#### 4.2. Inclusion Criteria

Subjects must meet all of the following criteria to be eligible for the study:

- 1. Male or female aged 18 or older at the time of signing the informed consent form (ICF), if local regulations are different in this regard, follow the local regulations.
- 2. Documented diagnosis of PNH.
- 3. Presence of the PNH white blood cell (WBC) clone, with a granulocyte or monocyte clone size of  $\geq 10\%$  by high-sensitivity flow cytometry at Screening.
- 4. Documented LDH level  $\geq 1.5 \times \text{ULN}$  at Screening.
- 5. History of transfusion for anaemia within 12 months prior to Screening or having PNH-related symptoms (e.g., fatigue, haemoglobinuria, abdominal pain, chest pain, shortness of breath [dyspnoea], dysphagia, erectile dysfunction) at Screening.
- 6. All subjects must be vaccinated against *Neisseria meningitidis* within 3 years prior to or on Day 1 in accordance with current local guidelines or Soliris® SmPC to reduce the risk of meningococcal infection.
- 7. Female subjects who are not pregnant or nursing at Screening and on initiation of study drug (Day 1) and who are not planning to become pregnant from Screening until 5 months after the last dose of study drug.
- 8. Subjects and their partners of childbearing potential (female or male) who agree to use of a highly effective contraceptive method (e.g., established use of oral, injected or implanted hormonal contraceptive, placement of an intrauterine device or intrauterine system, male sterilisation, or true abstinence [see Section 8.4.1]) from Screening until 5 months after the last dose of study drug.
- 9. Subjects must be able to understand the implications of taking part in the study and be willing to follow the study instructions and requirements fully.

10. Subjects must be able to provide informed consent, which must be obtained prior to any study related procedures.

#### 4.3. Exclusion Criteria

Subjects meeting any of the following criteria are not eligible for the study:

- 1. Previous treatment with a complement pathway inhibitor (including eculizumab).
- 2. Known hypersensitivity to the IP or any of the ingredients or excipients of the IP.
- 3. Known contraindication/hypersensitivity for meningococcal vaccine or the antibiotic to be used in the study.
- 4. Abnormal haematological parameters at Screening defined as the following:
  - a. Absolute neutrophil count (ANC)  $\leq 0.5 \times 10^3 / \mu L$
  - b. Platelet count  $< 70 \times 10^3 / \mu L$
- 5. History of meningococcal disease.
- 6. History of haematopoietic stem cell transplantation.
- 7. History of serious thrombotic event (e.g., stroke, myocardial infarction, pulmonary embolism, etc.).
- 8. Known or suspected active bacterial, virus, fungal infection within 30 days prior to initiation of study drug (Day 1).
- 9. Known history of human immunodeficiency virus (HIV) infection or have positive results at Screening.
- 10. Concomitant use of any of the following medications is prohibited if the following conditions apply.
  - a. Erythropoietin, systemic corticosteroids, low-molecular-weight heparins, iron supplements, and androgen therapy that have not been on a stable dose for at least 4 weeks prior to initiation of study drug (Day 1).
  - b. Warfarin with an unstable international normalised ratio (INR) for at least 4 weeks prior to initiation of study drug (Day 1) at the discretion of the Investigator.
  - c. Cyclosporine that has not been on a stable dose for at least 8 weeks prior to initiation of study drug (Day 1).
- 11. Subjects who have received or participated in another investigational drug, device, or procedures within 30 days or within 5 half-lives of that IP prior to Screening, whichever is greater.

- 12. History of malignancy within 5 years prior to Screening, except for curatively treated carcinoma in situ of uterine cervix, basal cell carcinoma of the skin, or squamous cell carcinoma of the skin.
- 13. Any other cardiac, hepatic, immunologic, pulmonary, rheumatoid disease, other conditions causing rise in LDH (e.g., tumours, muscular dystrophies, liver and bile disease, etc.), or the disorder which, at the discretion of the Investigator, will put the subjects at risk if they are enrolled.
- 14. Other unspecified reasons that, at the discretion of the Investigator or Sponsor, make the subjects unsuitable for enrolment.

# 4.4. Screen Failures and Re-screening

Screen failures are defined as subjects who consent to participate in the clinical trial but do not meet one or more criteria required for participation in the trial during the screening procedures. A minimal set of screen failure information is required.

Subjects who are screen failure due to technical issue, not medical issue, might be re-screened once based on discussion and agreement between the Investigator and the medical monitor.

During Coronavirus Disease 2019 (COVID-19) pandemic circumstances, eligibility may not be confirmed at Screening due to unexpected COVID-19 related restrictions. These cases may fall into screen failures due to out of 42 days screening window or consent withdrawal related with COVID-19 concern, etc. These will be considered as technical issue so that re-screening is applicable after COVID-19 related restrictions are relieved.

# 5. Treatment and Investigational Product

#### 5.1. Treatment of the Subjects

# 5.1.1. Dosing and Treatment Schedule

SB12 or Soliris® will be administered up to Week 50 (a total of 28 administrations of IP) unless they are early discontinued from study treatment. Dosing and treatment schedule should be kept as follows:

- 600 mg every  $7 \pm 2$  days for the first 4 weeks, followed by
- 900 mg for the fifth dose (Week 4)  $7 \pm 2$  days later, then
- 900 mg every  $14 \pm 2$  days thereafter

The treatment schedule is dependent on the previous treatment date rather than the absolute (i.e., fixed) number of days from Day 1. In other words, the next  $7 \pm 2$  days or  $14 \pm 2$  days treatment schedule described above is re-scheduled every time based on the date when the previous treatment is given.

The subject receiving SB12 or Soliris® therapy may require dosing interval adjustment within the recommended  $14 \pm 2$  days dosing schedule during the maintenance period (up to every 12 days) when it is deemed necessary at the discretion of the Investigator; e.g., two consecutive events of elevated LDH  $\geq$  2 × ULN combined with sign or symptom of intravascular haemolysis after prior LDH reduction to < 1.5 × ULN on treatment. If a 12 or 13 day dosing interval conflicts with administrative schedules (e.g., holidays or weekends) but a shortened dosing interval is considered necessary for safety of subject, consultation with medical monitor (or Sponsor) is recommended. For subjects whose dosing interval is adjusted to 12 days in Period 1, it is recommended that the dosing interval be switched back to 14 days after switching IP at Week 26. Once the above event has occurred, the Investigator should inform the

medical monitor and/or Sponsor immediately.

In special circumstances of a shortage of the comparator, to ensure continuity of study treatment for the duration of study, the Sponsor will provide SB12 instead of Soliris<sup>®</sup> in a blinded manner. Rules for allocation of remaining comparators during the comparator shortage situation will be prespecified prior to execution of the potential change of IP assignment from Soliris<sup>®</sup> to SB12 in a blinded manner. This is to avoid the risk of unblinding and potential bias.

# 5.1.2. Assignment of Subjects to Treatment Sequence

Subjects who meet all criteria for enrolment will be randomly assigned to treatment sequence I (SB12 to Soliris®) or II (Soliris® to SB12). The randomisation numbers will be generated by the interactive web response system (IWRS) to ensure that treatment sequence assignment is unbiased and concealed from subjects, Investigators, and other study personnel. These randomisation numbers are linked to the each treatment sequence, which in turn are linked to IP kit numbers.

Subjects will not be stratified and the assigned randomisation numbers will not be re-used.

# 5.1.3. Blinding

This study is double-blinded. Subjects, Investigators, and other study personnel will remain blinded to the treatment sequence assignment throughout the study period after randomisation.

To ensure the blinding for the treatment sequence assignment, one carton will contain only one IP vial (SB12 or Soliris®). The carton and IP vial will be packed and labelled in identical appearance.

Emergency unblinding is referred to Section 8.5.

#### 5.2. Investigational Product

# 5.2.1. Identity of Investigational Product

The IPs will be supplied to investigational site in one carton containing a single vial. These IP vials will be packed and labelled in a double-blinded manner for clinical use.

The Investigator shall take responsibility for all steps to maintain appropriate records and ensure appropriate supply, storage, handling, distribution, and usage of IPs in accordance with the protocol and any applicable laws and regulations.

A detailed guidance for IP preparation, administration, storage, and destruction will be provided in the pharmacy manual.

Details of the IPs are provided in Table 3.

**Table 3. Investigational Products Description** 

| Active Pharmaceutical Ingredient: Eculizumab | | |
|---|---|--|
| SB12 | | |
| Formulation | Solutions for IV infusion | |
| Contents | One vial of 30 mL contains 300 mg of eculizumab (10 mg/mL) | |
| Storage conditions | Stored in a refrigerator (2-8°C), do not freeze | |
| | Stored in the original package in order to protect from light | |
| Soliris <sup>®</sup> | | |
| Formulation | Solutions for IV infusion |
|---|---|
| Contents | One vial of 30 mL contains 300 mg of eculizumab (10 mg/mL) |
| Storage conditions | Stored in a refrigerator (2-8°C), do not freeze<br>Stored in the original package in order to protect from light |

## 5.2.2. Formulation, Packaging, and Labelling

Eculizumab (SB12 or Soliris®) will be supplied for use as a concentrate for solution for infusion (300 mg per vial for SB12, Soliris®).

Packaging and labelling of SB12 or Soliris® will follow standard operating procedure (SOP) of the manufacturing site and regulatory requirements in each country, as well as will be in accordance with ICH-Good Clinical Practice (GCP). SB12 or Soliris® will be pre-packaged and labelled in a double-blinded form. The labels will contain the following information: The pharmaceutical dosage form, route of administration, identification number, the protocol number, use by date, storage details, and all other details required by local regulations and Good Manufacturing Practice (GMP).

# 5.2.3. Product Storage and Stability

SB12 and Soliris® should be stored at 2-8°C (36-46°F) in the original carton in order to protect from light. The temperature will be monitored properly during the study period. If continuous monitoring is not available then manual temperature logs should be generated and recorded to ensure proper storage conditions. If a temperature deviation occurred, responsible person should contact the Sponsor to determine if the drug is still appropriate for use. The IPs should be stored in a secure area, clearly labelled, and stored away from other IPs or medication to prevent confusion (for example, in a clearly marked box on a separate shelf of the refrigerator).

Do not freeze and do not shake SB12 or Soliris® vials. The IPs must not be used beyond the expiration date.

#### 5.2.4. Preparation and Administration of Investigational Products

When IPs arrive at investigational sites, responsible site staff should check the IPs for damage, quantity, integrity, and temperature conditions during shipment, and report any deviations or product complaints (PC) to the Sponsor according to written procedure.

Dilution should be performed in accordance with good practices rules, particularly for the respect of asepsis. Withdraw the total amount of SB12 or Soliris® from the vials using a sterile syringe. Transfer the recommended dose to an infusion bag. Dilute SB12 or Soliris® to a final concentration of 5 mg/mL by addition to the infusion bag using sodium chloride 9 mg/mL (0.9%) solution for injection, sodium chloride 4.5 mg/mL (0.45%) solution for injection, or 5% dextrose in water, as the diluent.

The final admixed SB12 or Soliris® 5 mg/mL infusion volume is 120 mL for 600 mg doses and 180 mL for 900 mg doses. The solution should be clear and colourless. Gently agitate the infusion bag containing the diluted solution to ensure thorough mixing of the product and diluent. Although the chemical and physical stability of the diluted solution has been demonstrated for 24 hours at 2-8°C (36-46°F), the medicinal product should be used immediately after dilution. If not used immediately, in-use storage times and conditions prior to use are the responsibility of the user and would normally not be longer than 24 hours at 2-8°C, unless dilution has taken place in controlled and validated aseptic conditions. The diluted solution should be allowed to warm to room temperature (18-25°C, 64-77°F) prior to administration by exposure to ambient air and must not be heated in a microwave or with any

heat source.

The pharmacist and/or designee are responsible for preparing infusion setting for IP administration. Prior to administration, the IPs should be visually inspected for particulate matter and discolouration and checked to ensure match between subject number and assigned treatment.

IP injection will be performed by the Investigator and/or designee according to delegation of study personnel for this study. Do not administer IPs as an IV push or bolus injection. The diluted solution of IPs should be administered by IV infusion over 25-45 minutes via gravity feed, a syringe-type pump, or an infusion pump. It is not necessary to protect the diluted solution of IPs from light during administration to the subject.

Subjects should be monitored and documented for at least one hour following completion of the infusion for signs or symptoms of an infusion reaction. If an adverse reaction occurs during the administration of IPs, the infusion may be slowed or stopped at the discretion of the Investigator. If the infusion is slowed, the total infusion time may not exceed 2 hours.

## 5.2.5. Treatment Compliance and Investigational Product Accountability

Compliance will be assessed by the subject's source documents and electronic case report form (eCRF). All dosing information including exact date and time of IV infusion should be recorded in the subject's source documents and eCRF.

Also any reason for non-compliance should be documented. For example, insufficient compliance is defined when a subject missing more than one IP for reasons other than toxicity, missed scheduled study activities.

IP accountability and dispensing records must be kept current and contain the following information:

- The identification of the subjects to whom the drug was dispensed
- The dates and quantity of the drug dispensed to the subject
- The dispensing and inventory logs must be available for inspection by the study monitor

The Investigator and/or designee is responsible for accounting all unused IP and all used IP containers. The Investigator uses this information to maintain an accurate and complete dispensing and inventory record provided by the Sponsor.

IP supplies are shipped to the investigational site as needed. The monitor will review drug accounting during routine monitoring visits with the documents containing relevant information provided by the Sponsor. At the completion or termination of the study, a final drug accountability review and reconciliation must be completed; any discrepancies must be investigated and their resolution must be documented.

To avoid accidental unblinding, used drug kits (empty vials, vials with residual materials, and cartons) should be promptly discarded after the infusion bag is prepared and in accordance with the local destruction SOP/policies for clinical study drugs. All unused IPs should be returned to the Sponsor or designated vendor unless local destruction site is approved by the Sponsor. If destruction is authorised at the investigational site, the Investigator must ensure that the materials are destroyed in compliance with all applicable environmental regulations, institutional policies, and any instructions provided by the Sponsor. Destruction of the IPs must be adequately documented.

#### **5.3.** Concomitant Medication or Treatment

All medication including both prescription and non-prescription drugs, and any procedures undertaken between 4 weeks prior to Screening (except for immunosuppressant) and EOS should be recorded in the subject's source documents and eCRF. This record will include all prescription drugs, herbal products, vitamins, minerals, over-the-counter medications, and current medications for PNH. Details to be recorded include: Name (generic name preferred), dose number and unit, frequency of administration, route of administration, start and stop dates, reason for administration, and the AE it relates to (if applicable).

Medication ended prior to the first IP administration will be reported as a prior medication and medication ended on or after IP administration will be reported as a concomitant medication. It is the responsibility of the Investigator to ensure that details regarding all medications are recorded in full in the subject's source documents and eCRF.

#### 5.3.1. Permitted Concomitant Medications or Treatment

The following concomitant medications are allowed if given on a stable dose (only for chronic administration) during the study period. However, for the subject's welfare, medications can be adjusted under discussion between the Investigator and medical monitor and/or Sponsor.

- Erythropoietin, systemic corticosteroids, low-molecular-weight heparins, iron supplements, and androgen therapy with a stable dose from at least 4 weeks prior to initiation of study drug (Day 1).
- Warfarin with a stable INR from at least 4 weeks prior to initiation of study drug (Day 1).
- Cyclosporine with a stable dose from at least 8 weeks prior to initiation of study drug (Day 1).

#### 5.3.2. Prohibited Concomitant Medications or Treatment

Immunosuppressant except for cyclosporine is prohibited during the study period from randomisation including but not limited to:

• Anti-thymocyte globulin (ATG), cyclophosphamide, etc.

Investigator should discuss with the medical monitor and/or Sponsor before using any other immunosuppressant.

## 6. Study Assessment

## 6.1. Efficacy Assessment

## 6.1.1. Disease-related Laboratory Parameters

Blood samples will be collected before IP administration at the visits specified in Table 1 and Table 2. Blood samples for the parameters will be analysed in central laboratory. Laboratory reports will be available to the Investigator in a timely manner. The parameters include PNH clone size of RBC and WBC evaluated by high-sensitivity flow cytometry, LDH, reticulocyte count, haptoglobin, and free haemoglobin.

If the LDH level is not changed after the initiation of study drug (lack of efficacy), the Investigator and medical monitor and/or Sponsor should discuss to determine how to manage this case including whether or not to perform pharmacogenetic analysis (C5 gene polymorphism).

Detail instructions of collection, processing, labelling, storage, and shipment for blood samples will be Samsung Bioepis – * Information* 

provided in the laboratory manual.

## 6.1.2. Breakthrough Haemolysis

The Investigator and/or designee will record the breakthrough haemolysis in the source documents and eCRF during the study period.

The breakthrough haemolysis is defined as  $\geq 1$  new or worsening sign or symptom of intravascular haemolysis (fatigue, haemoglobinuria, abdominal pain, chest pain, shortness of breath, dysphagia, erectile dysfunction, anaemia [haemoglobin < 10 g/dL], or major adverse vascular event [MAVE] including thrombosis) in the presence of elevated LDH  $\geq 2 \times$  ULN after prior LDH reduction to < 1.5  $\times$  ULN on treatment.

If a suspected sign or symptom of breakthrough haemolysis occurs, blood collection is required for evaluation of LDH, PK, and PD parameters by central laboratory. If necessary, an unscheduled visit should occur for evaluation of the subject and collection of the required LDH, PK, and PD parameters. For purposes of confirming breakthrough haemolysis, assessment of LDH must be based on a central laboratory value.

#### 6.1.3. Transfusions

The subjects will receive pRBC transfusion in case the Investigator discovers a subject's haemoglobin warrants a transfusion;

- Haemoglobin value  $\leq 9$  g/dL with signs or symptoms, or
- Haemoglobin value  $\leq 7$  g/dL regardless of signs or symptoms

It is recommended that the transfusion would be performed within 48 hours of the haemoglobin assessment. The decision to give a transfusion may be based on either local or central laboratory haemoglobin values.

Transfusion record will be collected from the signing of the informed consent until EOS. Anaemia-related signs or symptoms, haemoglobin value, number of units of pRBCs will be documented on the source documents and eCRF.

## 6.1.4. Major Adverse Vascular Events

The description of MAVEs, anatomical site, method of diagnosis, date of diagnosis, and outcome will be recorded in the source documents and eCRF as AEs during the study period.

The MAVE is defined as following;

Thrombophlebitis/deep vein thrombosis, pulmonary embolus, cerebral arterial/venous
occlusion, myocardial infarction, transient ischemic attack, unstable angina, renal vein
thrombosis, mesenteric vein thrombosis, portal vein thrombosis (Budd-Chiari syndrome),
acute mesenteric ischaemia, etc.

## 6.1.5. Paroxysmal Nocturnal Haemoglobinuria-related Symptoms

The PNH-related symptom questionnaire will be completed by subjects. The questionnaire should be completed by subjects before IP administration at the visits specified in Table 1 and Table 2; at Screening, Weeks 0 (Day 1), 4, 14, 26, 30, 40, and 52.

The symptoms in the past 7 days will be rated by severity. The questionnaire is provided in APPENDIX A. Investigator and/or designee will record the presence or absence of the following signs and symptoms

#### of PNH;

• Fatigue, haemoglobinuria (discolouration of urine), chest pain, abdominal pain, dyspnoea (shortness of breath), dysphagia, and erectile dysfunction

## **6.2. Safety Assessment**

#### **6.2.1.** Adverse Events

All AEs will be recorded according to Section 8.

#### **6.2.2.** Clinical Laboratory Evaluations

Blood and urine sampling for clinical laboratory tests will be collected before IP administration at the visits specified in Table 1 and Table 2.

Blood and urine samples will be analysed in central laboratory except urine pregnancy test which will be performed at investigational site using centrally supplied pregnancy kit. A detailed process for clinical laboratory sampling, handling, storage, and shipping will be provided in the laboratory manual for safety lab testing. Laboratory reports will be available to the Investigator in a timely manner.

If laboratory tests are performed as per local practice and found to be abnormal, it is recommended that the Investigator uses their best clinical judgement to determine if the abnormal values would affect subjects' safety while participating in the study. It is highly recommended to test the abnormal parameter by central laboratory as well, if available.

During COVID-19 pandemic circumstances, it may be unable to get central laboratory values in time due to COVID-19 related restrictions. For those cases, local laboratory will be allowed in addition to central laboratory for scheduled visit after randomisation until COVID-19 restrictions are relieved under discussion with Sponsor.

The parameters for clinical laboratory tests are listed in the Table 4.

| Table 4. Parameters for Cl | inical Laboratory Tests | |
|---|---|---|
| Haematology | <ul> <li>WBC count</li> <li>RBC count</li> <li>Haemoglobin</li> <li>Haematocrit</li> <li>Platelet count</li> <li>Differential WBC count</li> <li>Nucleated RBC</li> </ul> | <ul> <li>Mean corpuscular haemoglobin (MCH)</li> <li>Mean corpuscular haemoglobin concentration (MCHC)</li> <li>Mean corpuscular volume (MCV)</li> <li>Mean platelet volume (MPV)</li> <li>Red cell distribution width (RDW)</li> </ul> |
| Chemistry | <ul> <li>Sodium</li> <li>Potassium</li> <li>Creatinine</li> <li>Blood urea nitrogen (BUN)</li> <li>Glucose</li> <li>Calcium</li> <li>Phosphorus</li> </ul> | <ul> <li>Total bilirubin</li> <li>Direct/indirect bilirubin</li> <li>Albumin</li> <li>Total protein</li> <li>Alanine aminotransferase (ALT)</li> <li>Aspartate aminotransferase (AST)</li> <li>Alkaline phosphatase (ALP)</li> <li>Gamma-glutamyl transpeptidase</li> </ul> |
| Coagulation Profile | <ul><li>Prothrombin time</li><li>Partial thromboplastin time</li><li>INR</li></ul> | |
| Urinalysis | <ul> <li>Protein</li> <li>Blood</li> <li>Leukocyte esterase</li> <li>Nitrate</li> <li>Ketone</li> <li>Glucose</li> <li>Ferritin</li> </ul> | <ul> <li>pH</li> <li>Specific gravity</li> <li>Bilirubin</li> <li>Urobilinogen</li> <li>Appearance</li> <li>Colour</li> <li>Serology (HIV-1 and HIV-2)</li> </ul> |
| Others | <ul> <li>Vitamin B<sub>12</sub></li> <li>Folate</li> </ul> | <ul> <li>Pregnancy test (serum or urine)<sup>1</sup></li> <li>Serum follicle stimulating hormone (FSH)<sup>2</sup></li> </ul> |

<sup>&</sup>lt;sup>1</sup> Pregnancy test will be performed for women of childbearing potential (serum or urine). Serum pregnancy test will be performed at Screening and 8 weeks after the last dose of study drug in case of ET and urine pregnancy test will be performed at other applicable visits before study drug administration.

The Investigator will check any laboratory values which have potential significance in subject's safety during the study period. The Investigator will also evaluate any change in laboratory values. Each out

<sup>&</sup>lt;sup>2</sup> Serum FSH levels will be measured at Screening and Week 26 in order to confirm postmenopausal status only for women who present natural (spontaneous) amenorrhea for at least 12 months prior to Screening regardless of the subjects' age.

of range result should be assessed as not clinically significant or clinically significant by the Investigator. All laboratory abnormalities that require intervention (i.e., IP temporary discontinuation, IP discontinuation, concomitant medication, etc.) should be assessed as clinically significant and the clinically significant abnormalities should be recorded as AEs (see Section 8.1).

## 6.2.3. Physical Examinations

Physical examination including height and weight will be performed at Screening and physical examination including weight before IP administration at the visits specified in Table 1 and Table 2.

Abnormal findings will be documented on the source documents and eCRF, and any clinically significant abnormality or worsening of a previously noted abnormality should be recorded as an AE (see Section 8.1).

## **6.2.4.** Twelve-lead Electrocardiograms

Twelve-lead ECG measurements will be performed before IP administration at the visits specified in Table 1 and Table 2.

## 6.2.5. Vital Signs

Vital signs (blood pressure, heart rate, and body temperature) will be assessed at the visits specified in Table 1 and Table 2. When vital signs are scheduled to be assessed at the same time point with blood sampling, it is recommended that the vital signs should be measured prior to the blood collection being performed.

The Investigator should assess all vital signs before IP administration on dosing days and any clinically significant abnormalities should be recorded as AEs (see Section 8.1).

#### **6.3. Other Assessments**

#### 6.3.1. Pharmacokinetic Assessments

Blood sampling for PK analysis will be performed in all randomised subjects before IP administration at the visits specified in Table 1 and Table 2. Blood samples should be collected at the same day of study drug administration. Subjects' samples may be used for PK analysis method development and/or method validation.

If the IP administration is delayed for any reasons after blood sample for PK is collected, blood sample for PK analysis should be repeated on actual dosing day and be used for analysis.

In all cases, the exact date and time of the PK sampling and IP administration must be carefully recorded in the source documents and eCRF. Detail instructions of handling, storage, and shipment for PK samples are described in the laboratory manual.

The Sponsor or its designated representative will store PK samples after the end of the clinical study for maximum 15 years in order to have the possibility to repeat the assay already performed (e.g., reanalysis requested by regulatory authorities or failure of first analysis [see Section 10.4]).

## **6.3.2.** Immunogenicity Assessments

The purpose of immunogenicity assay is to determine whether ADAs and NAbs against SB12 or Soliris® occur in similar rate and influence the safety or efficacy. Blood sampling for immunogenicity assay will be done before IP administration at the visits specified in Table 1 and Table 2. Blood samples should be collected at the same day of study drug administration. Subjects' samples may be used for immunogenicity testing assay method development and/or method validation.

Samsung Bioepis -  Information

If the IP administration is delayed for any reasons after blood sample for immunogenicity is collected, blood sample for immunogenicity assay should be repeated on actual dosing day and be used for analysis.

In all cases, the exact date and time of the ADAs and NAbs sampling and IP administration must be carefully recorded in the source documents and eCRF. Detail instructions of handling, storage, and shipment for immunogenicity samples are described in the laboratory manual.

The Sponsor or its designated representative will store immunogenicity samples after the end of the clinical study for maximum 15 years in order to have the possibility to repeat the assay already performed (e.g., re-analysis requested by regulatory authorities or failure of first analysis [see Section 10.4]).

## 6.3.3. Pharmacodynamic Assessments

Blood samples for PD analysis will be collected at prior to infusion before IP administration at the visits specified in Table 1 and Table 2. Blood samples should be collected at the same day of study drug administration. Subjects' samples may be used for PD analysis method development and/or method validation.

Complement activity will be measured within the secured sample stability period by the validated method by the Sponsor or its designated representative.

If the IP administration is delayed for any reasons after blood sample for PD is collected, blood sample for PD analysis should be repeated on actual dosing day and be used for analysis.

In all cases, the exact date and time of the PD sampling and IP administration must be carefully recorded in the source documents and eCRF. Detail instructions of handling, storage, and shipment for PD samples are described in the laboratory manual.

The Sponsor or its designated representative will store PD samples after the end of the clinical study for maximum 15 years in order to have the possibility to repeat the assay already performed (e.g., reanalysis requested by regulatory authorities or failure of first analysis [see Section 10.4]).

#### **6.3.4. Pharmacogenetic Assessments**

Blood sample will be collected for pharmacogenetic analysis, ideally on Day 1 before initiation of study drug, or at the next scheduled blood sampling.

Genetic variants in C5 is associated with poor response to eculizumab since C5 mutation causes the structural change in binding site of eculizumab, resulting in less suppression of complement-mediated haemolysis. These blood samples can be used for extraction and analysis of DNA in order to investigate the mutational status of the subjects including, but not limited to C5. The analysis will be performed during or after the study for subjects who present poor response to study drug, or only if scientifically appropriate and data required.

The exact date and time of blood sampling for pharmacogenetic analysis must be recorded in the source documents and eCRF. Detail instructions of handling, storage, and shipment for pharmacogenetic samples are described in the laboratory manual.

The Sponsor or its designated representative will store pharmacogenetic samples after the end of the clinical study for maximum 15 years in order to have the possibility to repeat the assay already performed (e.g., re-analysis requested by regulatory authorities or failure of first analysis [see Section 10.4]).

# 7. Study Procedures

## 7.1. Study Flow and Visit Schedule

During this study, efficacy, safety, PK, immunogenicity, and PD assessments will be performed. The complete schedule of activities is outlined in Table 1 and Table 2.

## 7.1.1. Screening Period

## 7.1.1.1. Screening Visit (D-63 to D-22)

Screening should be performed within 42 days before randomisation. All subjects must provide written informed consent prior to any study related procedures being performed.

An eligibility screening form (ESF) documenting the subject's fulfilment of the entry criteria is to be completed by the Investigator or designee for all individuals considered for the study and subsequently included or excluded from the study. ESF should be reviewed by study monitor and submitted to medical monitor to determine the eligibility. Subjects who are confirmed to meet all criteria for enrolment will be randomly assigned in a 1:1 ratio to receive SB12 or Soliris<sup>®</sup>. Subjects who are considered for study entry but fail to meet the eligibility requirements should also have an ESF completed with the reason for lack of eligibility included, since this provides information on the selected study population. All ESFs should be kept in the study files at the investigational sites.

The following procedures and assessments should be performed within 42 days before randomisation. Retesting or re-evaluation is allowed within the screening period, but the latest result will be used to determine the eligibility.

- Written informed consent
- Demographic data
- Review of medical history including clinically significant diseases especially related to eligibility criteria (see Section 4.3), surgical procedures, and thrombosis history
- Review of transfusion history (anaemia-related signs or symptoms which precipitated transfusion, haemoglobin level before transfusion, number of units of pRBCs, date of transfusion, if available) within 12 months prior to Screening
- Physical examination (including height and body weight)
- Vital signs (blood pressure, heart rate, and body temperature)
- Twelve-lead ECG
- FSH test (serum) for women with at least 12 months natural (spontaneous) amenorrhea prior to Screening.
- Pregnancy test (serum) for women of childbearing potential. Female subjects of nonchildbearing potential are defined as:
  - a. At least 12 months natural amenorrhea and FSH > 40 U/L confirmed by serum blood test OR
  - b. Those with history of hysterectomy, ligation of both fallopian tubes, surgical removal of both ovaries, or appropriate sterilisation operation. Documentation of surgical procedure

performed at least 90 days prior to Screening or appropriate medical documentation is required for confirmation of surgical sterilisation.

- Review of laboratory results
  - Disease-related laboratory parameters: PNH clone size of RBC and WBC evaluated by high-sensitivity flow cytometry, LDH, reticulocyte count, haptoglobin, and free haemoglobin
  - Haematology: Haemoglobin, haematocrit, RBC count, total WBC count including differential count, platelet count, nucleated RBC, MCH, MCHC, MCV, MPV and RDW
    - ✓ <u>Note</u>: If concurrent bone marrow failure is suspected, bone marrow examination is highly recommended to rule out the combined disease (e.g., myelodysplastic syndrome, severe aplastic anaemia, etc.).
  - Chemistry: Sodium, potassium, serum creatinine, BUN, glucose, calcium, phosphorus, total bilirubin, direct/indirect bilirubin, albumin, total protein, ALT, AST, ALP, and gamma-glutamyl transpeptidase
  - Coagulation profile: Prothrombin time, partial thromboplastin time, and INR
  - Urinalysis: Protein, blood, leukocyte esterase, nitrite, ketone, glucose, pH, specific gravity, bilirubin, urobilinogen, appearance, and colour (if urinalysis result is abnormal, urine microscopic examination will be performed)
  - Serology: HIV-1 and HIV-2
  - Others: Ferritin, vitamin B<sub>12</sub>, and folate
- PNH symptomatology will be assessed.
- AEs assessment
- Review of previous medication (within 4 weeks prior to Screening except immunosuppressant, which will be assessed for 8 weeks prior to Screening)
- Review of MAVEs
- Evaluate subject compliance with all eligibility criteria

## 7.1.1.2. Vaccination for *Neisseria meningitidis*

Due to its mechanism of action, the use of SB12 or Soliris<sup>®</sup> increases the subject's susceptibility to meningococcal infection (*Neisseria meningitidis*). Meningococcal disease due to any serogroup may occur.

To reduce the risk of meningococcal infection, all subjects must be vaccinated against *Neisseria meningitidis* prior to or on Day 1 in accordance with current local guidelines or Soliris® SmPC. Vaccines against serogroups A, C, Y, W135, and B where available, are recommended in preventing the commonly pathogenic meningococcal serogroups. In case subjects were vaccinated against meningococcal infection within 3 years prior to Day 1, which is properly documented, vaccination for this study could be omitted. For the information including formulation, preparation, and storage of vaccine, refer to the prescribing information in SmPC of vaccine. Subjects must be revaccinated later during the study if local guidelines indicate to do so.

Subjects who initiate SB12 or Soliris<sup>®</sup> treatment less than 14 days after receiving a meningococcal vaccine must receive treatment with appropriate prophylactic antibiotics until 14 days after vaccination. Vaccination for *Neisseria meningitidis* and the prophylactic antibiotics should be recorded in the source documents and eCRF. As vaccination might not be sufficient to prevent meningococcal infection, appropriate use of antibiotics may be considered according to the current local guidelines and/or at the discretion of the Investigator.

As vaccination may further activate complement, subjects with PNH may experience increased signs and/or symptoms of their underlying disease, such as haemolysis. Therefore, subjects should be closely monitored for disease symptoms after vaccination.

To raise risk awareness of meningococcal infection and its signs and/or symptoms, subjects will be given the safety card to carry with them during the study period.

The safety card will contain following:

- Signs and symptoms of infection and sepsis
- Warning to seek immediate medical care if signs and/or symptoms of meningococcal infection are present
- Statement that the patient is receiving eculizumab
- Contact details where a health care practitioner can receive further information

#### 7.1.2. Randomisation

Investigator should check the whole eligibility criteria of the subjects based on the laboratory report, medical history, and subjects' assessment. After a subject's eligibility is confirmed by the Investigator and medical monitor, subject should be randomised to either treatment sequence through an IWRS.

Once the subject is confirmed eligible for the study, the subject will be advised on study restrictions such as contraception, prohibited medications, and other study requirements if any.

During COVID-19 pandemic circumstances, Day 1 (1st dosing) may not be started within 21 days of randomisation due to unexpected COVID-19 related restrictions. In such cases, the subject will be monitored for safety per Investigator's discretion. Day 1 will be started after the COVID-19 related restrictions are relieved.

#### 7.1.3. Treatment Period

The Investigator should check if the subject does not meet the discontinuation criteria before the initiation of study drug at Day 1.

All procedures and assessments will be performed at the visits specified in Table 1 and Table 2, and before IP administration on same day or up to 2 days prior, unless otherwise specified.

Laboratory assessments will be performed at central laboratory. Detail instructions of collecting, processing, storing, and shipping for blood samples are described in the laboratory manual. Laboratory reports will be available to the Investigator in a timely manner for clinical management of subjects during treatment period.

The Investigator will evaluate the assessment results and manage subjects based on the medicinal judgement and/or knowledge.

In special circumstances of a shortage of the comparator, to ensure continuity of study treatment for the duration of study, the Sponsor will provide SB12 instead of Soliris® in a blinded manner. Investigators and subjects will be informed prior to the execution of the potential change of IP assignment. Subjects willing to continue the study treatment after knowing that they may receive SB12 instead of Soliris® in a blinded manner during the study, should have their agreement both documented in the source document and an ICF. If the Investigators or subjects do not agree to the potential change of IP assignment, then subjects may withdraw from the study and be closely monitored for at least 8 weeks after last dose of study drug.

## 7.1.3.1. Treatment Period 1 (before Cross-over)

- Blood sampling for pharmacogenetic analysis (C5 gene polymorphism) will be performed at Week 0 (Day 1). If missing, it would be taken at the next scheduled blood sampling time.
- Physical examination (including body weight) will be performed at each scheduled visit.
- Vital signs (blood pressure, heart rate, and body temperature) will be checked at each scheduled visit.
- Twelve-lead ECG will be performed at Week 14.
- Pregnancy test (urine) will be performed at the visits specified in Table 1 for women of childbearing potential only.
- Clinical laboratory tests including haematology, chemistry (includes or does not include ferritin, vitamin B<sub>12</sub>, and folate), coagulation profile, and urinalysis will be performed at the visits specified in Table 1.
- Blood sample collection for disease-related laboratory parameters will be performed at the visits specified in Table 1.
- Blood sample collection for PK analysis will be performed at pre-dose of Week 0 (Day 1), Week 2, Week 4, Week 6, Week 10, Week 14, Week 18, and Week 22.
- Blood sample collection for immunogenicity assay will be performed at pre-dose of Week 0 (Day 1), Week 2, Week 4, Week 6, Week 10, Week 14, Week 18, and Week 22.
- Blood sample collection for PD analysis will be performed at pre-dose of Week 0 (Day 1), Week 2, Week 4, Week 6, Week 10, and Week 14.
- PNH symptomatology will be assessed at the visits specified in Table 1.
- AEs, concomitant medications, MAVEs, and transfusion record will be assessed and recorded.

## IP administration

• IP administrations by IV infusion for 35 ± 10 minutes (600 mg every week for first 4 weeks and 900 mg for the fifth week, followed by 900 mg every 2 weeks, the visit window allowed for each visit is ± 2 days)

## 7.1.3.2. Visit 16 (Week 26/Day 183)

Each subject will cross-over from the treatment initially assigned to another treatment at Visit 16 (Week 26) and IPs will be given until Visit 28 (Week 50).

- Physical examination (including body weight)
- Vital signs (blood pressure, heart rate, and body temperature)
   Samsung Bioepis  Information

- Twelve-lead ECG
- FSH test (serum) for women with at least 12 months natural (spontaneous) amenorrhea prior to Screening.
- Pregnancy test (urine) for women of childbearing potential only.
- Clinical laboratory tests including haematology, chemistry (includes ferritin, vitamin B<sub>12</sub>, and folate), coagulation profile, and urinalysis.
- Blood sample collection for disease-related laboratory parameters.
- Blood sample collection for PK analysis will be performed at pre-dose.
- Blood sample collection for immunogenicity assay will be performed at pre-dose.
- Blood sample collection for PD analysis will be performed at pre-dose.
- PNH symptomatology will be assessed.
- AEs, concomitant medications, MAVEs, and transfusion record will be assessed and recorded.

## IP administration

• IP administration by IV infusion for  $35 \pm 10$  minutes (900 mg)

#### 7.1.3.3. Treatment Period 2 (after Cross-over)

- Physical examination (including body weight) will be performed at each scheduled visit.
- Vital signs (blood pressure, heart rate, and body temperature) will be checked at each scheduled visit.
- Twelve-lead ECG will be performed at Week 40 and Week 52.
- Pregnancy test (urine) will be performed at the visits specified in Table 2 for women of childbearing potential only.
- Clinical laboratory tests including haematology, chemistry (includes or does not include ferritin, vitamin B<sub>12</sub>, and folate), coagulation profile, and urinalysis will be performed at the visits specified in Table 2.
- Blood sample collection for disease-related laboratory parameters will be performed at the visits specified in Table 2.
- Blood sample collection for PK analysis will be performed at pre-dose of Week 28, Week 30, Week 32, Week 36, Week 40, Week 44, Week 48, and Week 52.
- Blood sample collection for immunogenicity assay will be performed at pre-dose of Week 28, Week 30, Week 32, Week 36, Week 40, Week 44, Week 48, and Week 52.
- Blood sample collection for PD analysis will be performed at pre-dose of Week 28, Week 30, Week 32, Week 36, Week 40, and Week 52.
- PNH symptomatology will be assessed at the visits specified in Table 2.
- AEs, concomitant medications, MAVEs, and transfusion record will be assessed and recorded.

#### IP administration

• IP administrations by IV infusion for  $35 \pm 10$  minutes (900 mg every  $14 \pm 2$  days)

# 7.1.3.4. Safety Follow-up (Week 58/Day 407)

Safety follow-up will be done at Week 58 ( $\pm$  7 days) which is 8 weeks after the last dose of SB12 or Soliris® for subjects who complete the study treatments until Week 50, regardless whether subject receives extended supply of SB12 or not to ensure subject's safety. These activities will be conducted either by visit or by phone call based on subjects' preference.

AEs, concomitant medications, MAVEs, and transfusion record will be assessed and recorded.

#### 7.1.3.5. Early Termination Visit

ET visit is defined as 8 weeks ( $\pm$  7 days) after the last dose of SB12 or Soliris<sup>®</sup> during the treatment period.

- Physical examination (including body weight)
- Vital signs (blood pressure, heart rate, and body temperature)
- Pregnancy test (serum) for women of childbearing potential only.
- Clinical laboratory tests including haematology, chemistry, and urinalysis
- Blood sample collection for disease-related laboratory parameters
- Blood sample collection for immunogenicity assay
- AEs, concomitant medications, MAVEs, and transfusion record will be assessed and recorded.

#### 7.1.4. Unscheduled Visits

If a sign or symptom of breakthrough haemolysis is suspected, an unscheduled visit should be occurred and samples should be collected for LDH, PK, and PD assessment for central laboratory at that time. Additionally, other unscheduled visits are permitted at the discretion of the Investigator. Any tests, procedures, or assessments performed at the unscheduled visits must be recorded in the source documents and eCRF.

#### 7.2. Discontinuation

## 7.2.1. Subject Discontinuation from Study Treatment

The study treatment must be discontinued for a subject in the event of the following:

- Consent withdrawal by subject
  - Subjects may withdraw from the study or study specific procedures at any time for any reason during the entire duration of the study without prejudicing future treatment.
  - If subjects withdraw his/her consent, the Investigator must inquire the reasons for consent withdrawal as to whether it is related to the study (e.g., documented lack of efficacy, AE, or pregnancy); however, the subject could refuse to provide such reason.
  - If the main reason for consent withdrawal is considered related to the study, the Investigator may select appropriate reason among the reasons listed below other than consent withdrawal.
- Pregnancy (study treatment should be immediately stopped when a pregnancy is made known

and the pregnant woman will be removed from the study)

- Unblinding the study treatment to the Investigator or subject (i.e., breaking the double-blind).
- Other complement inhibitor use

The Investigator should discuss with the medical monitor prior to discontinuing a subject's study treatment in case of the following criteria, but not limited to:

- Conditions or intercurrent illness that preclude compliance with the protocol in terms of their safety or well-being
- Lack of efficacy (e.g., C5 gene polymorphism)

<u>Note</u>: If the LDH level is not changed after the initiation of study drug (lack of efficacy), the Investigator and medical monitor and/or Sponsor should discuss to determine how to manage this case including whether or not to perform pharmacogenetic analysis (C5 gene polymorphism).

- Unacceptable toxicity including meningococcal infection or anaphylaxis
- Serious protocol deviations (PDs) including lack of subject's compliance (e.g., repeated delay in study treatment and lost to follow-up) that preclude continuation of the study

<u>Note</u>: Before a subject is deemed lost to follow-up, the Investigator or designee will make every effort to regain contact with the subject.

• Investigator discretion or other reasons

Discontinuation from study treatment does not mean immediate discontinuation from the study, and remaining study procedures should be completed as indicated by the study protocol. Subjects who discontinue from the study at any time post-Day 1 (after the initiation of study drug) before completion of last study treatment at Week 50 will be required to have an ET visit. The data to be collected at the 8 weeks after the last dose of study drug are described in the Section 7.1.3.5. Every effort will be employed to keep subjects who discontinued from study treatment to undertake the scheduled ET visit procedures.

Subjects who discontinue study treatment after being exposed to study treatment will be monitored closely for signs of a potentially life-threatening haemolytic breakthrough event. Serious haemolysis is identified by serum LDH levels greater than the pre-treatment level, along with any of the following:

- Greater than 25% absolute decrease in PNH clone size (in the absence of dilution due to transfusion) in 1 week or less
- A haemoglobin level of < 5 g/dL or a decrease of > 4 g/dL in 1 week or less
- Angina
- Change in mental status
- A 50% increase in serum creatinine level
- Thrombosis as defined by MAVEs

Any subject who discontinues SB12 or Soliris® should be monitored for at least 8 weeks after last dose of study drug to detect serious haemolysis and other reactions. If serious haemolysis occurs after SB12 or Soliris® discontinuation, consider the following procedures and/or treatments:

- Blood transfusion (pRBCs) or exchange transfusion if the PNH RBCs are > 50% of the total RBCs by flow cytometry
- Anticoagulation
- Corticosteroids
- Complement inhibitors

## 7.2.2. Investigational Site Discontinuation

Investigational site participation may be discontinued if the Sponsor, the Investigator, or the Institutional Review Board (IRB)/Independent Ethics Committee (IEC) of the investigational site judge it necessary for any reason. Health authorities and IRB/IEC will be informed about the discontinuation of the study in accordance with applicable regulations.

# 7.3. Early Termination of the Study

The study can be terminated at any time for medical or ethical reasons by the Sponsor. If the study is terminated or discontinued prematurely, the Sponsor will promptly notify to the Investigator. Investigator may be informed of additional procedures to be followed in order to assure that adequate consideration is given to the protection of the subject's interests.

Health authorities and IRB/IEC will be informed about the discontinuation of the study in accordance with applicable regulations.

# 8. Safety Monitoring and Reporting

#### 8.1. Adverse Events

#### 8.1.1. Definition of Adverse Event

An AE is any untoward medical occurrence in a patient or clinical investigation subject administered the medicinal (investigational) product or other protocol-imposed intervention and which does not necessarily have to have a causal relationship with this treatment or intervention. An AE can therefore be an unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of any dose of a medicinal (investigational) product or other protocol-imposed intervention regardless of attribution.

All AEs during the period of observation (as specified in Section 8.1.2) including the events that occurred prior to administration of an IP should be reported as an AE.

Pre-existing conditions and any abnormal findings from assessments during the screening period which are not related to protocol-imposed intervention should not be reported as AEs; however, pre-existing conditions which worsen (i.e., increase in severity) that meet the definition of an AE during the study are to be reported as AEs.

Diagnostic and therapeutic non-invasive and invasive procedures, such as surgery, should not be reported as AEs. However, the medical condition for which the procedure was performed should be reported if it meets the definition of an AE. For example, an acute appendicitis that begins during the AE reporting period should be reported as an AE and the resulting appendectomy should be recorded as treatment of the AE.

The AEs that emerge during treatment with an IP (i.e., treatment-emergent AE [TEAE]) will be analysed for the purposes of safety analyses.

## **8.1.1.1.** Clinically Significant Abnormality

If there are any abnormalities discovered during the laboratory tests, physical examinations, vital signs, and/or other safety assessments and the abnormality is assessed clinically significant by the Investigator, it should be reported as an AE. This does not apply to pre-existing conditions which have been documented at Screening or if the abnormality is consistent with a current diagnosis (underlying disease or other AEs). If it is not specified or defined elsewhere in the protocol, clinically significant abnormality may include the events that led to an intervention, including withdrawal of the IP treatment, significant additional concomitant medication, and others evaluated as clinically significant by the Investigator.

If the clinically significant laboratory or other abnormality from safety assessment is not a sign of a disease or syndrome, the abnormality itself should be reported as an AE. If the abnormality can be characterised by a precise clinical term, the clinical term should be reported as the AE. For example, an elevated serum potassium level of 7.0 mEq/L should be reported as 'hyperkalaemia'. Observations of the same clinically significant abnormality from visit to visit should not be repeatedly reported as AEs, unless their severity, seriousness, or aetiology changes.

#### 8.1.2. Period of Observation for Adverse Events

AEs will be reported from the time of signing the ICF until EOS.

SAEs must be reported to the Sponsor or its designated representative according to Section 8.2.2.

Unresolved AEs during the study period should be followed up until EOS. The Investigator should observe the AEs for appropriate medical care of the subject until AE resolution or stabilisation.

If the subject has an ongoing SAE at EOS, these cases will be followed until event resolution or stabilisation (see Section 8.2.2).

#### 8.1.3. Reporting Adverse Events

AEs are to be reported in the eCRF and reviewed by the Investigator. When reporting an AE, a diagnosis (when possible and appropriate) rather than each individual sign and symptom should be reported.

Each AE is to be assessed to determine if it meets the criteria of an SAE (see Section 8.2.1 for SAE definition). If an AE is classified as a SAE, it must be reported to the Sponsor, or its designated representative, promptly according to the timeline specified in Section 8.2.2. For an SAE, a diagnosis with a description of signs and symptoms as well as other supporting information that led to the diagnosis should be described in the SAE form provided by the Sponsor (see Section 8.2.2).

#### 8.1.4. Severity Assessment

The Investigator is responsible for assessing and reporting the severity of AEs in accordance with National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0.

The following general guideline can be used to describe the severity of the AE. A grading (severity) scale for each specific AE is provided in NCI-CTCAE v5.0.

Table 5. Severity Grade of NCI-CTCAE v5.0

| Grade | Clinical Description of Severity |
|---|---|
| Grade 1 | Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. |

| Grade | Clinical Description of Severity |
|---|---|
| Grade 2 | Moderate; minimal, local or non-invasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL) <sup>a</sup> . |
| Grade 3 | Severe or medically significant but not immediately life-threatening; hospitalisation or prolongation of hospitalisation indicated; disabling; limiting self-care ADL <sup>b</sup> . |
| Grade 4 | Life-threatening consequences; urgent intervention indicated. |
| Grade 5 | Death related to AE. |

<sup>&</sup>lt;sup>a</sup> Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.

## 8.1.5. Causality Assessment

The Investigator is responsible for assigning a causal relationship to each AE. The causal relationship between the IP and the AE should be defined as not related (no) or related (yes).

Events should be classified as 'related' if there is a reasonable possibility that the IP caused the AE. This means that there are facts (evidence) or arguments to suggest a causal relationship.

Events should be classified as 'not related' if there is no reasonable possibility that the IP caused the AE.

#### 8.1.6. Expectedness Assessment

Expectedness of AEs will be assessed by reference safety information (RSI) in IB. More detailed information on expectedness assessment will be explained in IB. The latest Soliris® SmPC [10] will be used to assess the expectedness for the reference product after database lock or emergency unblinding.

#### 8.1.7. Withdrawal due to Adverse Events

Subject withdrawal from the study due to an AE should be distinguished from withdrawal due to personal reasons and recorded in the source documents and appropriate eCRF section. Subjects withdrawn due to an AE should be followed up until the time point specified in Section 7.2.1. When a subject withdraws from the study due to an SAE, the SAE must be reported and followed in accordance with the requirements outlined in Section 8.2.2.

Subjects who discontinue the administration of IPs because of serious or significant safety issues should be followed closely until the events are fully and permanently resolved or stabilised.

#### 8.2. Serious Adverse Events

#### 8.2.1. Definition of Serious Adverse Event

An SAE is any untoward medical occurrence at any dose that:

- Results in death,
- Is life-threatening,
- Requires inpatient hospitalisation or prolongation of existing hospitalisation,

<sup>&</sup>lt;sup>b</sup> Self-care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden

- Results in persistent or significant disability/incapacity,
- Results in congenital anomaly/birth defects,
- Is medically important.

Medical and scientific judgement should be exercised in deciding whether expedited reporting is appropriate in other situations, such as important medical events that may not be immediately life-threatening or result in death or hospitalisation. However, if it is determined that the event may jeopardise the subject and may require intervention to prevent one of the other outcomes listed in the definition above, the important medical event should be reported as serious. Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalisation or development of drug dependency or drug abuse.

The term 'severe' is often used to describe the intensity (severity) of a specific event (as in mild, moderate, or severe myocardial infarction); the event itself, however, may be of relatively minor medical significance (such as severe headache). This is not the same as 'serious,' which is based on subject/event outcome or action criteria usually associated with events that pose a threat to a subject's life or functioning.

## 8.2.1.1. Life-threatening

The term 'life-threatening' in the definition of 'serious' refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe.

## 8.2.1.2. Hospitalisation

AEs reported from clinical studies associated with inpatient hospitalisation or prolongations of hospitalisation are considered serious. Staying at an observation unit in the emergency room for more than 24 hours qualifies for hospitalisation. Any events leading to subsequent emergency room visit for less than 24 hours should be in the discretion of the Investigator to assess serious as medically important.

Hospitalisation or prolongation of hospitalisation in the absence of a precipitating clinical AE is not in itself an SAE. Examples include:

- Admission for treatment of a pre-existing condition not associated with the development of a new AE or with a worsening of the pre-existing condition (e.g., for work-up of persistent pre-treatment lab abnormality),
- Social admission for convenience (e.g., admission of a subject who does not have a carer),
- Administrative admission (e.g., for a yearly physical exam),
- Protocol-specified admission during a clinical study (e.g., for a procedure required by the study protocol),
- Optional admission not associated with a precipitating clinical AE (e.g., for elective cosmetic surgery).

Pre-planned treatments or surgical procedures should be noted in the relevant source document for the individual subject.

## 8.2.2. Reporting Serious Adverse Events

SAEs must be collected until 8 weeks ( $\pm$  7 days) from the last dose of study drug (five half-lives of the study drug).

SAEs that occurred at or before EOS must be reported to the Sponsor or its designated representative via eCRF SAE report form at least within 24 hours of the Investigator becoming aware of the event.

SAEs that occurred after EOS must be reported to the Sponsor or its designated representative using the paper SAE report form at least within 24 hours of the Investigator becoming aware of the event.

Date and time (wherever possible) of the Investigator becoming aware of the SAE will be recorded in the SAE form and source document properly.

In particular, if the SAE is fatal or life-threatening, the Sponsor must be notified immediately, irrespective of the extent of available AE information. This timeframe also applies to additional (follow-up) information that becomes available on previously forwarded SAE reports. Sponsor will then follow expedited reporting procedures according to local and international regulations as appropriate.

The Investigator is obligated to pursue and provide information to the Sponsor on all SAEs in accordance with the timeframes for reporting specified above. In addition, an Investigator may be requested by the Sponsor to obtain specific additional follow-up information in an expedited fashion. In general, this will include a description of the SAE, which should be provided in sufficient detail so as to allow for a complete medical assessment of the case and independent determination of possible causality. Information on other possible causes of the event, such as concomitant medications and illnesses must be provided. In the case of a subject death, a summary of available autopsy findings must be submitted as soon as possible to the Sponsor or its designated representative.

All SAEs will be followed until event resolution or stabilisation (for chronic events), if possible, even when a subject is withdrawn from treatment. For chronic events that do not fully resolve until years later, the outcome should be reported as 'resolved with sequelae' as soon as the event has stabilised or returned to baseline. Follow-up information for the SAE should be actively sought and submitted as the information becomes available.

#### 8.3. Adverse Events of Special Interest

#### **8.3.1.** Meningococcal Infection

Due to its mechanism of action, the use of SB12 or Soliris® increases the subject's susceptibility to meningococcal infection (*Neisseria meningitidis*). These subjects might be at risk of disease by serogroups (particularly Y, W135, and X), although meningococcal disease due to any serogroup may occur. To reduce the risk of infection, all subjects will be vaccinated against *Neisseria meningitidis* prior to or on Day 1. Subjects must be revaccinated later during the study if local guidelines indicate to do so. However, vaccination may not be sufficient to prevent meningococcal infection. Consideration should be given to current local guidelines and/or the discretion of the Investigator on the appropriate use of antibacterial agents. Cases of serious or fatal meningococcal infections have been reported in Soliris®-treated patients. All subjects should be monitored for early signs of meningococcal infection, evaluated immediately if infection is suspected, and treated with appropriate antibiotics if necessary.

Subjects should immediately call the Investigator or seek emergency medical care, if subjects experience any of the following symptoms:

- Headache with nausea or vomiting
- Headache and a fever
- Headache with a stiff neck or stiff back
- Fever
- Fever and a rash
- Confusion
- Muscle aches with flu-like symptoms
- Eyes sensitive to light

Subjects should be informed of these signs and symptoms and steps taken to seek medical care immediately. Subjects who are undergoing treatment for serious meningococcal infections should discontinue SB12 or Soliris® treatment, and the Investigator must discuss the benefits and risks of SB12 or Soliris® treatment with subjects and provide them with medical instructions.

## **8.3.2.** Other Systemic Infections

SB12 or Soliris® blocks terminal complement activation; therefore subjects may have increased susceptibility to infections, especially with encapsulated bacteria. Serious infection with *Neisseria species* (other than *Neisseria meningitidis*), including disseminated gonococcal infections, have been reported after Soliris® treatment. Additionally, *Aspergillus* infections have occurred in immunocompromised and neutropenic patients. Subjects should immediately call the Investigator or seek emergency medical care, if subjects experience other systemic infections.

## 8.3.3. Infusion-related Reactions

Administration of SB12 or Soliris<sup>®</sup> may result in infusion reactions or immunogenicity that could cause allergic or hypersensitivity reactions (including anaphylaxis). In clinical trials, 1 (0.9%) gMG patient experienced an infusion reaction which required discontinuation of Soliris<sup>®</sup>. No PNH, aHUS, or NMOSD patients experienced an infusion reaction which required discontinuation of Soliris<sup>®</sup> in clinical trials.

Administration of SB12 or Soliris® should be performed in a setting with emergency equipment and site staff who are trained to medical emergencies.

If an infusion reaction occurs during the administration of IPs, the infusion may be slowed or stopped at the discretion of the Investigator. If the infusion is slowed, the total infusion time may not exceed 2 hours. The subject will be monitored until resolution of any observed symptoms. The majority of subjects will be resolved for symptoms and subsequently will receive further infusions. Subjects should be warned of the possibility of late onset reactions and should be instructed to contact their Investigator if these reactions occur. Subjects who experience infusion-related symptoms may be premedicated with paracetamol and antihistamines for subsequent infusions.

When a severe hypersensitivity reaction such as anaphylaxis occurs, the infusion should be interrupted immediately and supportive care including oxygen, epinephrine, beta-agonists, and corticosteroids should be administered with continuous vital sign monitoring by trained site staff until the symptoms are resolved.

#### 8.4. Pregnancy

Any pregnancy, including those of female partners of male subjects treated with the IP, should be reported to the Sponsor. If the female partner of a male subject becomes pregnant, a written consent must be obtained from the female partner before collecting any pregnancy-related information. All pregnancies associated with the subject, from the time the subject receives the first dose of study drug until 5 months after the last dose of study drug should be reported to the Sponsor. Pregnancy reports should be made within 24 hours of the Investigator becoming aware of the pregnancy using the "pregnancy notification and outcome report form".

Although pregnancy is not an AE, all pregnancies must be followed up until 6-8 weeks after the outcome of the pregnancy becomes available, unless the subject is lost to follow-up. The pregnancy outcome should be notified to the Sponsor by submitting a follow-up pregnancy notification and outcome report form. If the outcome of the pregnancy meets SAE criteria then the Investigator should report this case according to the SAE reporting process (Section 8.2.2).

## 8.4.1. Pregnancy Prevention

In order to minimise the risk to a foetus or embryo for including women of childbearing potential in this study, female subjects of childbearing potential and male subjects with female partner of childbearing potential must agree to use at least one highly effective birth control method. The Investigator and/or designee will discuss with the subject the need to use highly effective contraception consistently and correctly and document such conversation on the subject's source documents.

Highly effective birth control method includes the following:

- Combined (oestrogen and progesterone containing) hormonal contraception associated with inhibition of ovulation:
  - Oral, intravaginal, transdermal
- Progesterone-only hormonal contraception associated with inhibition of ovulation:
  - Oral, injectable, implantable
- Intrauterine device
- Intrauterine hormone-releasing system
- Bilateral tubal occlusion
- Vasectomised partner
- True abstinence

<u>Note:</u> True abstinence could be considered sufficient only for subjects who do not have a partner.

Followings are not highly effective birth control method and cannot be used for this study:

Progesterone-only oral hormonal contraception where inhibition of ovulation is not the
primary mode of action, male or female condom with or without spermicide,
cap/diaphragm/sponge with spermicide, periodic abstinence (calendar, symptothermal, postovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational

amenorrhoea method

## 8.5. Emergency Unblinding of Assigned Treatment

Unblinding should be considered only when knowledge of the treatment assignment is deemed essential for the subject's safety by their Investigator or a regulatory body. Emergency unblinding should be decided based on the medical decision by the Investigator considering subjects safety. In general, unblinding of subjects during the conduct of the clinical study should only be performed where there are compelling medical or safety reasons to do so. The responsibility to break the treatment code in emergency situations resides solely with the Investigator.

The IWRS will be used to break the blind and details on how to do this are provided in the IWRS manual. The Sponsor must be notified immediately after a subject and/or the Investigator is unblinded during the course of the study along with the reason for breaking the blind. Pertinent information regarding the circumstances of unblinding of a subject's treatment code must be documented on the subject's source documents. This includes who performed the unblinding, the subject(s) affected, the reason for the unblinding, the date of the unblinding, and the relevant IP information.

## 8.6. Independent Data and Safety Monitoring Board

An independent DSMB will be assigned for this study. The DSMB will consist of external experts (e.g., haematologists, clinical pharmacologists, and biostatisticians) and will review the safety and tolerability data from the study at pre-specified intervals. The details of the safety data and time points for review will be described in the DSMB charter and in the DSMB statistical analysis plan (SAP).

In addition, an ongoing blinded review of AEs, including clinical laboratory data will be regularly and continuously undertaken by the Sponsor medical monitor and pharmacovigilance team.

# 9. Statistical Methods and Data Analysis

Further information on the statistical methods for this study will be provided in the SAP, which will be finalised prior to the database lock for reporting the clinical study report (CSR).

Statistical analysis and reporting will be performed as follows:

#### • Interim safety analysis for independent DSMB meeting:

A DSMB SAP, describing the methodology and presentation of results and access to results will be prepared as a separate document. The safety reports for the DSMB data review meetings will be prepared according to the DSMB SAP.

The statistical analysis will be performed by an independent statistical reporting team and the results will be communicated to the DSMB directly by an independent unblind statistician.

#### • CSR:

The analysis will take place after the last subject completes the procedures at Week 58 or the corresponding visit. All study data will be analysed and reported for CSR.

## 9.1. Statistical Hypotheses

This is a cross-over study to demonstrate equivalence in terms of LDH between SB12 and Soliris<sup>®</sup>. The null hypothesis tested for the primary efficacy analysis is that either (1) SB12 is inferior to Soliris<sup>®</sup> or (2) SB12 is superior to Soliris<sup>®</sup> based on a pre-specified equivalence margin.

for those who are in favour of the time-adjusted AUEC of LDH, the treatment effect will be measured by time-adjusted AUEC of LDH between two different time points in each period, from Week 14 to Week 26 and from Week 40 to Week 52. The equivalence will be declared if the 90% confidence interval (CI) of the ratio between treatment effects is entirely contained within the pre-defined equivalence margin of [0.77, 1.29].

for those who are in favour of the LDH level at a single time point, equivalence will be declared if the 95% CI of the difference between treatments in LDH level at Week 26 is entirely contained within the pre-defined equivalence margin of  $[-1.2 \times \text{ULN}, 1.2 \times \text{ULN}]$  where ULN of LDH to be specified in the central laboratory specification for this study.

If normal range of LDH is gender specific, the smaller/smallest ULN will be used for the equivalence margin; otherwise ULN is not gender specific, unified ULN will be used for the equivalence margin.

## 9.2. Analysis Sets

The following sets will be used for the analyses performed in the study:

- Randomised Set (RAN) consists of all subjects who have received a randomisation number.
- Modified Full Analysis Set (M-FAS) consists of all RAN subjects who do not have positive result of pharmacogenetic analysis (C5 gene polymorphism). However, subjects who do not have any efficacy assessment result after randomisation and do not receive IP during the study period will be excluded from this analysis set. Following the intent-to-treat principle, subjects will be analysed according to the treatment sequence they are assigned to at randomisation.
- Per-Protocol Set for AUEC of LDH (PPS-AUEC) consists of all M-FAS subjects who have sufficient LDH assessments for AUEC calculation without any major PDs that have impact on efficacy assessment. Subjects excluded from the primary analysis will be pre-defined on a case-by-case basis prior to unblinding the treatment sequence assignment for analyses. In addition, subjects who received different treatment from the randomised treatment sequence due to a shortage of the comparator will be excluded from this analysis set.
- Per-Protocol Set for LDH at a single time point (PPS-single) consists of all M-FAS subjects who have LDH assessment at Week 26 without any major PDs that have impact on efficacy assessment. Subjects excluded from the primary analysis will be pre-defined on a case-by-case basis prior to unblinding the treatment sequence assignment for analyses. In addition, subjects who received different treatment in Period 1 from the randomised treatment sequence due to a shortage of the comparator will be excluded from this analysis set.
- Safety Set (SAF) consists of all subjects who receive at least one IP during the study period. Subjects will be analysed according to the treatment received.
- PK Analysis Set (PKS) consists of all subjects in the SAF who have at least one PK sample analysed.
- PD Analysis Set (PDS) consists of all subjects in the SAF who have at least one PD sample analysed.

## 9.3. Subject Demographic and Baseline Characteristics

The baseline value will be defined as the last available measurement value prior to or on the date of the

initiation of study drug.

Subject demographics and baseline disease characteristics will be summarised by treatment sequence for the RAN. Continuous variables (e.g., age, weight, height) will be summarised with descriptive statistics (n, mean, standard deviation [SD], median, minimum, maximum) and categorical variables (e.g., gender, race, ethnicity) will be summarised with count and percentage.

Comparison between treatment sequences in demographics and baseline disease characteristics will be performed using the chi-square test or *F*-test as appropriate. The results of these tests will be provided including the *p*-value only for descriptive purposes and will not be used as a formal basis to determine the factors to be included in primary or secondary efficacy analysis models. If baseline imbalances are detected for any of the factors, additional analyses may be performed to adjust for these baseline differences.

Relevant medical history, transfusion history, and continuing medical conditions will be summarised by treatment sequence for the RAN.

## 9.4. Analysis of the Primary Objectives

for those who are in favour of the time-adjusted AUEC of LDH, the primary efficacy analysis will be performed for the PPS-AUEC using a linear mixed model with treatment, sequence, period, and gender as fixed effects, and subject nested within sequence as a random effect. The analysis will be performed with log<sub>e</sub>-transformed time-adjusted AUEC of LDH estimating the difference in least squares means and its 90% CI, and back transformation of those values will provide the ratio of geometric means and 90% CI. The equivalence will be declared if the two-sided 90% CI of the ratio of geometric means in time-adjusted AUEC of LDH between SB12 and Soliris<sup>®</sup> lies within the pre-defined equivalence margin of [0.77, 1.29].

for those who are in favour of the LDH level at a single time point, the primary efficacy analysis will be performed for the PPS-single using a linear mixed model with treatment, and gender as a fixed effect. The analysis will be performed with loge-transformed LDH at Week 26 estimating the difference in least squares means and its 95% CI, and the delta method will be used to provide the mean difference and 95% CI in original scale. The equivalence will be declared if the two-sided 95% CI of the mean difference in LDH level at Week 26 between SB12 and Soliris® lies within the pre-defined equivalence margin of [-1.2 × ULN, 1.2 × ULN] where ULN of LDH to be specified in the central laboratory specification for this study.

No formal adjustment of Type I error rates will be performed.

For the primary analysis with the M-FAS, missing data will be imputed for subjects who drop out for the study prior to the primary analysis time point. A missing-at-random approach will assume that subjects who withdraw from a study had similar missing values to peer subjects who completed the study in that treatment sequence. This approach ensures that evidence of lack of equivalence is not diluted when there are missing data. Multiple imputation method will be used with the assumption of monotone missing pattern and regression method. For the sensitivity analyses, complete case analysis will be performed.

## 9.5. Analysis of the Secondary Objectives

## 9.5.1. Efficacy Variable Analyses

As a secondary efficacy endpoint, number of units of pRBCs transfused will be summarised descriptively by treatment sequence and treatment sequence within period and will be analysed using

Samsung Bioepis -  Information

Wilcoxon rank-sum test. And mean LDH profile will be presented over time.

## 9.5.2. Safety Analyses

All reported terms for AEs will be coded using Medical Dictionary for Regulatory Activities (MedDRA®). AEs will be collected and classified according to NCI-CTCAE v5.0. For all AE and SAE tables, subjects will be counted once for each preferred term and each system organ class.

A TEAE will be defined as any AE with an onset date on or after the date of the initiation of study drug. AEs which are already present before the initiation of study drug and increase in severity after the initiation of study drug will be considered as TEAEs. Pre-existing AEs before the initiation of study drug with no increase in severity after the initiation of study drug will not be considered as TEAEs.

All TEAEs and SAEs will be summarised respectively by count and percentage of subjects experiencing events by system organ class, preferred term. TEAEs leading to IP discontinuation and TEAEs by causality and severity will be summarised similarly. All AEs including those pre-existing before the initiation of study drug will be listed by subject.

In addition, infection-related AEs including meningococcal infection and other systemic infection, and IRRs will also be summarised.

Duration of exposure to IP and number of IV infusion will be summarised by treatment sequence within period with descriptive statistics for the SAF. Prior and concomitant medications, and significant non-drug therapies will be summarised with count and percentage.

Changes in vital signs and clinical laboratory parameters will be summarised descriptively by treatment sequence and visit. Other safety variables will be summarised unless otherwise specified, and all safety variables will be listed.

All safety analyses will be performed using the SAF. Additional analyses will be performed for the subjects who received different treatment from the randomised treatment sequence due to a shortage of the comparator if needed. For example, AEs and concomitant medications will be analysed based on the actual switched treatment.

#### 9.5.3. Pharmacokinetic Analyses

PK analysis will be performed for the PKS. C<sub>trough</sub> will be summarised with descriptive statistics by treatment sequence, period, and time point.

#### 9.5.4. Immunogenicity Analyses

ADA and NAb results (e.g., 'positive' or 'negative') will be summarised with count and percentage by treatment sequence and visit. In addition, incidence of overall ADA will be summarised by treatment sequence and period.

Immunogenicity analyses will be performed using the SAF.

## 9.5.5. Pharmacodynamic Analyses

PD analysis will be performed for the PDS. The absolute values, and change from baseline in terminal complement activities will be summarised by treatment sequence and visit. PD data for each subject will also be listed.

# 9.6. Sample Size Calculations

The equivalence margin for the mean difference of LDH at Week 26 is derived from two historical

studies with Soliris®. In TRIUMPH study, the mean (SD) of LDH at Week 26 is 327.3 (432.9) U/L and 2,418.9 (930.6) U/L for eculizumab and non-eculizumab arms, respectively. PNH registry study reported the mean of LDH at 6 months is 352.1 (224.0) U/L and 1,201.0 (815.6) U/L for eculizumab and non-eculizumab arms, respectively.

**Table 6. LDH Level from Reference Studies** 

| | E | culizumab | No | on-eculizumab | Note |
|---|---|---|---|---|---|
| | N | Mean (SD) | N | Mean (SD) | 11010 |
| TRIUMPH study (2006) <sup>a</sup> | 41 | 327.3 (432.9) | 44 | 2,418.9 (930.6) | Results at Week 26 |
| International PNH registry (2016) | 38 | 352.1 (224.0) | 102 | 1,201.0 (815.6) | Results at 6 months |
| Meta-analysis for mean difference with 95% CIs | -1,152.5 [-1,303.4, -1,001.7] | | | | |

<sup>&</sup>lt;sup>a</sup> SD for TRIUMPH study was derived from the standard error in the reference paper.

A meta-analysis with fixed-effect model estimates -1,152.5 U/L of LDH mean at Week 26 with a 95% CI [-1,303.4,-1,001.7]. The of upper limit of 95% CI was approximately U/L, which implies that at least treatment effect is obtained to preserve the treatment effect over placebo if the U/L was statistically chosen as the equivalence limit.

In the clinical study, LDH detection level or normal range of LDH would depend on the specification of laboratory parameters chosen for the study. Therefore, it is not likely to be clinically meaningful to propose any specific LDH level as the equivalence margin without the consideration of normal range of LDH level.



Therefore, the equivalence margin will be [-1.2 × ULN, 1.2 × ULN] for the comparison with the 95% CI of the mean difference in LDH at Week 26 where ULN of LDH to be specified in the central laboratory specification for this study. For sample size calculation, [-268 U/L, 268 U/L] is chosen to be 23 subjects per treatment sequence with the assumptions of no mean difference and common SD of 270 U/L at the overall 5% significance level. Assuming a 5% loss from randomised subjects after 26 weeks, a sample size of 25 subjects per treatment sequence (overall sample size of 50) will give 23 completers per treatment sequence after 26 weeks, which is estimated to give 80% power to detect the equivalence within the margin of 268 U/L.

The nQuery Advisor® option two-group *t*-tests (two one-sided test [TOST]) of equivalence in means (equal n's) gives the following statement to estimate the n per group to show the equivalence: "When the sample size in each group is 23, a two group design will have 80% power to reject both the null hypothesis that the test mean minus the standard mean is below –268 and the null hypothesis that the test mean minus the standard mean is above 268 i.e., that the test and standard are not equivalent, in favor of the alternative hypothesis that the means of the two groups are equivalent, assuming that the expected difference in means is 0, the common standard deviation is 270 and that each test is made at the 2.5% level."

For calculation of the equivalence margin for time-adjusted AUEC of LDH, mean and coefficient of

variation (%CV) were referred from TRIUMPH study. The mean (%CV) of AUEC of LDH at Week 26 is  $81,140.0~\text{U/L} \times \text{day}$  (142.45%) and 429,874.1 U/L × day (33.49%) for eculizumab and non-eculizumab arms, respectively.



With the given equivalence margin of [0.77, 1.29], 22 subjects per treatment sequence was calculated with the assumptions of the mean ratio of 1, common %CV of 42% at the overall 10% significance level. Assuming a 10% loss from randomised subjects after 52 weeks, a sample size of 25 subjects per treatment sequence (overall sample size of 50) will give 22 completers per treatment sequence after 52 weeks, which is estimated to give 80% power to detect the equivalence within the margin of [0.77, 1.29].

The nQuery Advisor® option two-group t-tests (TOST) of equivalence for ratio of means (log-scale) gives the following statement to estimate the n per group to show the equivalence: "When the sample size in each sequence group is 22 (and the total sample size is 44), a crossover design will have 80% power to reject both the null hypothesis that the ratio of the test mean to the standard mean is below 0.77 and the null hypothesis that the ratio of test mean to the standard mean is above 1.29; i.e., that the test and standard are not equivalent, in favor of the alternative hypothesis that the means of the two treatments are equivalent, assuming that the expected ratio of means is 1, the Crossover ANOVA,  $\sqrt{MSE}$  (In scale) is  $\frac{1}{2}$  (the SD differences,  $\sigma$  (In scale) is  $\frac{1}{2}$ ), that data will be analyzed in the natural log scale using t-tests for differences in means, and that each t-test is made at the 5% level."

Therefore, the sample size of 50 allows enough power to detect the equivalence in both situations.

# 10. Data Collection and Management

## 10.1. Data Confidentiality

Information about study subjects will be kept confidential. Study information will be labelled with a code number, and will not include the subject's name, hospital number or other information that could identify them. A list linking the code and the subject's name will be kept in the site files as required by ICH-GCP to protect the subject's confidentiality.

The coded information will be sent to the Sponsor (or designee) who will analyse it and report the study results both to regulatory and ethical authorities. The Sponsor may also place data on public websites or publish journal articles based upon these results. Care will be taken to prevent subjects being identified through these publications. In addition, data may be shared with other companies or researchers to aid further research into complement inhibitor. Such data sharing practices will be covered by confidentiality agreements. No-one outside the investigational site will have access to subject-identifiable information.

#### 10.2. Monitoring

The Sponsor has engaged the services of a contract research organisation (CRO) to perform all monitoring functions within this clinical study. The monitors will work in accordance with the CRO SOPs and have the same rights and responsibilities as monitors from the Sponsor. Monitors will establish and maintain regular contact between the Investigator and the Sponsor.

Monitors will evaluate the competence of each investigational site and inform the Sponsor about any problems relating to facilities, technical equipment or investigational site staff. During the study, Samsung Bioepis – * Information* 

monitors will check that written informed consent has been obtained correctly from all subjects and that data are recorded correctly and completely. Monitors will also perform source data verification by comparing entries in the eCRF with corresponding source data and informing the Investigator of any errors or omissions. Monitors will verify adherence to the protocol at the investigational site. All PDs will be reported to the Sponsor via the monitoring visit reports. Monitors will arrange for the supply of IP and ensure appropriate storage conditions are maintained.

Monitoring visits will be conducted at regular intervals according to ICH-GCP. The monitor will provide written reports to the Sponsor on each occasion they contact with the Investigator regardless of whether it is by phone or in person.

Further details on the monitoring processes and the level of source data verification to be performed will be outlined in the monitoring plan.

# 10.3. Data Handling and Record Keeping

The Investigator must maintain essential study documents (protocol and protocol amendments, completed eCRFs, signed ICFs and its revisions, relevant correspondence, and all other supporting documentation) until at least 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or at least 2 years after the formal discontinuation of clinical development of the IP or 15 years from completion of the study. These documents should be retained for a longer period if required by the applicable regulatory requirements or the investigational sites, institution or private practice in which the study is being conducted. Subject identification codes (subject names and corresponding study numbers) will be retained for the same period of time. These documents may be transferred to another responsible party, deemed acceptable by the Sponsor, and who agrees to abide by the retention policies. Written notification of transfer must be submitted to the Sponsor. The Investigator must contact the Sponsor prior to disposing of any study records and obtain written permission to do so.

## 10.4. Future Use of Stored Specimens and Data

The Sponsor or designated representative can store PK, immunogenicity, PD, and/or pharmacogenetic samples for maximum 15 years after the end of the clinical study. The Sponsor or designated representative should operate under the same regulations related to and take the same responsibility to save personal data. The sample may be used for additional assay to be performed if considered scientific relevant or requested by regulatory authorities in order to have the possibility to perform the assay.

## 10.5. Database Management and Coding

Data generated within this clinical study will be handled according to the relevant SOPs of the data management and biostatistics departments of the Sponsor (or an appropriate company designated by the Sponsor to perform these activities). Subject data will be captured in an eCRF and reviewed by the monitor in order to check adherence to the protocol and to detect any data inconsistency or discrepancy.

The Investigator must ensure that the clinical data required by the study protocol are carefully reported in the eCRF. He/she must also check that the data reported in the eCRF correspond to those in the medical records.

Data must be entered into eCRFs in English by the designated investigational site staffs in a timely manner. Forms should be available during periodic visits by study monitors to enable review for completeness and acceptability. Any correction to the data entered into the eCRF must be carried out by the Investigator or a designated investigational site staffs. These changes may be made either on the initiative of the investigational site staffs or in response to monitoring or data queries. Any changes to

written data must be made using ICH-GCP corrections and any change to electronic data should be made in a system which can provide an audit trail. Monitors and clinical data managers will review the eCRF for accuracy and can generate queries to the investigational site staffs for resolution. Corrections will be recorded in an audit trail that records the original information, the corrected information, and identification of the person making the changes, date of correction made and reason for change. The Investigator must sign and date the eCRF pages as indicated.

Medical/surgical history and underlying diseases and AEs will be coded using the MedDRA<sup>®</sup>. Concomitant medications will be coded using the World Health Organization-Drug Dictionary Enhanced (WHO-DDE). The versions of coding dictionaries used will be stated in the CSR.

## 10.6. Quality Control and Quality Assurance

During the conduct of the study, the Sponsor or its agent will conduct periodic monitoring visits to ensure that the protocol and ICH-GCP are being followed. The monitors may review source documents to confirm that the data recorded are accurate. The Investigator and institution will allow the domestic and foreign regulatory authorities, the Sponsor's monitors and auditors' direct access to source documents to perform this verification. The investigational site may be subject to review by the IRB/IEC, and/or to quality assurance audits performed by the Sponsor, and/or to inspection by appropriate regulatory authorities. It is important that the Investigators and their relevant personnel are available during the monitoring visit, possible audits and/or regulatory inspection(s) and that sufficient time is devoted to the process.

#### 10.7. Protocol Deviation

PDs will be pre-defined prior to subject enrolment and documented separately named as "protocol deviation definition list" which includes category (e.g., violation of inclusion/exclusion criteria, use of prohibited medication, non-compliance with treatment), deviation description, severity (major or minor), time point for PDs. Major PDs are defined as those deviations from the protocol likely to have an impact on the perceived efficacy and/or safety of study treatments.

PDs will be reviewed and confirmed prior to database lock to decide which subjects and/or subject data will be excluded from certain analyses. Decisions regarding the exclusion of subjects and/or subject data from analyses will be documented and approved prior to database lock.

## 11. Ethics Considerations and Administrative Procedures

## 11.1. Institutional Review Boards and Independent Ethics Committees

The Investigator and the Sponsor will follow all local laws and regulations relating to contact with and approvals from the IRB/IEC.

The Investigator must provide the Sponsor with documentation of IRB/IEC approval of the protocol and informed consent before the study may begin at the investigational site. The Investigator will supply documentation to the Sponsor relating to the annual renewal of the protocol from the IRB/IEC and any approvals of revisions to the ICF or amendments to the protocol.

The Investigator will report promptly to the IRB/IEC any new information that may adversely affect the safety of subjects or the conduct of the study. Similarly, the Investigator will submit written summaries of the study status to the IRB/IEC on a regular basis and in accordance with the timelines required locally. Upon completion of the study, the Investigator will provide the ethics committee with a report on the outcome of the study if required by local regulations.

## 11.2. Ethical Conduct of the Study

This study will be conducted and informed consent will be obtained from each subject according to the ethical principles stated in the Declaration of Helsinki (2013), the applicable guidelines for ICH-GCP and the applicable drug and data protection laws and regulations of the countries where the study will be conducted.

#### 11.3. Written Informed Consent

The written informed consent will be used to explain the risks and benefits of study participation to the subject in simple terms before the subject enters into the study. The ICF contains a statement that the consent is freely given, that the subject is aware of the risks and benefits of entering the study, and that the subject is free to withdraw from the study at any time. Written consent must be given by the subject and/or legal representative, after the receipt of detailed information on the study.

The Investigator is responsible for ensuring that informed consent is obtained from each subject or legal representative and for obtaining the appropriate signatures and dates on the ICF prior to the performance of any protocol procedures and prior to the administration of IP. The Investigator will provide each subject with a copy of the signed and dated ICF and this will be documented on the subject's source document.

## 11.4. Investigator Information

## 11.4.1. Investigator Obligations

This study will be conducted in accordance with the ICH-GCP, the ethical principles that have their origin in the Declaration of Helsinki (2013) and local laws and regulations.

The Investigator is responsible for ensuring that the study is conducted according to the signed Investigator statement, the study protocol and applicable regulations; for protecting the rights, safety, and welfare of subjects under the Investigator's care; and for the control of drugs under investigation. The Investigator must obtain the informed consent of each subject to whom IP is administered.

## 11.4.2. Training of Investigational Site Personnel

Before the first subject is enrolled into the study, the Sponsor representative will review and discuss the requirements of the clinical study protocol and related documents with the investigational site staff and will also train them in any study-specific procedures.

The Investigator will ensure that appropriate training relevant to the study is given to all investigational site staff and that any new information relevant to the performance of this study is forwarded to the investigational site staff involved.

The Investigator will maintain a record of all individuals involved in the study (medical, nursing, and other investigational site staff).

#### 11.4.3. Protocol Signatures

The Investigator must sign the Investigator signature page of this protocol prior to starting recruitment for the study. By signing the protocol, the Investigator confirms in writing that he/she has read, understands and will strictly adhere to the study protocol and will conduct the study in accordance with ICH-GCP and applicable regulatory requirements. The study will not be able to start at any investigational site where the Investigator has not signed the protocol.

## 11.4.4. Financing and Insurance

Samsung Bioepis is the Sponsor of this study and will be providing the finances to cover the operation of the study. Details of financial agreements are provided in the clinical trial agreement with the investigational sites and in contracts with other companies involved in the running of the study.

The Sponsor has obtained suitable insurance for this study. A copy of the insurance details will be provided to each Investigator who will be responsible for providing the IRB/IEC with these details according to local requirements.

# 12. Publication Policy

The Sponsor supports the efforts of health authorities to increase the transparency of medical research conducted in human subjects. The Sponsor will register and maintain the information of clinical studies on a public registry program. The Sponsor is committed to the public disclosure of the results from clinical studies through posting on public clinical study data banks. The Sponsor will comply with the guidelines of regulatory authorities with regards to public registration and disclosure of clinical study data.

# 13. Extended Supply

After completion of activities at Week 52, an open-label extended supply of SB12 will be provided for up to 2 calendar years starting from Week 52 to subjects who have benefited from study treatment and opt to participate in extended supply under an ethical basis.

Before entering an extended supply, the Investigator will review the subject status including reduction of PNH disease activity, such as improvement of symptoms or laboratory parameters, during eculizumab treatment to decide if the subject will benefit from participation in extended supply. Once subjects are considered to benefit from extended supply, subjects will be asked if he/she would like to receive an extended supply. For receiving an extended supply, subjects should agree with signing ICF for extended supply and with required activities including refraining from pregnancy, maintaining a highly effective contraceptive method, and receiving meningococcal vaccination (if required by local regulations) to ensure subject's safety during extended supply.

During extended supply, Investigators will treat subjects with 900 mg of SB12 every  $14 \pm 2$  days for up to 2 years (104 weeks). SB12 will be packaged and labelled using open label and dispensed through the IWRS. Investigators should ensure the compliance and accountability of SB12 during the course of extended supply. Any PC must be reported to Sponsor.

SAEs that occur during this phase must be reported to the Sponsor, which will be reported to regulatory authorities by the Sponsor according to local/national requirements via expedited reporting and periodic reporting such as Development Safety Update Report (DSUR) or Periodic Safety Update Report (PSUR). Pregnancy should also be reported until 5 months after the last SB12 treatment. Other particular activities will not be imposed and no data collection or reporting will occur for extended supply.

Discontinuation of study treatment can be decided if unacceptable toxicity, pregnancy, other complement inhibitor use or lack of efficacy occurs, or at the discretion of the Investigator or by subject's consent withdrawal. Specific study procedures are not required for subjects who have discontinued prematurely except for SAEs reporting and pregnancy reporting.

During the period of extended supply, the Investigator and the Sponsor will follow all local laws and regulations relating to contact with and approvals from the IRB/IEC. The Investigator is responsible for ensuring that the study is conducted according to the signed Investigator statement, the study protocol and applicable regulations; for protecting the rights, safety, and welfare of subjects under the Investigator's care; and for the control of drugs under investigation.

The Investigators must maintain essential study documents until at least 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or at least 2 years after the formal discontinuation of clinical development of the IP or 15 years from completion of the extended supply, if applicable.

Investigational sites participation may be discontinued if the Sponsor, Investigator or IRB/IEC consider necessary. Extended supply may be terminated by the Sponsor if medically or ethically indicated, and in such cases will be promptly notified to the Investigator. In any case, health authorities and IRB/IEC will be informed for the action in accordance with applicable regulations.

## 14. References

- [1] Hillmen P, Lewis S, Bessler M, et al. Natural history of paroxysmal nocturnal hemoglobinuria. *N Engl J Med.* 1995; 333 (19): 1253-8.
- [2] Moyo V, Mukhina G, Garrett E, et al. Natural history of paroxysmal nocturnal haemoglobinuria using modern diagnostic assays. *Br J Haematol*. 2004; 126 (1): 133-8.
- [3] Nishimura J, Kanakura Y, Ware R, et al. Clinical course and flow cytometric analysis of paroxysmal nocturnal hemoglobinuria in the United States and Japan. *Medicine (Baltimore)*. 2004; 83 (3): 193-207.
- [4] Sharma V. Paroxysmal nocturnal hemoglobinuria: pathogenesis, testing, and diagnosis. *Clin Adv Hematol Oncol*. 2013; 11 Suppl 13 (9): 2-8.
- [5] Parker C, Omine M, Richards S, et al. Diagnosis and management of paroxysmal nocturnal hemoglobinuria. *Blood*. 2005; 106 (12): 3699-709.
- [6] Hartmann R, Jenkins D, Mckee L, et al. Paroxysmal nocturnal hemoglobinuria: clinical and laboratory studies relating to iron metabolism and therapy with androgen and iron. *Medicine* (*Baltimore*). 1966; 45 (5): 331-63.
- [7] Hill A, Hillmen P, Richards S, et al. Sustained response and long-term safety of eculizumab in paroxysmal nocturnal hemoglobinuria. *Blood*. 2005; 106 (7): 2559-65.
- [8] Hillmen P, Young N, Schubert J, et al. The complement inhibitor eculizumab in paroxysmal nocturnal hemoglobinuria. *N Engl J Med*. 2006; 355 (12): 1233-43.
- [9] Brodsky R, Young N, Antonioli E, et al. Multicenter phase 3 study of the complement inhibitor eculizumab for the treatment of patients with paroxysmal nocturnal hemoglobinuria. *Blood*. 2008; 111 (4): 1840-7.
- [10] Soliris<sup>®</sup> EPAR Product Information. EMA (Jul 01, 2020). Retrieved Jul 13, 2020 from <a href="https://www.ema.europa.eu/en/documents/product-information/soliris-epar-product-information en.pdf">https://www.ema.europa.eu/en/documents/product-information/soliris-epar-product-information en.pdf</a>
- [11] Guideline on similar biological medicinal products monoclonal antibodies. EMA. (May 2012). EMA/CHMP/BMWP/403543/2010. Retrieved Jun 04, 2018 from <a href="http://www.ema.europa.eu/docs/en\_GB/document\_library/Scientific\_guideline/2012/06/WC500128686.pdf">http://www.ema.europa.eu/docs/en\_GB/document\_library/Scientific\_guideline/2012/06/WC500128686.pdf</a>
- [12] Rother RP, Bell L, Hillmen P, et al. The clinical sequelae of intravascular hemolysis and extracellular plasma hemoglobin: a novel mechanism of human disease. *JAMA*. 2005; 293 (13): 1653-62.
- [13] Hill A, Rother R, Wang X, et al. Effect of eculizumab on haemolysis-associated nitric oxide depletion, dyspnoea, and measures of pulmonary hypertension in patients with paroxysmal nocturnal haemoglobinuria. *Br J Haematol*. 2010; 149 (3): 414-25.
- [14] Weitz I. Thrombosis in Paroxysmal Nocturnal Hemoglobinuria insights into the role of complement in thrombosis. *Thromb Res.* 2010; 125 Suppl 2: S106-7.
- [15] Helley D, de Latour R, Porcher R, et al. Evaluation of hemostasis and endothelial function in patients with paroxysmal nocturnal hemoglobinuria receiving eculizumab. *Haematologica*. 2010; 95 (4): 574-81.
- [16] Hillmen P, Muus P, Dührsen U, et al. Effect of the complement inhibitor eculizumab on

thromboembolism in patients with paroxysmal nocturnal hemoglobinuria. Blood. 2007; 110 (12): 4123-8.

- [17] The Most Expensive Prescription Drugs in the World. Kathlyn Stone. (Updated Aug 26, 2018/Dec 11, 2017/Apr 24, 2017). Retrieved Oct 04, 2018 from <a href="https://www.thebalance.com/the-8-most-expensive-prescription-drugs-in-the-world-2663232">https://www.thebalance.com/the-8-most-expensive-prescription-drugs-in-the-world-2663232</a>
- [18] Devalet B, Mullier F, Chatelain B, et al. Pathophysiology, diagnosis, and treatment of paroxysmal nocturnal hemoglobinuria: a review. *Eur J Haematol*. 2015; 95 (3): 190-8.
- [19] de Latour R, Mary J, Salanoubat C, et al. Paroxysmal nocturnal hemoglobinuria: natural history of disease subcategories. *Blood.* 2008; 112 (8): 3099-106.
- [20] Kato G, McGowan V, Machado R, et al. Lactate dehydrogenase as a biomarker of hemolysis-associated nitric oxide resistance, priapism, leg ulceration, pulmonary hypertension, and death in patients with sickle cell disease. *Blood.* 2006; 107 (6): 2279-85.
- [21] Soliris® Prescribing Information. FDA (Nov 20, 2020). Retrieved Nov 26, 2020 from <a href="https://www.accessdata.fda.gov/drugsatfda">https://www.accessdata.fda.gov/drugsatfda</a> docs/label/2020/125166s434lbl.pdf

# APPENDIX A. Paroxysmal Nocturnal Haemoglobinuria Symptoms Subject Questionnaire

Following signs and symptoms are associated with PNH.

If you have had the symptom in the past 7 days, please circle the number below that describe your severity for each sign or symptom.

| J | | 2 | 1 | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| 1) ] | Fatigue | | | | | | | | | |
| 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| None | <u>.</u> | <u>-</u> | <u>-</u> | | <u></u> | <u></u> | | | | Severe |
| 2) ] | Haemoglo | obinuria ( | discolour | ation of u | rine) | | | | | |
| 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| None | <u> </u> | <u> </u> | <u> </u> | <u> </u> | <u>i</u> | <u> </u> | <u> </u> | <u> </u> | <u> </u> | Severe |
| 3) ( | Chest pair | 1 | | | | | | | | |
| 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| None | | | <b>-</b> | | | | | | | Severe |
| 4) | Abdomina | al pain | | | | | | | | |
| 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| None | | | | | | | | | | Severe |
| 5) ] | Dyspnoea | (shortnes | ss of brea | th) | | | | | | |
| 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| None | · | <u> </u> | · | | ·£ | | | | | Severe |
| 6) ] | Dysphagia | a | | | | | | | | |
| 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| None | <u></u> | <u> </u> | <u> </u> | · <del>·</del> | <u></u> | <u>-i</u> | <u>.</u> | · <del>·</del> | <u></u> | Severe |
| 7) ] | Erectile d | ysfunction | n (if appl | icable) | | | | | | |
| 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| None | <u>i</u> | <u>L</u> | <u>L</u> | <u>i</u> | <u>i</u> | <u>i</u> | <u>i</u> | <u>i</u> | <u>.</u> | Severe |
# **Protocol Signature Pages**

#### SIGNATURE PAGE

### **Declaration of Sponsor Representative**

**Protocol Title**: A Phase III Randomised, Double-blind, Multicentre Study to Compare the Efficacy, Safety, Pharmacokinetics, and Immunogenicity between SB12 (proposed eculizumab biosimilar) and Soliris® in Subjects with Paroxysmal Nocturnal Haemoglobinuria

This clinical study protocol was subjected to critical review. The information it contains is consistent with current knowledge of the risks and benefits of the investigational medicinal product, as well as with the moral, ethical, and scientific principles governing clinical research as set out in the Declaration of Helsinki, 2013 and the guidelines on Good Clinical Practice applicable to this clinical study.

#### Sponsor Representative

| Name: | | | |
|--------------|---------------------------|-------|----------------|
| Institution: | Samsung Bioepis Co., Ltd. | | |
| Signature: | | Date: | Nov 27, 2020. |
| | | | (MMM DD, YYYY) |

### SIGNATURE PAGE

### **Declaration of the Coordinating Investigator**

**Protocol Title**: A Phase III Randomised, Double-blind, Multicentre Study to Compare the Efficacy, Safety, Pharmacokinetics, and Immunogenicity between SB12 (proposed eculizumab biosimilar) and Soliris® in Subjects with Paroxysmal Nocturnal Haemoglobinuria

This clinical study protocol was subjected to critical review. The information it contains is consistent with current knowledge of the risks and benefits of the investigational medicinal product, as well as with the moral, ethical, and scientific principles governing clinical research as set out in the Declaration of Helsinki, 2013 and the guidelines on Good Clinical Practice applicable to this clinical study.

### **Coordinating Investigator**



### SIGNATURE PAGE

### **Declaration of the Principal Investigator**

**Principal Investigator** 

**Protocol Title**: A Phase III Randomised, Double-blind, Multicentre Study to Compare the Efficacy, Safety, Pharmacokinetics, and Immunogenicity between SB12 (proposed eculizumab biosimilar) and Soliris® in Subjects with Paroxysmal Nocturnal Haemoglobinuria

This clinical study protocol was subjected to critical review. The information it contains is consistent with current knowledge of the risks and benefits of the investigational medicinal product, as well as with the moral, ethical, and scientific principles governing clinical research as set out in the Declaration of Helsinki, 2013 and the guidelines on Good Clinical Practice applicable to this clinical study.

| • | S | | |
|--------------|---|-------|----------------|
| Name: | | | |
| Institution: | | | |
| Signature: | | Date: | |
| _ | | | (MMM DD, YYYY) |

# CHANGE HISTORY OF PROTOCOL AMENDMENT

Amendment 1: Version 2.0, Oct 08, 2018

| Section<br>Affected | Ori | ginal Content | | | Amen | ded/New Cont | tent | Rationale |
|---|---|---|---|---|---|---|---|---|
| SYNOPSIS<br>Exclusion<br>Criteria | <ul><li>4. Abnormal haematologicathe following:</li><li>a. Absolute neutrophi</li><li>b. Platelet count &lt; 80,</li></ul> | l count (ANC) | - | ed as | <ul><li>4. Abnormal haematologic the following:</li><li>a. Absolute neutroph</li><li>b. Platelet count &lt; 86</li></ul> | il count (ANC) | $) \le 500/\text{mm}^3$ | To change platelet count criteria |
| Figure 1 | Confirmed PNH (m=50) Treatment-naive 1 ls years W-8 W-2 W0 <sup>5</sup> W4 <sup>4</sup> W1 <sup>4</sup> Screening 1 <sup>2</sup> dosing* Period 1 | Period I AUECe → W266e | W40 V Period 2 | Soliris* | Sequence I (n=25) Confirmed PNH (n=50) Treatment-curve 2 it years W-5 W-5 W-5 W-5 W-5 Sequence II (n=25) Sequence II (n=25) Freshold Sequence II (n=25) Freshold Sequence II (n=25) Freshold Sequence II (n=25) Freshold Freshold Sequence II (n=25) | Period 1 AUEC <sup>d</sup> | SB12 Soliris* Period 2 AUEC* W40 W52 EQS Period 2 | To extend the period from randomisation to initiation of study drug taking account of IP shipment |
| Figure 1<br>Footnote | a. Randomisation will triginvestigational site. The done within 14 days of | e initiation of s | study drug should | | a. Randomisation will tr<br>investigational site. To<br>done within <b>14-21 day</b> | he initiation of | study drug should be | To extend the period from randomisation to initiation of study drug taking account of IP shipment |
| Table 1 | Assessments Study Visit Week | Scree<br>-ning | -sation | | Assessments Study Visit Week | Scree<br>-ning | Randomisation | To extend the period from randomisation to initiation of study |
| | Day (± Visit Window) | -56 to -15 | -14 to -1 | ••• | Day (± Visit Window) | =56 to -15<br>-63 to -22 | = <del>14 to -1</del><br>-21 to -1 | drug taking account of IP |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | | | shipment |
| Table 1<br>Footnote | 4. All screening procedures must be completed and reviewed within 42 days prior to randomisation. All eligibility criteria must be reviewed and confirmed prior to randomisation. The initiation of study drug (Day 1) should be done within 14 days of randomisation. | 4. All screening procedures must be completed and reviewed within 42 days prior to randomisation. All eligibility criteria must be reviewed and confirmed prior to randomisation. The initiation of study drug (Day 1) should be done within 14-21 days of randomisation. | To extend the period from randomisation to initiation of study drug taking account of IP shipment |
| Table 1<br>Footnote | 8. Both white blood cell (WBC) and red blood cell (RBC) clone size will be measured by flow cytometry prior to dosing at Screening, Day 1, and Week 52. () | 8. Both white blood cell (WBC) and red blood cell (RBC) clone size will be measured by flow cytometry prior to dosing at Screening, and prior to dosing at Day 1,—and Week 52. () | To clarify the meaning because no dosing will be done at Screening |
| Table 1<br>Footnote | 11. Parameters included in haematology test are WBC count, RBC count, haemoglobin, haematocrit, platelet count, differential WBC count, nucleated RBC, mean corpuscular haemoglobin (MCH), mean corpuscular haemoglobin concentration (MCHC), mean corpuscular volume (MCV), mean platelet volume (MPV), and red cell distribution width (RDW). () | 11. Parameters included in haematology test are WBC count, RBC count, haemoglobin, haematocrit, platelet count, differential WBC count, and nucleated RBC, mean corpuscular haemoglobin (MCH), mean corpuscular haemoglobin concentration (MCHC), mean corpuscular volume (MCV), mean platelet volume (MPV), and red cell distribution width (RDW). () | To remove several haematology test parameters |
| Table 2<br>Footnote | 5. Both WBC and RBC clone size will be measured by flow cytometry prior to dosing at Screening, Day 1, and Week 52. () | 5. Both WBC and RBC clone size will be measured by flow cytometry prior to dosing at Screening, and prior to dosing at Day 1, and Week 52. () | To clarify the meaning because no dosing will be done at Screening |
| Table 2<br>Footnote | 8. Parameters included in haematology test are WBC count, RBC count, haemoglobin, haematocrit, platelet count, differential WBC | 8. Parameters included in haematology test are WBC count, RBC count, haemoglobin, haematocrit, platelet count, differential WBC | To remove several haematology test parameters |

| Section<br>Affected | | Original Conten | t | | Amended/New Content | Rationale |
|---|---|---|---|---|---|---|
| | | count, nucleated RB0 MPV, and RDW. ( | C, MCH, MCHC, MCV, | | count, and nucleated RBC <del>, MCH, MCHC,</del> MCV, MPV, and RDW. () | |
| LIST OF<br>ABBREVIA<br>-TIONS | MCHC I | Mean corpuscular haen<br>Mean corpuscular haen<br>Mean corpuscular volu<br>Mean platelet volume | noglobin concentration | MCHC<br>MCV | Mean corpuscular hacmoglobin Mean corpuscular hacmoglobin concentration Mean corpuscular volume | To remove several haematology test parameters |
| | RDW I | Red cell distribution w | idth | MPV<br>RDW | Mean platelet volume Red cell distribution width | |
| LIST OF<br>STUDY<br>STAFF | Clinical Research Scientist Safety Physician | | | Clinical<br>Research<br>Scientist<br>Safety<br>Physician | | Administrative change due to study staff change |
| 4.3.<br>Exclusion<br>Criteria | the following: a. Absolute: | natological parameters neutrophil count (ANC ount < 80,000/mm <sup>3</sup> | at Screening defined as $C \le 500/\text{mm}^3$ | the following: a. Absolut | ematological parameters at Screening defined as e neutrophil count (ANC) $\leq 500/\text{mm}^3$ count $< 80,000 70,000/\text{mm}^3$ | To change platelet count criteria |
| Table 4. Parameters for Clinical Laboratory | Haematology | WBC count RBC count | Mean corpuscular<br>haemoglobin<br>(MCH) | Haematology | WBC count Mean | To remove several haematology test parameters |

Samsung Bioepis -  Information

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| Tests | Haemoglobin Haematocrit Platelet count Differential WBC count Nucleated RBC Mean corpuscular volume (MCV) Mean platelet volume (MPV) Red cell distribution width (RDW) | <ul> <li>Haemoglobin</li> <li>Haematocrit</li> <li>Platelet count</li> <li>Differential WBC count</li> <li>Nucleated RBC</li> <li>Mean concentration (MCHC)</li> <li>Mean corpuscular concentration (MCHC)</li> <li>Mean corpuscular corpuscular corpuscular volume (MCV)</li> <li>Mean platelet volume (MPV)</li> <li>Red cell distribution width (RDW)</li> </ul> | |
| 6.2.3.<br>Physical<br>Examination<br>s | Physical examination including height and weight will performed before IP administration at Screening and physical examination including weight at the visits specified in Table 1 and Table 2. () | | To clarify the meaning because no dosing will be done at Screening |
| 7.1.1.1.<br>Screening<br>Visit (D-63<br>to D-22) | 7.1.1.1. Screening Visit (D-56 to D-15) | 7.1.1.1. Screening Visit ( <del>D=56</del> D=63 to <del>D=15</del> D=22) | To extend the period from randomisation to initiation of study drug taking account of IP shipment |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| 7.1.1.1.<br>Screening<br>Visit (D–63<br>to D–22) | Review of laboratory results Haematology: Haemoglobin, haematocrit, RBC count, total WBC count including differential count, platelet count, nucleated RBC, MCH, MCHC, MCV, MPV, and RDW | <ul> <li>Review of laboratory results</li> <li>Haematology: Haemoglobin, haematocrit, RBC count, total WBC count including differential count, platelet count, and nucleated RBC, MCH, MCHC, MCV, MPV, and RDW</li> </ul> | To remove several haematology test parameters |
| 7.1.1.1.<br>Screening<br>Visit (D–63<br>to D–22) | Review of laboratory results Urinalysis: Protein, blood, leukocytes, nitrite, ketone, glucose, pH, specific gravity, bilirubin, urobilinogen, appearance, and colour (if urinalysis result is abnormal, urine microscopic examination will be performed) | <ul> <li>Review of laboratory results</li> <li>Urinalysis: Protein, blood, leukocytes esterase, nitrite, ketone, glucose, pH, specific gravity, bilirubin, urobilinogen, appearance, and colour (if urinalysis result is abnormal, urine microscopic examination will be performed)</li> </ul> | To change urinalysis parameter to be consistent with Table 4 |
| 7.1.1.1.<br>Screening<br>Visit (D–63<br>to D–22) | Review of laboratory results | <ul> <li>Review of laboratory results</li> <li>Others: Ferritin, vitamin B<sub>12</sub>, and folate</li> </ul> | To add laboratory<br>tests to be<br>consistent with<br>Table 1 |
| 8.3.2. Other<br>Systemic<br>Infections | SB12 or Soliris® blocks terminal complement activation; therefore subjects may have increased susceptibility to infections, especially with encapsulated bacteria. Additionally, aspergillus infections have occurred in immunocompromised and neutropenic patients. Subjects should immediately call the Investigator or seek emergency medical care, if subjects experience other systemic infections. | SB12 or Soliris® blocks terminal complement activation; therefore subjects may have increased susceptibility to infections, especially with encapsulated bacteria. Serious infection with Neisseria species (other than Neisseria meningitidis), including disseminated gonococcal infections, have been reported after Soliris® treatment. Additionally, aspergillus infections have occurred in immunocompromised and neutropenic patients. Subjects should immediately call the Investigator or seek emergency medical care, if subjects experience other systemic infections. | To add the updated safety information according to the latest version of regulatory document |
| 13. | [17] The Most Expensive Prescription Drugs in the World. Kathlyn Stone. (Updated Dec 11, 2017/Apr 24, 2017). Retrieved | [17] The Most Expensive Prescription Drugs in the World. Kathlyn Stone. (Updated <b>Aug 26, 2018/Dec 11, 2017/</b> Apr 24, | To refer the latest |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| References | Mar 09, 2018 from <a href="https://www.thebalance.com/the-8-most-expensive-prescription-drugs-in-the-world-2663232">https://www.thebalance.com/the-8-most-expensive-prescription-drugs-in-the-world-2663232</a> | 2017). Retrieved Mar 09, 2018 Oct 04, 2018 from <a href="https://www.thebalance.com/the-8-most-expensive-prescription-drugs-in-the-world-2663232">https://www.thebalance.com/the-8-most-expensive-prescription-drugs-in-the-world-2663232</a> | information |
| 13.<br>References | [21] Soliris® Prescribing Information. FDA (Feb 28, 2018). Retrieved Apr 25, 2018 from <a href="https://www.accessdata.fda.gov/drugsatfda_docs/label/2018/125166s426lbl.pdf">https://www.accessdata.fda.gov/drugsatfda_docs/label/2018/125166s426lbl.pdf</a> | [21] Soliris® Prescribing Information. FDA (Feb 28 Jul 25, 2018). Retrieved Apr 25 Oct 04, 2018 from https://www.accessdata.fda.gov/drugsatfda_docs/label/2018/125166s426lbl.pdf https://www.accessdata.fda.gov/drugsatfda_docs/label/2018/125166s047s048lbl.pdf | To refer the latest<br>version of<br>regulatory<br>document |

### Amendment 2: Version 3.0, Dec 12, 2018

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| SYNOPSIS<br>Exclusion<br>Criteria | N/A | 7. History of serious thrombotic event (e.g., stroke, myocardial infarction, pulmonary embolism, etc.) | To add exclusion criteria |
| SYNOPSIS<br>Secondary<br>Endpoints | <ul> <li>Immunogenicity endpoints</li> <li>Incidence of anti-drug antibodies (ADAs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and end of study (EOS)</li> <li>Incidence of neutralising antibodies (NAbs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and EOS</li> </ul> | <ul> <li>Immunogenicity endpoints</li> <li>Incidence of anti-drug antibodies (ADAs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and end of study (EOS)/early termination (ET)</li> <li>Incidence of neutralising antibodies (NAbs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and EOS/ET</li> </ul> | To add time point to be consistent with Table 2 |
| SYNOPSIS<br>Statistical<br>Methods | PK analyses PK analysis will be performed for the PK Analysis Set (PKS). Serum trough concentration will be summarised descriptively by treatment sequence, period, and time point. | PK analyses PK analysis will be performed for the PK Analysis Set (PKS). Serum trough concentration C <sub>trough</sub> will be summarised descriptively by treatment sequence, period, and time point. | To apply abbreviation |
| Figure 1<br>Footnote | ® = Randomisation; AUEC = Area under the Effect Curve; EOS = End of Study | <ul> <li>R = Randomisation; AUEC = Area under the Effect Curve; EOS</li> <li>End of Study; PNH = Paroxysmal Nocturnal</li> <li>Haemoglobinuria; W = Week</li> </ul> | To add abbreviations |
| 2.2.2.<br>Secondary<br>Endpoints | Immunogenicity endpoints • Incidence of anti-drug antibodies (ADAs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and end of study (EOS) | Immunogenicity endpoints • Incidence of anti-drug antibodies (ADAs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and end of study (EOS)/early termination (ET) | To add time point to be consistent with Table 2 |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | • Incidence of neutralising antibodies (NAbs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and EOS | • Incidence of neutralising antibodies (NAbs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and EOS/ET | |
| 3.2.1.<br>Scientific<br>Rationale for<br>Study<br>Design | for analysis of haemolysis reduction as measured by AUEC of LDH between two different time points in each period, the primary objective is to demonstrate comparable clinical efficacy of SB12 and Soliris® in terms of AUEC of LDH from Week 14 to Week 26 and from Week 40 to Week 52. The primary objective is to demonstrate comparable clinical efficacy of SB12 and Soliris® in terms of the LDH level (U/L) at Week 26. | () , for analysis of haemolysis reduction as measured by AUEC of LDH between two different time points in each period, the primary objective is to demonstrate comparable clinical efficacy of SB12 and Soliris® in terms of AUEC of LDH from Week 14 to Week 26 and from Week 40 to Week 52. , for analysis of haemolysis reduction as measured by the LDH level at single time point, the primary objective is to demonstrate comparable clinical efficacy of SB12 and Soliris® in terms of the LDH level (U/L) at Week 26 | To add phrase to be consistent within the document |
| 4.3.<br>Exclusion<br>Criteria | N/A | 7. History of serious thrombotic event (e.g., stroke, myocardial infarction, pulmonary embolism, etc.) | To add exclusion criteria |
| 5.1.1. Dosing and Treatment Schedule | SB12 or Soliris® will be administered up to Week 52 (a total of 29 administrations of IP) unless they are early discontinued from study treatment. | SB12 or Soliris® will be administered up to Week 52 (a total of 29 administrations of IP) unless they are early discontinued from study treatment. | To clarify dosing and treatment schedule |
| | • 600 mg every 7 ± 2 days for the first 4 weeks, followed by | • 600 mg every 7 ± 2 days for the first 4 weeks, followed by | |
| | <ul> <li>900 mg for the fifth dose 7 ± 2 days later, then</li> <li>900 mg every 14 ± 2 days thereafter</li> </ul> | <ul> <li>900 mg for the fifth dose 7 ± 2 days later, then</li> <li>900 mg every 14 ± 2 days thereafter</li> </ul> | |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| Anecteu | In case a dosing is delayed, next dosing visit date should not be altered. The subject receiving SB12 or Soliris® therapy may require dose adjustment within the recommended $14 \pm 2$ days dosing schedule during the maintenance period (up to every 12 days) when it is deemed necessary at the discretion of the Investigator; e.g., two consecutive events of elevated LDH $\geq 2 \times \text{ULN}$ after prior LDH reduction to $< 1.5 \times \text{ULN}$ on treatment. () | In case a dosing is delayed, next dosing visit date should not be altered. In case previous IP administration was out of window, next visit schedule should be adjusted to keep intervals of IP administration as indicated above. The subject receiving SB12 or Soliris® therapy may require dose adjustment within the recommended $14 \pm 2$ days dosing schedule during the maintenance period (up to every 12 days) when it is deemed necessary at the discretion of the Investigator; e.g., two consecutive events of elevated LDH $\geq 2 \times \text{ULN}$ combined with sign or symptom of intravascular haemolysis after prior LDH reduction to $< 1.5 \times \text{ULN}$ on treatment. | |
| | | () | |
| 5.2.5. Treatment Compliance and Investigation -al Product Accountabili -ty | Unless otherwise notified, empty vials and vials with residual materials should be kept for inspection and accountability by the study monitor prior to their destruction or handled per local pharmacy SOP for clinical study drugs. All unused IPs should be returned to the Sponsor or designated vendor unless local destruction site is approved by the Sponsor. If destruction is authorised at the investigational site, the Investigator must ensure that the materials are destroyed in compliance with all applicable environmental regulations, institutional policies, and any instructions provided by the Sponsor. Destruction of the IPs must be adequately documented. | Unless otherwise notified, empty vials and vials with residual materials should be kept for inspection and accountability by the study monitor prior to their destruction or handled per local pharmacy SOP for clinical study drugs. All unused IPs should be returned to the Sponsor or designated vendor unless local destruction site is approved by the Sponsor. If destruction is authorised at the investigational site, the Investigator must ensure that the materials are destroyed in compliance with all applicable environmental regulations, institutional policies, and any instructions provided by the Sponsor. Destruction of the IPs must be adequately documented. In case of expanded access of SB12 to subjects, the | To add IP accountability during additional SB12 provision |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | | Investigator is responsible for maintaining the SB12 records which include information on amounts delivered, dispensed, and returned/destroyed; for ensuring proper storage conditions are maintained and documented including details of dates, quantities, batch numbers, expiry dates; ensuring the SB12 is only used as specified by the expanded access; for reconciling all SB12 received from the Sponsor. Further details will be provided in a guideline for expanded access. | |
| 5.3.<br>Concomitant<br>Medication<br>or Treatment | All medication including both prescription and non-prescription drugs, and any procedures undertaken during the study period (from the study informed consent has been signed to EOS/early termination [ET] visit) should be recorded in the subject's source documents and eCRF. () | All medication including both prescription and non-prescription drugs, and any procedures undertaken during the study period (from the study informed consent has been signed to EOS/early termination [ET] visit) should be recorded in the subject's source documents and eCRF. () | To apply abbreviation |
| 7.1.3.<br>Treatment<br>Period | All procedures and assessments will be performed at the visits specified in Table 1 and Table 2. Samples for laboratory assessments will be collected before IP administration. () | All procedures and assessments will be performed at the visits specified in Table 1 and Table 2. Samples for laboratory assessments will be collected before IP administration on same day or up to 2 days prior, unless otherwise specified. () | To clarify the window for sample collection |
| 7.2.1.<br>Subject<br>Discontinuat<br>ion from<br>Study<br>Treatment | <ul> <li>() The Investigator should discuss with the medical monitor prior to discontinuing a subject's study treatment in case of the following criteria, but not limited to: <ul> <li>Conditions or intercurrent illness that preclude compliance with the protocol in terms of their safety or well-being</li> </ul> </li> </ul> | <ul> <li>() The Investigator should discuss with the medical monitor prior to discontinuing a subject's study treatment in case of the following criteria, but not limited to: <ul> <li>Conditions or intercurrent illness that preclude compliance with the protocol in terms of their safety or well-being</li> </ul> </li> </ul> | To clarify the meaning of lack of subject's compliance |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | <ul> <li>Lack of efficacy (e.g., C5 gene polymorphism) Note: If the LDH level is not changed after the initiation of study drug (lack of efficacy), the Investigator and medical monitor and/or Sponsor should discuss to determine how to manage this case including whether or not to perform pharmacogenetic analysis (C5 gene polymorphism). </li> <li>Unacceptable toxicity</li> <li>Lack of subject's compliance (e.g., a subject who missed two consecutive doses, lost to follow-up) Note: Before a subject is deemed lost to follow-up, the Investigator or designee will make every effort to regain contact with the subject. </li> <li>Investigator discretion or other reasons</li> <li>()</li> </ul> | <ul> <li>Lack of efficacy (e.g., C5 gene polymorphism) Note: If the LDH level is not changed after the initiation of study drug (lack of efficacy), the Investigator and medical monitor and/or Sponsor should discuss to determine how to manage this case including whether or not to perform pharmacogenetic analysis (C5 gene polymorphism). </li> <li>Unacceptable toxicity <ul> <li>Lack of subject's compliance (e.g., a subject who missed two consecutive doses, repeated delay in study treatment and lost to follow-up)</li> <li>Note: Before a subject is deemed lost to follow-up, the Investigator or designee will make every effort to regain contact with the subject.</li> <li>Investigator discretion or other reasons</li> </ul> </li> </ul> | |
| 7.2.1.<br>Subject<br>Discontinuat<br>ion from<br>Study<br>Treatment | Any subject who discontinues SB12 or Soliris® should be monitored for at least 8 weeks after last study drug to detect serious haemolysis and other reactions. If serious haemolysis occurs after SB12 or Soliris® discontinuation, consider the following procedures and/or treatments: • Blood transfusion (pRBCs) or exchange transfusion if the PNH RBCs are > 50% of the total RBCs by flow cytometry | Any subject who discontinues SB12 or Soliris® should be monitored for at least 8 weeks after last study drug to detect serious haemolysis and other reactions. If serious haemolysis occurs after SB12 or Soliris® discontinuation, consider the following procedures and/or treatments: • Blood transfusion (pRBCs) or exchange transfusion if the PNH RBCs are > 50% of the total RBCs by flow cytometry | To add the additional information for SB12 provision |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| - Anteced | <ul> <li>Anticoagulation</li> <li>Corticosteroids</li> <li>Complement inhibitors</li> </ul> | <ul> <li>Anticoagulation</li> <li>Corticosteroids</li> <li>Complement inhibitors</li> <li>According to the Investigator's medical judgement, if complement inhibitor should be administered again due to serious haemolysis and other reactions which occur within 8 weeks after completion of the study treatment with SB12 or Soliris®, the Investigator should discuss with Sponsor for an expanded access of SB12 to such subjects. Accordingly, the Sponsor will provide SB12 to those subjects as an expanded access up to 1 year period, where applicable, in accordance with relevant local regulations and/or law.</li> </ul> | |
| 8.1.2. Period of Observation for Adverse Events | () However, SAEs that are considered to be related to the IP can be collected until 10.5 weeks from the last dose of study drug (five half-lives of the study drug). SAEs that occurred after EOS visit or ET visit and that are considered to be related to the IP must be reported to the Sponsor or its designated representative using the paper SAE report form at least within 24 hours of the Investigator becoming aware of the event (see Section 8.2.2). Unresolved AEs during the study period should be followed up until the EOS and recorded in the eCRF. The Investigator should observe the AEs for appropriate medical care of the subject until AE resolution or stabilisation. () | However, SAEs must that are considered to be related to the IP can be collected until 10.5 weeks from the last dose of study drug (five half-lives of the study drug). SAEs that occurred after EOS visit or ET visit and that are considered to be related to the IP must be reported to the Sponsor or its designated representative using the paper SAE report form at least within 24 hours of the Investigator becoming aware of the event (see Section 8.2.2). Unresolved AEs during the study period should be followed up until the EOS and recorded in the eCRF. The Investigator should observe the AEs for appropriate medical care of the subject until AE resolution or stabilisation. () | To expand the collection scope of SAE from serious adverse reaction to serious adverse event. |

| 0.1.2 | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| 8.1.3. Reporting Adverse Events | Each AE is to be assessed to determine if it meets the criteria of an SAE (see Section 8.2.1 for SAE definition). If an AE is classified as an SAE, it must be reported to the Sponsor, or its designated representative, promptly according to the timeline specified in Section 8.2.2. For an SAE, a diagnosis with a description of signs and symptoms as well as other supporting information that led to the diagnosis should be described in the SAE form provided by the Sponsor (see Section 8.2.2). | Each AE is to be assessed to determine if it meets the criteria of an SAE (see Section 8.2.1 for SAE definition). If an AE is classified as an SAE, it must be reported to the Sponsor, or its designated representative, promptly according to the timeline specified in Section 8.2.2. For an SAE, a diagnosis with a description of signs and symptoms as well as other supporting information that led to the diagnosis should be described in the SAE form provided by the Sponsor (see Section 8.2.2). If the subject who received the additional SB12 provision according to Section 7.2.1 has an AE, it must be reported to the Sponsor or its designated representative using the paper AE report form. If the AE is classified as a SAE, it must be reported to Sponsor or its designated representative using the paper SAE report form at least within 24 hours of the Investigator becoming aware of the event (see Section 8.2.2). | To add the safety reporting during additional SB12 provision |
| 8.2.2.<br>Reporting<br>Serious<br>Adverse<br>Events | SAEs that occurred at or before EOS visit or ET visit must be reported to the Sponsor or its designated representative via eCRF SAE report form at least within 24 hours of the Investigator becoming aware of the event. SAEs that occurred after EOS visit or ET visit and that are considered to be related to the IP must be reported to the Sponsor or its designated representative using the paper SAE report form at least within 24 hours of the Investigator becoming aware of the event. () | SAEs must be collected until 10.5 weeks from the last dose of study drug (five half-lives of the study drug). SAEs that occurred at or before EOS visit or ET visit must be reported to the Sponsor or its designated representative via eCRF SAE report form at least within 24 hours of the Investigator becoming aware of the event. SAEs that occurred after EOS visit or ET visit and that are considered to be related to the IP must be reported to the Sponsor or its designated representative using the paper SAE report form at least within 24 hours of the Investigator becoming aware of the event. SAEs that occurred from the subject who received the | To clarify the reporting period for SAEs and add the safety reporting during additional SB12 provision |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | | additional SB12 must be reported to the Sponsor or its designated representative using the paper SAE report form at least within 24 hours of the Investigator becoming aware of the event. () | |
| 9.1.<br>Statistical<br>Hypotheses | , the treatment effect will be measured by AUEC of LDH between two different time points in each period, from Week 14 to Week 26 and from Week 40 to Week 52. The equivalence will be declared if the 90% confidence interval (CI) of the ratio between treatment effects is entirely contained within the pre-defined equivalence margin of [0.77, 1.29]. , equivalence will be declared if the 95% CI of the difference between treatments in LDH level at Week 26 is entirely contained within the pre-defined equivalence margin of [-1.2 × ULN, 1.2 × ULN] where ULN of LDH to be specified in the central laboratory specification for this study. | for those who are in favour of the AUEC of LDH, the treatment effect will be measured by AUEC of LDH between two different time points in each period, from Week 14 to Week 26 and from Week 40 to Week 52. The equivalence will be declared if the 90% confidence interval (CI) of the ratio between treatment effects is entirely contained within the predefined equivalence margin of [0.77, 1.29]. for those who are in favour of the LDH level at a single time point, equivalence will be declared if the 95% CI of the difference between treatments in LDH level at Week 26 is entirely contained within the pre-defined equivalence margin of [-1.2 × ULN, 1.2 × ULN] where ULN of LDH to be specified in the central laboratory specification for this study. | To add phrase to be consistent within the document |
| 9.5.3.<br>Pharmacokin<br>-etic<br>Analyses | PK analysis will be performed for the PKS. Serum trough concentration will be summarised with descriptive statistics by treatment sequence, period, and time point. | PK analysis will be performed for the PKS. Serum trough-<br>concentration C <sub>trough</sub> will be summarised descriptively by<br>treatment sequence, period, and time point. | To apply abbreviation |
| 13. | [10] Soliris <sup>®</sup> EPAR – Product Information. EMA (Jan 18, 2018). Retrieved Apr 25, 2018 from | [10] Soliris <sup>®</sup> EPAR – Product Information. EMA (Jan 18 Oct 24, 2018). Retrieved Apr 25 Dec 11, 2018 from | To refer the latest version of |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| References | http://www.ema.europa.eu/docs/en_GB/document_library/EPA<br>R Product_Information/human/000791/WC500054208.pdf | http://www.ema.europa.eu/docs/en_GB/document_library/E<br>PAR<br>Product_Information/human/000791/WC500054208.pdf<br>https://www.ema.europa.eu/documents/product-<br>information/soliris-epar-product-information_en.pdf | regulatory<br>document |
| All Sections | N/A | All sections were updated to follow consistent usage of punctuation. | Administrative<br>update irrelevant to<br>study design and/or<br>procedures |

## Amendment 3: Version 4.0, Nov 29, 2019

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| SYNOPSIS<br>Planned<br>Study Period | After Screening, the duration of study participation will be 60 weeks per subject including 52-week treatment period and 8-week post-treatment follow-up period. | After Screening, the duration of study participation will be 60—weeks per subject including-52-week randomised treatment period and 8-week post-treatment follow-up an extension period of up to 2 years. | To reflect the changes due to 2-year extension period |
| SYNOPSIS<br>Study<br>Design | This is a randomised Phase III, double-blind, multicentre, crossover study to compare the efficacy, safety, pharmacokinetics, and immunogenicity between SB12 and Soliris® in subjects with PNH. Subjects will be randomised in a 1:1 ratio to treatment sequence I (SB12 to Soliris®) or treatment sequence II (Soliris® to SB12). Subjects who are randomised to initially receive SB12 will be switched to receive Soliris® and subjects who are randomised to initially receive Soliris® will be switched to receive SB12 at Week 26. | This multicentre Phase III study is composed of the Main Part and Extension Part. The Main Part is a randomised Phase III, double-blind period, multicentre, cross-over study to compare the efficacy, safety, pharmacokinetics, and immunogenicity between SB12 and Soliris® in subjects with PNH. The Extension Part is an open-label, single-arm, 2-year extension period to provide SB12 in subjects with PNH for an extended duration under an ethical basis. For the Main Part, subjects Subjects will be randomised in a 1:1 ratio to treatment sequence I (SB12 to Soliris®) or treatment sequence II (Soliris® to SB12). Subjects who are randomised to initially receive SB12 will be switched to receive Soliris® and subjects who are randomised to initially receive Soliris® will be switched to receive SB12 at Week 26. End of the Main Part is defined as completion of pre-dose activities at Week 52. Subjects who complete the Main Part will enter the Extension Part. For the Extension Part, all subjects will receive SB12 for 2 years. | To reflect the changes due to 2-year extension period |
| SYNOPSIS<br>Inclusion<br>Criteria | 3. Presence of the PNH white blood cell (WBC) clone ≥ 10% by high-sensitivity flow cytometry at Screening. | 3. Presence of the PNH white blood cell (WBC) clone, with a granulocyte or monocyte clone size of ≥ 10% by high-sensitivity flow cytometry at Screening. | To clarify the inclusion criteria |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| SYNOPSIS<br>Exclusion<br>Criteria | <ul> <li>4. Abnormal haematological parameters at Screening defined as the following:</li> <li>a. Absolute neutrophil count (ANC) ≤ 500/mm³</li> <li>b. Platelet count &lt; 70,000/mm³</li> </ul> | <ul> <li>4. Abnormal haematological parameters at Screening defined as the following:</li> <li>a. Absolute neutrophil count (ANC) ≤ 500/mm³ 0.5 × 10³/μL</li> <li>b. Platelet count &lt; 70,000/mm³ 70 × 10³/μL</li> </ul> | To change the unit of haematology parameters |
| SYNOPSIS<br>Exclusion<br>Criteria | 6. History of bone marrow transplantation. | 6. History of bone marrow haematopoietic stem cell transplantation. | To clarify the exculsion criteria |
| SYNOPSIS<br>Exclusion<br>Criteria | <ul> <li>10. Concomitant use of any of the following medications is prohibited if the following conditions apply.</li> <li>b. Warfarin with an unstable international normalized ratio (INR) for at least 4 weeks prior to initiation of study drug (Day 1).</li> </ul> | <ul> <li>10. Concomitant use of any of the following medications is prohibited if the following conditions apply.</li> <li>b. Warfarin with an unstable international normalized normalised ratio (INR) for at least 4 weeks prior to initiation of study drug (Day 1) at the discretion of the Investigator.</li> </ul> | To clarify the exculsion criteria |
| SYNOPSIS<br>Investigation<br>-al Products | • Dose regimen: 600 mg every 7 days for the first 4 weeks (initial phase) and 900 mg for the fifth week, followed by 900 mg every 14 ± 2 days until Week 52 (maintenance phase). | • Dose regimen: 600 mg every 7 days for the first 4 weeks (initial phase) and 900 mg for the fifth week, followed by 900 mg every 14 ± 2 days until Week 52, thereafter (maintenance phase). | To reflect the changes due to 2-year extension period |
| SYNOPSIS<br>Main<br>Criteria for<br>Evaluation | <ul> <li>Primary endpoints</li> <li>LDH level (U/L) at Week 26</li> <li>Area under the effect curve (AUEC) of LDH from Week 14 to Week 26 and from Week 40 to Week 52</li> </ul> | <ul> <li>Primary endpoints</li> <li>LDH level (U/L) at Week 26</li> <li>Area-Time-adjusted area under the effect curve (AUEC) of LDH from Week 14 to Week 26 and from Week 40 to Week 52</li> </ul> | To clarify the primary endpoint |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| SYNOPSIS | Secondary endpoints | Secondary endpoints | To reflect the |
| Main<br>Criteria for<br>Evaluation | Efficacy endpoints • LDH profile over time • Number of units of pRBCs transfused throughout the study duration for each period Safety endpoints • Incidence of adverse events (AEs) and serious AEs (SAEs) • Incidence of infection-related AEs • Meningococcal infection • Other systemic infections • Incidence of infusion-related reactions (IRRs) () Immunogenicity endpoints • Incidence of anti-drug antibodies (ADAs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and end of study (EOS)/early termination (ET) • Incidence of neutralising antibodies (NAbs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and EOS/ET | <ul> <li>Efficacy endpoints</li> <li>LDH profile over time during the Main Part</li> <li>Number of units of pRBCs transfused throughout the study duration for each period during the Main Part</li> <li>Safety endpoints</li> <li>Incidence of adverse events (AEs) and serious AEs (SAEs)</li> <li>Incidence of serious AEs (SAEs)</li> <li>Incidence of infection-related AEs</li> <li>Meningococcal infection</li> <li>Other systemic infections</li> <li>Incidence of infusion-related reactions (IRRs)</li> <li>()</li> <li>During the Extension Part, only SAEs will be collected.</li> <li>Immunogenicity endpoints</li> <li>Incidence of anti-drug antibodies (ADAs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and end of study (EOS)/early termination (ET)</li> <li>Incidence of neutralising antibodies (NAbs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and EOS/ET</li> </ul> | changes in secondary endpoints due to 2-year extension period |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| SYNOPSIS<br>Statistical<br>Methods | for those who are in favour of the AUEC of LDH, the primary efficacy analysis will be performed for the PPS-AUEC using a linear mixed model with treatment, subject, sequence, and period as fixed effects and, subject nested within sequence as a random effect. The analysis will be performed with logetransformed AUEC of LDH estimating the difference in least squares means and its 90% confidence interval (CI), and back transformation of those values will provide the ratio of geometric means and 90% CI. The equivalence will be declared if the two-sided 90% CI of the ratio of geometric means in AUEC of LDH between SB12 and Soliris® lies within the predefined equivalence margin of [0.77, 1.29]. for those who are in favour of the LDH level at a single time point, the primary efficacy analysis will be performed for the PPS-single using a linear mixed model with treatment as a fixed effect. () () As a secondary efficacy endpoint, the number of units of pRBCs transfused will be analysed using Wilcoxon rank-sum test for each period. And mean LDH profile will be presented over time. Safety analyses Safety analyses will be performed for the Safety Set (SAF). | for those who are in favour of the time-adjusted AUEC of LDH, the primary efficacy analysis will be performed for the PPS-AUEC using a linear mixed model with treatment, subject, sequence, and period, and gender as fixed effects, and subject nested within sequence as a random effect. The analysis will be performed with loge-transformed time-adjusted AUEC of LDH estimating the difference in least squares means and its 90% confidence interval (CI), and back transformation of those values will provide the ratio of geometric means and 90% CI. The equivalence will be declared if the two-sided 90% CI of the ratio of geometric means in time-adjusted AUEC of LDH between SB12 and Soliris® lies within the pre-defined equivalence margin of [0.77, 1.29]. Or those who are in favour of the LDH level at a single time point, the primary efficacy analysis will be performed for the PPS-single using a linear mixed model with treatment, and gender as a fixed effect. () If normal range of LDH is gender specific, the smaller/smallest ULN will be used for the equivalence margin; otherwise ULN is not gender specific, unified ULN will be used for the equivalence margin. () | To clarify the primary endpoint and efficacy/safety analysis To reflect the local amendment To reflect changes in the statistical methods due to 2-year extension period |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | All reported terms for AEs will be coded using the latest version of Medical Dictionary for Regulatory Activities (MedDRA®). AEs will be collected and classified according to National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) v5.0. All AE data will be summarised by count and percentage of subjects experiencing events by system organ class, preferred term, treatment sequence, and period. () | As a secondary efficacy endpoint, the number of units of pRBCs transfused during the Main Part will be analysed using Wilcoxon rank-sum test for each period. And mean LDH profile during the Main Part will be presented over time. Safety analyses Safety analyses will be performed for in the Safety Set (SAF) for the Main Part (SAF1) and Safety Set for the Extension Part (SAF2). | |
| | Changes in vital signs and clinical laboratory parameters will be summarised descriptively by treatment sequence, period, and time point. () Immunogenicity analyses The immunogenicity analyses will be performed for the SAF. ADA and NAb results will be summarised with count and percentage by treatment sequence, period, and time point. The incidence of overall ADA will be summarised by treatment sequence and period. | All reported terms for AEs will be coded using the latest version of Medical Dictionary for Regulatory Activities (MedDRA®). AEs will be collected and classified according to National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) v5.0. All AE data reported during the Main Part will be summarised by count and percentage of subjects experiencing events by system organ class, preferred term, treatment sequence, and period for the SAF1. () | |
| | Sample size () | Changes in vital signs and clinical laboratory parameters will be summarised descriptively by treatment sequence, period, and time point <b>for the SAF1</b> . () | |
| | For calculation of the equivalence margin for AUEC of LDH, mean and coefficient of variation (%CV) were referred from TRIUMPH study. The mean (%CV) of AUEC of LDH at Week 26 is 81140.0 U/L × day (142.45%) and 429874.1 U/L × day (33.49%) for eculizumab and non-eculizumab arms, respectively. | All SAEs reported during the Extension Part will be summarised by count and percentage of subjects experiencing events by system organ class and preferred term for the SAF2. Immunogenicity analyses | |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | From the results in the reference study, mean ratio of AUEC of LDH is estimated to be 0.19 with a 90% CI [0.1308, 0.2724]. The upper limit of the equivalence margin is calculated as where it preserves at least of eculizumab treatment effect over the placebo, but the equivalence margin will be [0.77, 1.29] for the comparison with the 90% CI of mean ratio of AUEC of LDH. () | The immunogenicity analyses will be performed for the SAF SAF1. ADA and NAb results will be summarised with count and percentage by treatment sequence, period, and time point. The incidence of overall ADA will be summarised by treatment sequence and period. Sample size () For calculation of the equivalence margin for time-adjusted AUEC of LDH, mean and coefficient of variation (%CV) were referred from TRIUMPH study. The mean (%CV) of AUEC of LDH at Week 26 is 81140.0 U/L × day (142.45%) and 429874.1 U/L × day (33.49%) for eculizumab and non-eculizumab arms, respectively. | |
| | | From the results in the reference study, mean ratio of AUEC of LDH is estimated to be 0.19 with a 90% CI [0.1308, 0.2724]. The upper limit of the equivalence margin is calculated as where it preserves at least equivalence margin will be [0.77, 1.29] for the comparison with the 90% CI of mean ratio of time-adjusted AUEC of LDH. () | |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| Figure 1 | Sequence (a=25) SB12 Soliris | Sequence I (n=25) SB12 Soliris* | To reflect the changes due to 2-year extension period |
| Figure 1<br>Footnote | <ul> <li>® = Randomisation; AUEC = Area under the Effect Curve; EOS = End of Study; PNH = Paroxysmal Nocturnal Haemoglobinuria; W = Week</li> <li>c. From Week 4, 900 mg of SB12 or Soliris® every 14 ± 2 days up to Week 52 ()</li> <li>f. EOS visit is defined as 8 weeks after the last dose of SB12 or Soliris®.</li> </ul> | <ul> <li>Randomisation; AUEC = Area under the Effect Curve; EOS = End of Study; n = No. of Subjects; PNH = Paroxysmal Nocturnal Haemoglobinuria; W = Week</li> <li>From Week 4, 900 mg of SB12 or Soliris® every 14 ± 2 days up to Week 52-50. During the Extension Part, SB12 will be given to all subjects.</li> <li>EOS visit Completion of pre-dose activities at Week 52 is defined as end of the Main Part 8 weeks after the last dose of SB12 or Soliris®.</li> <li>EOS is defined as the date of last subject's last visit in the Extension Part.</li> </ul> | To add abbreviations To reflect the changes due to 2-year extension period |
| Table 1 | Table 1. Schedule of Activities (Period 1, before Cross-over) | Table 1. Schedule of Activities (Main Part: Period 1, before Cross-over) | To reflect the changes due to 2-year extension period |
| Table 1<br>Footnote | 4. All screening procedures must be completed and reviewed within 42 days prior to randomisation. All eligibility criteria must be reviewed and confirmed prior to randomisation. The initiation of study drug (Day 1) should be done within 21 days of randomisation. | 4. All screening procedures must be completed and reviewed within 42 days prior to randomisation. All eligibility criteria not dependent on Day 1 must be reviewed and confirmed prior to randomisation. The initiation of study drug (Day 1) should be done within 21 days of randomisation. Eligibility criteria that are dependent on | To clarify the randomisation process including eligibility confirmation process |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | | Day 1 should be checked at Day 1 and if found in violation then should be withdrawn according to discontinuation criteria. | |
| Table 1<br>Footnote | 7. Females of childbearing potential only. Serum pregnancy test at Screening and EOS (or 8 weeks after the last dose of study drug in case of early termination [ET]); urine pregnancy test at other applicable visits. | 7. Females of childbearing potential only. Serum pregnancy test at Screening and EOS (or 8 weeks after the last dose of study drug in case of early termination [ET]) (ET) during the Main Part; urine pregnancy test at other applicable visits before study drug administration. | To reflect the changes due to 2-year extension period and clarify the timeframe |
| Table 1<br>Footnote | 10. LDH will be measured at pre-dose on each visit and will also be measured throughout the study period if the suspected sign or symptom of breakthrough haemolysis occurs. | 10. LDH will be measured at pre-dose on each visit and will also be measured <b>throughout the study period</b> if the suspected sign or symptom of breakthrough haemolysis occurs. | To reflect the changes due to 2-year extension period |
| Table 1<br>Footnote | 11. Parameters included in haematology test are WBC count, RBC count, haemoglobin, haematocrit, platelet count, differential WBC count, and nucleated RBC. () | 11. Parameters included in haematology test are WBC count, RBC count, haemoglobin, haematocrit, platelet count, differential WBC count, and nucleated RBC, mean corpuscular haemoglobin (MCH), mean corpuscular haemoglobin concentration (MCHC), mean corpuscular volume (MCV), mean platelet volume (MPV), and red cell distribution width (RDW). () | To add several haematology parameters |
| Table 1<br>Footnote | 12. Blood sample for PK analysis will be taken prior to dosing at Weeks 0, 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, and 52. Blood samples should be collected at the same day of study drug administration. If the administration of IPs is delayed for any reasons after predose blood sampling for PK analysis, blood sample should be re-collected on actual dosing day and be used for analysis. PK samples will also be collected throughout the | 12. Blood sample for PK analysis will be taken prior to dosing at Weeks 0, 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, and 52. Blood samples should be collected at the same day of study drug administration. If the administration of IPs is delayed for any reasons after pre-dose blood sampling for PK analysis, blood sample should be recollected on actual dosing day and be used | To reflect the changes due to 2-year extension period |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | study period if the suspected sign or symptom of breakthrough haemolysis occurs. | for analysis. PK samples will also be collected throughout the study period if the suspected sign or symptom of breakthrough haemolysis occurs. | |
| Table 1<br>Footnote | 13. Blood sample for PD (terminal complement activity) analysis will be taken prior to dosing at Weeks 0, 2, 4, 6, 10, 14, 26, 28, 30, 32, 36, 40, and 52. Blood samples should be collected at the same day of study drug administration. If the administration of IPs is delayed for any reasons after pre-dose blood sampling for PD analysis, blood sample should be re-collected on actual dosing day and be used for analysis. PD samples will also be collected throughout the study period if the suspected sign or symptom of breakthrough haemolysis occurs. | 13. Blood sample for PD (terminal complement activity) analysis will be taken prior to dosing at Weeks 0, 2, 4, 6, 10, 14, 26, 28, 30, 32, 36, 40, and 52. Blood samples should be collected at the same day of study drug administration. If the administration of IPs is delayed for any reasons after pre-dose blood sampling for PD analysis, blood sample should be re-collected on actual dosing day and be used for analysis. PD samples will also be collected throughout the study period if the suspected sign or symptom of breakthrough haemolysis occurs. | To reflect the changes due to 2-year extension period |
| Table 1<br>Footnote | 14. Blood sample for immunogenicity assay will be taken prior to dosing at Weeks 0, 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and EOS/ET. Blood samples should be collected at the same day of study drug administration except for EOS/ET. If the administration of IPs is delayed for any reasons after pre-dose blood sampling for immunogenicity assay, blood sample should be recollected on actual dosing day and be used for analysis. | 14. Blood sample for immunogenicity assay will be taken prior to dosing at Weeks 0, 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and EOS/ET. Blood samples should be collected at the same day of study drug administration except for EOS/ET visit. If the administration of IPs is delayed for any reasons after pre-dose blood sampling for immunogenicity assay, blood sample should be re-collected on actual dosing day and be used for analysis. | To reflect the changes due to 2-year extension period |
| Table 1<br>Footnote | 19. Adverse events (AEs) will be collected from the time of signing the informed consent until EOS (or 8 weeks after the last dose of study drug in case of ET). | 19. Adverse events (AEs) will be collected from the time of signing the informed consent until EOS end of the Main Part (or 8 weeks after the last dose of study drug in case of ET during the Main Part). | To reflect the changes due to 2-year extension period |

| Section<br>Affected | Origi | nal Content | Amende | d/New | Content | Rationale |
|---|---|---|---|---|---|---|
| Table 1<br>Footnote | 20. Previous medications (vexcept immunosuppress immunosuppressant) with medications will be reco | to Screen<br>weeks pri<br>immunos<br>concomit<br>throughe<br>the Main | ing exc<br>ior to So<br>uppress<br>ant med<br>out the<br>Part (<br>tudy di | tions (within 4 weeks prior ept immunosuppressant, 8 creening for sant) will be recorded and dications will be recorded study period until end of or 8 weeks after the last rug in case of ET during | To reflect the changes due to 2-year extension period | |
| Table 1<br>Footnote | | be collected from the time of nsent until EOS (or 8 weeks after ug in case of ET). | 21. Transfusion record will signing the informed core Part (or 8 weeks after the ET during the Main Part Part (or 8 weeks after the ET during the Main Part | To reflect the changes due to 2-year extension period | | |
| Table 2 | Table 2. Schedule of Activitie Cross-over) | es (Period 2 and EOS/ET, after | OS/ET, after Table 2. Schedule of Activities (Main Part: Period 2 and EOS/ET, after Cross-over) | | | |
| Table 2 | Assessments | Study Period | Assessments | | Study Period | To reflect the |
| | Study Visit | 29 EOS/ET <sup>20</sup> | Study Visit | 29 | EOS/ET <sup>20</sup> ET <sup>21</sup> | changes due to 2- |
| | Week Day (± Visit Window) | 52 60<br>365<br>(±2) 421 (±7) | Week | 52 <sup>20</sup> | 60<br>8 (±1) weeks after the<br>last dose of study drug | year extension period |
| | IP administration <sup>15</sup> | ✓ | Day (± Visit Window) | 365<br>(±2) | 4 <del>21 (±7)</del> | |
| Table 2<br>Footnote | EOS = End of Study; | | IP administration <sup>15</sup> EOS = End of Study; | + | | To reflect the changes due to 2-year extension period |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| Table 2<br>Footnote | 4. Females of childbearing potential only. Serum pregnancy test at Screening and EOS (or 8 weeks after the last dose of study drug in case of ET); urine pregnancy test at other applicable visits. | 4. Females of childbearing potential only. Serum pregnancy test at Screening and EOS (or 8 weeks after the last dose of study drug in case of ET) during the Main Part; urine pregnancy test at other applicable visits before study drug administration. | To reflect the changes due to 2-year extension period and clarify the timeframe |
| Table 2<br>Footnote | 7. LDH will be measured at pre-dose on each visit and will also be measured throughout the study period if the suspected sign or symptom of breakthrough haemolysis occurs. | 7. LDH will be measured at pre-dose on each visit and will also be measured <b>throughout the study period</b> if the suspected sign or symptom of breakthrough haemolysis occurs. | To reflect the changes due to 2-year extension period |
| Table 2<br>Footnote | 8. Parameters included in haematology test are WBC count, RBC count, haemoglobin, haematocrit, platelet count, differential WBC count, and nucleated RBC. () | 8. Parameters included in haematology test are WBC count, RBC count, haemoglobin, haematocrit, platelet count, differential WBC count, and nucleated RBC, MCH, MCHC, MCV, MPV, and RDW. () | To add several<br>haematology<br>parameters |
| Table 2 Footnote | 9. Blood sample for PK analysis will be taken prior to dosing at Weeks 0, 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, and 52. Blood samples should be collected at the same day of study drug administration. If the administration of IPs is delayed for any reasons after predose blood sampling for PK analysis, blood sample should be re-collected on actual dosing day and be used for analysis. PK samples will also be collected throughout the study period if the suspected sign or symptom of breakthrough haemolysis occurs. | 9. Blood sample for PK analysis will be taken prior to dosing at Weeks 0, 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, and 52. Blood samples should be collected at the same day of study drug administration. If the administration of IPs is delayed for any reasons after pre-dose blood sampling for PK analysis, blood sample should be recollected on actual dosing day and be used for analysis. PK samples will also be collected throughout the study period if the suspected sign or symptom of breakthrough haemolysis occurs. | To reflect the changes due to 2-year extension period |
| Table 2<br>Footnote | 10. Blood sample for PD (terminal complement activity) analysis will be taken prior to dosing at Weeks 0, 2, 4, 6, 10, 14, 26, 28, 30, 32, 36, 40, and 52. Blood samples should be collected at the same day of study drug administration. If the administration of IPs is delayed for | 10. Blood sample for PD (terminal complement activity) analysis will be taken prior to dosing at Weeks 0, 2, 4, 6, 10, 14, 26, 28, 30, 32, 36, 40, and 52. Blood samples should be collected at the same day of study drug | To reflect the changes due to 2-year extension period |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | any reasons after pre-dose blood sampling for PD analysis, blood sample should be re-collected on actual dosing day and be used for analysis. PD samples will also be collected throughout the study period if the suspected sign or symptom of breakthrough haemolysis occurs. | administration. If the administration of IPs is delayed for any reasons after pre-dose blood sampling for PD analysis, blood sample should be re-collected on actual dosing day and be used for analysis. PD samples will also be collected throughout the study period if the suspected sign or symptom of breakthrough haemolysis occurs. | |
| Table 2<br>Footnote | 11. Blood sample for immunogenicity assay will be taken prior to dosing at Weeks 0, 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and EOS/ET. Blood samples should be collected at the same day of study drug administration except for EOS/ET. If the administration of IPs is delayed for any reasons after pre-dose blood sampling for immunogenicity assay, blood sample should be recollected on actual dosing day and be used for analysis. | 11. Blood sample for immunogenicity assay will be taken prior to dosing at Weeks 0, 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and EOS/ET. Blood samples should be collected at the same day of study drug administration except for EOS/ET visit. If the administration of IPs is delayed for any reasons after pre-dose blood sampling for immunogenicity assay, blood sample should be re-collected on actual dosing day and be used for analysis. | To reflect the changes due to 2-year extension period |
| Table 2<br>Footnote | 17. Adverse events (AEs) will be collected from the time of signing the informed consent until EOS (or 8 weeks after the last dose of study drug in case of ET). | 17. Adverse events (AEs) will be collected from the time of signing the informed consent until EOS end of the Main Part (or 8 weeks after the last dose of study drug in case of ET during the Main Part). | To reflect the changes due to 2-year extension period |
| Table 2<br>Footnote | 18. Concomitant medications will be recorded throughout the study period. | 18. Concomitant medications will be recorded throughout the study period until end of the Main Part (or 8 weeks after the last dose of study drug in case of ET during the Main Part). | To reflect the changes due to 2-year extension period |
| Table 2<br>Footnote | 19. Transfusion record will be collected from the time of signing the informed consent until EOS (or 8 weeks after the last dose of study drug in case of ET). | 19. Transfusion record will be collected from the time of signing the informed consent until EOS end of the Main Part (or 8 weeks after the last dose of study drug in case of ET during the Main Part). | To reflect the changes due to 2-year extension period |

| Section<br>Affected | | Original Content | | | Amendo | ed/New Content | | Rationale |
|---|---|---|---|---|---|---|---|---|
| Table 2<br>Footnote | - | or ET visit is defined as 8 weeks after the last 312 or Soliris <sup>®</sup> . | | 20 | <del>after the</del><br>End of t | it or ET visit is de<br>last dose of SB12<br>he Main Part is d<br>ion of pre-dose ac | <del>l or Soliris<sup>®</sup></del><br>efined as | To reflect the changes due to 2-year extension period |
| Table 2<br>Footnote | N/A | | 21. | | | 8 weeks after the<br>y be up to Week 5 | | To reflect the changes due to 2-year extension period |
| Table 3 | N/A | | SB12 adm | | Part: 2-year Extension Period eeks 52" 540 560 580 V 0 V 0 V 0 V 0 | Study Period 50 62 64 140 142 142 143 144 145 145 146 147 148 148 | 144 148 150 152 154 Extension | To reflect the changes due to 2-year extension period |
| Table 3<br>Footnote | N/A | | 1.<br>2.<br>3. | IV infusion<br>Only SAEs<br>from start<br>End of the<br>the last do<br>subjects do | for 35 ± 1<br>s will be col<br>of study tro<br>Extension<br>se of SB12. | will be administer of minutes for all sometiment at Week sometiment at Week sometimed as Prematurely discretany specific sture. | ubjects.<br>Extension Part<br>52.<br>8 weeks after<br>ontinued | To reflect the changes due to 2-year extension period |
| LIST OF<br>ABBREVIA<br>-TIONS | IB INR N/A SAF | Investigators' Brochure International normalized ratio N/A Safety Set | | R<br>CH<br>CHC | Internation | ors <sup>2</sup> Investigator <sup>2</sup> al <del>normalized</del> not ouscular haemogl corpuscular | malised ratio | To revise/add<br>abbreviations<br>according to<br>updated contents |
| | | | M | CV | | ouscular volume | | |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | | MFDS Ministry of Food and Drug Safety MPV Mean platelet volume NMOSD Neuromyelitis optica spectrum disorder RDW Red cell distribution width SAF1 Safety Set for the Main Part SAF2 Safety Set for the Extension Part | |
| LIST OF<br>STUDY<br>STAFF | Sponsor: Samsung Bioepis Co., Ltd. 107, Cheomdan-daero, Yeonsu-gu, Incheon, 21987 Republic of Korea Tel: +82 (32) 455 3114 Fax: +82 (32) 455 6799 Clinical Development Lead Statistician | Sponsor: Samsung Bioepis Co., Ltd. 107, Cheomdan-daero, Yeonsu-gu, Incheon, 21987 Republic of Korea Tel: +82 (32) 455 6114 3114 Fax: +82 (32) 455 6799 Clinical Development Lead Statistician | Administrative change |
| 1.1. Paroxysmal Nocturnal Haemoglobi- | () Soliris® (eculizumab, Alexion Pharmaceuticals, Inc.) is a humanised monoclonal antibody that blocks terminal | () Soliris® (eculizumab, Alexion Pharmaceuticals, Inc.) is a humanised monoclonal antibody that blocks terminal | To refer the latest information |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| nuria | complement by binding to C5 and is the only approved therapy for PNH. | complement by binding to C5 and is the <b>only</b> approved therapy for PNH. | |
| 1.2.<br>Overview of<br>SB12 | SB12 has been developed as a similar biological medicinal product to Soliris® (eculizumab, Alexion Pharmaceuticals, Inc.). Soliris® is currently indicated for the treatment of patients with PNH, atypical haemolytic uremic syndrome (aHUS), and refractory generalised myasthenia gravis (gMG) [10]. () | SB12 has been developed as a similar biological medicinal product to Soliris® (eculizumab, Alexion Pharmaceuticals, Inc.). Soliris® is currently indicated for the treatment of patients with PNH, atypical haemolytic uremic syndrome (aHUS), and refractory generalised myasthenia gravis (gMG), and neuromyelitis optica spectrum disorder (NMOSD) [10; 21]. () | To refer the latest<br>version of<br>regulatory<br>document |
| 1.2.2.<br>Clinical<br>Pharmacolog<br>-y of SB12 | As clinical studies using SB12 have not been conducted up to date, clinical data is currently not available. Based on biosimilarity between SB12 and Soliris®, which was demonstrated through extensive quality and non-clinical similarity exercise, a Phase I study will be conducted in healthy subjects to compare the pharmacokinetic (PK), safety, tolerability, immunogenicity, and pharmacodynamic (PD) profiles and a Phase III study will be conducted in subjects with PNH to compare the efficacy, safety, pharmacokinetics, and immunogenicity of SB12 to Soliris®. Information on the safety of SB12 based on the product information of Soliris® and non-clinical exercise is presented in the Investigators' Brochure (IB). The safety results of the Phase I study will be updated when the results become available. | As clinical studies using SB12 have not been conducted up to date, clinical data is currently not available. Based on biosimilarity between SB12 and Soliris®, which was demonstrated through extensive quality and non-clinical similarity exercise, a Phase I study will be was conducted in healthy subjects to compare the pharmacokinetic (PK), safety, tolerability, immunogenicity, and pharmacodynamic (PD) profiles and a Phase III study will be conducted in subjects with PNH to compare the efficacy, safety, pharmacokinetics, and immunogenicity of SB12 to Soliris®. Information on the safety of SB12 based on the product information of Soliris® and, non-clinical, and clinical exercise is presented in the Investigators' Investigator's Brochure (IB). The safety results of the Phase I study will be updated when the results become available. | To reflect updated study progress (Phase I study completion) |
| 1.3.2.<br>Clinical Data<br>of Soliris® | In 40 patients with PNH, a 1-compartmental model was used to estimate PK parameters after multiple doses. Mean clearance was $0.31 \pm 0.12$ mL/hr/kg, mean volume of distribution was $110.3 \pm 17.9$ mL/kg, and mean elimination half-life was $11.3 \pm 3.4$ days. Based on these data, the onset of steady state is predicted to be approximately 49-56 days. | In 40 patients with PNH, a 1-compartmental model was used to estimate PK parameters after multiple doses. Mean clearance was $0.31 \pm 0.12$ mL/hr/kg, mean volume of distribution was $110.3 \pm 17.9$ mL/kg, and mean elimination half-life was $11.3 \pm 3.4$ days-Based on these data, the onset of The steady state is predicted to be approximately 49-56 days achieved by 4 weeks using the | To refer the latest<br>version of<br>regulatory<br>document |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| 1.5.1.<br>Known<br>Potential<br>Risks | According to Soliris® Summary of Product Characteristics (SmPC) [10], supportive safety data were collected from 29 completed and one ongoing clinical studies that included 1,407 patients exposed to eculizumab in ten disease populations, including PNH, aHUS, and refractory gMG. () () () Subjects will have a safety follow-up at the end of study (EOS) visit 8 weeks after the last dose of study drug. An independent Data and Safety Monitoring Board (DSMB) will convene at pre-specified intervals to conduct interim monitoring of accumulating safety data. Following each data review, the DSMB will make recommendations regarding the conduct of the study, including continuation of the study without modifications, termination of the study for safety reasons, or modification of the study design for safety reasons. | PNH adult dosing regimen. () According to Soliris® Summary of Product Characteristics (SmPC) [10], supportive safety data were collected from 29 30 completed and one ongoing clinical studies that included 1,407 1,503 patients exposed to eculizumab in ten complementmedicated disease populations, including PNH, aHUS, and refractory gMG, and NMOSD. () () () Subjects will have a safety follow-up at the end of study (EOS) visit until 8 weeks after the last dose of study drug. An independent Data and Safety Monitoring Board (DSMB) will convene at pre-specified intervals to conduct interim monitoring of accumulating safety data. Following each data review, the DSMB will make recommendations regarding the conduct of the study, including continuation of the study without modifications, modification of the protocol, pausing of subject enrolment until the resolution of issues, or termination of the study for safety reasons, or modification of the study design for safety reasons. | To refer the latest version of regulatory document To reflect the changes due to 2-year extension period To further clarify the DSMB actions |
| 1.5.2.<br>Known<br>Potential<br>Benefits | Soliris® is the only approved therapy for PNH and is indicated for the treatment patients with aHUS and gMG [10]. The drug is highly effective in stopping intravascular haemolysis, eliminating or decreasing the need for RBC transfusions, improving quality of life, and reducing the risk of thrombosis, the leading cause of mortality from PNH [7; 8; 9]. () | Soliris <sup>®</sup> is the <b>only</b> approved therapy for PNH and is indicated for the treatment patients with aHUS, <b>and</b> gMG, <b>and NMOSD</b> [10; 21]. The drug is highly effective in stopping intravascular haemolysis, eliminating or decreasing the need for RBC transfusions, improving quality of life, and reducing the risk of thrombosis, the leading cause of mortality from PNH [7; 8; 9]. | To refer the latest<br>version of<br>regulatory<br>document |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| 2.2.1.<br>Primary<br>Endpoints | <ul> <li>Primary endpoints</li> <li>LDH level (U/L) at Week 26</li> <li>Area under the effect curve (AUEC) of LDH from Week 14 to Week 26 and from Week 40 to Week 52</li> </ul> | <ul> <li>Primary endpoints</li> <li>LDH level (U/L) at Week 26</li> <li>Area Time-adjusted area under the effect curve (AUEC) of LDH from Week 14 to Week 26 and from Week 40 to Week 52</li> </ul> | To clarify the primary endpoint |
| 2.2.2.<br>Secondary<br>Endpoints | Secondary endpoints Efficacy endpoints LDH profile over time Number of units of pRBCs transfused throughout the study duration for each period Safety endpoints Incidence of AEs and serious AEs (SAEs) Incidence of infection-related AEs Meningococcal infection Other systemic infections Incidence of infusion-related reactions (IRRs) Immunogenicity endpoints Incidence of anti-drug antibodies (ADAs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and EOS/early termination (ET) Incidence of neutralising antibodies (NAbs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and EOS/ET | Secondary endpoints Efficacy endpoints LDH profile over time during the Main Part Number of units of pRBCs transfused throughout the study duration for each period during the Main Part Safety endpoints Incidence of AEs and serious AEs (SAEs) Incidence of serious AEs (SAEs) Incidence of infection-related AEs Meningococcal infection Other systemic infections Incidence of infusion-related reactions (IRRs) () During the Extension Part, only SAEs will be collected. Immunogenicity endpoints Incidence of anti-drug antibodies (ADAs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and EOS/early termination (ET) | To reflect the changes in secondary endpoints due to 2-year extension period |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | | • Incidence of neutralising antibodies (NAbs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and <b>EOS/</b> ET | |
| 3.1.<br>Overview of<br>Study<br>Design | This is a randomised Phase III, double-blind, multicentre, cross- over study to compare the efficacy, safety, pharmacokinetics, and immunogenicity between SB12 and Soliris® in subjects with PNH. () IPs will be given until Week 52. Details of assessment that will be conducted and treatment that will be administered are presented in Table 1 and Table 2. The last assessment will be done at Week 60 or 8 weeks after the last dose of study drug. | This multicentre Phase III study is composed of the Main Part and Extension Part. The Main Part is a randomised Phase III, double-blind period, multicentre, cross over study to compare the efficacy, safety, pharmacokinetics, and immunogenicity between SB12 and Soliris® in subjects with PNH. The Extension Part is an openlabel, single-arm, 2-year extension period to provide SB12 in subjects with PNH for an extended duration under an ethical basis. () IPs SB12 or Soliris® will be given until Week 52 50. End of the Main Part is defined as completion of pre-dose activities at Week 52. Subjects who complete the Main Part will enter the Extension Part. For the Extension Part, all subjects will receive SB12 for 2 years. Details of assessment that will be conducted and treatment that will be administered are presented in Table 1, and Table 2, and Table 3. The last assessment for the Main Part will be done performed at pre-dose of Week 60 52 or 8 weeks after the last dose of study drug in case of ET during the Main Part. The last assessment for the Extension Part will be performed at 8 weeks after the last dose of SB12. | To reflect the changes due to 2-year extension period |
| 3.2.1.<br>Scientific<br>Rationale for | () | () , for | To clarify the primary endpoint and reflect the |
| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| Study<br>Design | analysis of haemolysis reduction as measured by AUEC of LDH between two different time points in each period, the primary objective is to demonstrate comparable clinical efficacy of SB12 and Soliris® in terms of AUEC of LDH from Week 14 to Week 26 and from Week 40 to Week 52. , for analysis of haemolysis reduction as measured by the LDH level at single time point, the primary objective is to demonstrate comparable clinical efficacy of SB12 and Soliris® in terms of the LDH level | analysis of haemolysis reduction as measured by <b>time-adjusted</b> AUEC of LDH between two different time points in each period, the primary objective is to demonstrate comparable clinical efficacy of SB12 and Soliris® in terms of <b>time-adjusted</b> AUEC of LDH from Week 14 to Week 26 and from Week 40 to Week 52. s, for analysis of haemolysis reduction as measured by the LDH level at single | local amendment |
| | (U/L) at Week 26. | time point, the primary objective is to demonstrate comparable clinical efficacy of SB12 and Soliris® in terms of the LDH level (U/L) at Week 26. | |
| 3.2.3.<br>Rationale for<br>Pharmacokin<br>-etic<br>Assessments | A randomised, three-arm, parallel, single-dose Phase I PK study will be conducted in healthy subjects to demonstrate similarity in PK profiles of SB12, European Union (EU) sourced Soliris®, and US sourced Soliris®. However, since target-mediated clearance of eculizumab can be more accurately investigated in patients, additional PK assessments will be performed in this Phase III study to provide supportive evidence to PK similarity. | A randomised, three-arm, parallel, single-dose Phase I PK study will be was conducted in healthy subjects to demonstrate similarity in PK profiles of SB12, European Union (EU) sourced Soliris®, and US sourced Soliris®. However, since target-mediated clearance of eculizumab can be more accurately investigated in patients, additional PK assessments will be performed in this Phase III study to provide supportive evidence to PK similarity. | To reflect updated<br>study progress<br>(Phase I study<br>completion) |
| 3.3. Duration<br>of Study<br>Participation | After Screening, the duration of study participation will be 60 weeks per subject including 52-week treatment period and 8-week post-treatment follow-up period | After Screening, the duration of study participation will be 60—weeks per subject including-52-week randomised treatment period and 8-week post-treatment follow-up an extension period of up to 2 years. | To reflect the changes due to 2-year extension period |
| 3.5. End of<br>Study<br>Definition | A subject is considered to have completed the study if he or she has completed all study treatment including the last visit or the last scheduled procedure shown in Table 2. The EOS is defined as completion of the last scheduled visit shown in Table 2. The | A subject is considered to have completed the <b>each part of</b> study if he or she has completed all study treatment including the last visit or the last scheduled procedure shown in Table 2 and Table 3. The EOS is defined as completion of the last | To reflect the changes due to 2-year extension period |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | end of this clinical study is defined as completion of the last subject's EOS. | scheduled visit shown in Table 2. The end of this clinical study the Main Part is defined as completion of the last subject's EOS pre-dose activities at Week 52 for subjects. The end of the Extension Part is defined as 8 weeks after the last dose of SB12. The end of study (EOS) is defined as the date of last subject's last visit in the Extension Part. | |
| 4.2.<br>Inclusion<br>Criteria | 3. Presence of the PNH white blood cell (WBC) clone ≥ 10% by high-sensitivity flow cytometry at Screening. | 3. Presence of the PNH white blood cell (WBC) clone, with a granulocyte or monocyte clone size of ≥ 10% by high-sensitivity flow cytometry at Screening. | To clarify the inclusion criteria |
| 4.3.<br>Exclusion<br>Criteria | <ul> <li>4. Abnormal haematological parameters at Screening defined as the following:</li> <li>a. Absolute neutrophil count (ANC) ≤ 500/mm³</li> <li>b. Platelet count &lt; 70,000/mm³</li> </ul> | <ul> <li>4. Abnormal haematological parameters at Screening defined as the following:</li> <li>a. Absolute neutrophil count (ANC) ≤ 500/mm³ 0.5 × 10³/μL</li> <li>b. Platelet count &lt; 70,000/mm³ 70 × 10³/μL</li> </ul> | To change the unit of haematology parameters |
| 4.3.<br>Exclusion<br>Criteria | 6. History of bone marrow transplantation. | 6. History of bone marrow haematopoietic stem cell transplantation. | To clarify the exculsion criteria |
| 4.3.<br>Exclusion<br>Criteria | <ul> <li>10. Concomitant use of any of the following medications is prohibited if the following conditions apply.</li> <li>b. Warfarin with an unstable international normalized ratio (INR) for at least 4 weeks prior to initiation of study drug (Day 1).</li> </ul> | <ul> <li>10. Concomitant use of any of the following medications is prohibited if the following conditions apply.</li> <li>b. Warfarin with an unstable international normalized normalised ratio (INR) for at least 4 weeks prior to initiation of study drug (Day 1) at the discretion of the Investigator.</li> </ul> | To clarify the exculsion criteria |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| 5.1.1. Dosing and Treatment | SB12 or Soliris® will be administered up to Week 52 (a total of 29 administrations of IP) unless they are early discontinued from study treatment. | SB12 or Soliris® will be administered up to Week 52 (a total of 29 administrations of IP) unless they are early discontinued from study treatment. | To clarify dosing and treatment schedule |
| Schedule | <ul> <li>600 mg every 7 ± 2 days for the first 4 weeks, followed by</li> <li>900 mg for the fifth dose 7 ± 2 days later, then</li> <li>900 mg every 14 ± 2 days thereafter</li> <li>In case previous IP administration was out of visit window, next visit schedule should be adjusted to keep intervals of IP administration as indicated above.</li> <li>The subject receiving SB12 or Soliris® therapy may require dose adjustment within the recommended 14 ± 2 days dosing schedule during the maintenance period (up to every 12 days) when it is deemed necessary at the discretion of the Investigator; e.g., two consecutive events of elevated LDH ≥ 2 × ULN combined with sign or symptom of intravascular haemolysis after prior LDH reduction to &lt; 1.5 × ULN on treatment. Once the above event has occurred, the Investigator should inform the medical monitor and/or Sponsor immediately.</li> </ul> | Dosing and treatment schedule of SB12 or Soliris® should be kept as follows: • 600 mg every 7 ± 2 days for the first 4 weeks, followed by • 900 mg for the fifth dose (Week 4) 7 ± 2 days later, then • 900 mg every 14 ± 2 days thereafter In case previous IP administration was out of visit window, next visit schedule should be adjusted to keep intervals of IP administration as indicated above. The treatment schedule is dependent on the previous treatment date rather than the absolute (i.e., fixed) number of days from Day 1. In other words, the next 7 ± 2 days or 14 ± 2 days treatment schedule described above is re-scheduled every time based on the date when the previous treatment is given. The subject receiving SB12 or Soliris® therapy may require dose dosing interval adjustment within the recommended 14 ± | To reflect the changes due to 2-year extension period |
| | | 2 days dosing schedule during the maintenance period (up to every 12 days) when it is deemed necessary at the discretion of the Investigator; e.g., two consecutive events of elevated LDH $\geq$ 2 × ULN combined with sign or symptom of intravascular haemolysis after prior LDH reduction to < 1.5 × ULN on treatment. For subjects whose dosing interval is adjusted to | |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | | 12 days in Period 1 of the Main Part, it is recommended that the dosing interval be switched back to 14 days after switching IP at Week 26. Once the above event has occurred, the Investigator should inform the medical monitor and/or Sponsor immediately during the Main Part, but in the Extension Part, the event can be managed at the discretion of the Investigator. | |
| 5.1.3.<br>Blinding | This study is double-blinded. Subjects, Investigators, and other study personnel will remain blinded to the treatment sequence assignment throughout the study period after randomisation. () | This The Main Part of this study is double-blinded. Subjects, Investigators, and other study personnel will remain blinded to the treatment sequence assignment throughout the study period until end of the Main Part after randomisation. () | To reflect the changes due to 2-year extension period |
| 5.2.1.<br>Identify of<br>Investigation<br>-al Product | The IPs will be supplied to investigational site in one carton containing a single vial. These IP vials will be packed and labelled in a double-blinded manner for clinical use. () | The IPs will be supplied to investigational site in one carton containing a single vial. These IP vials will be packed and labelled in a double-blinded manner for elinical use the Main Part. For the Extension Part, SB12 will also be supplied to investigational site in one carton containing a single vial. These SB12 vials will be packed and labelled using open label for the Extension Part. () | To reflect the changes due to 2-year extension period |
| 5.2.2.<br>Formulation,<br>Packaging,<br>and<br>Labelling | Eculizumab (SB12 or Soliris®) will be supplied for use as a concentrate for solution for infusion (300 mg per vial for SB12, EU sourced Soliris®). (). SB12 or Soliris® will be pre-packaged and labelled in a double-blinded form. () | Eculizumab (SB12 or Soliris®) will be supplied for use as a concentrate for solution for infusion (300 mg per vial for SB12, EU sourced Soliris®). (). SB12 or Soliris® will be pre-packaged and labelled in a double-blinded form for the Main Part. For the Extension Part, SB12 will be packaged and labelled using open label. () | To reflect the changes due to 2-year extension period |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| 5.2.4. Preparation and Administrati -on of Investigation -al Products | Dilution should be performed in accordance with good particles rules, particularly for the respect of asepsis. Withdraw the total amount of SB12 or Soliris® from the vials using a sterile syringe. Transfer the recommended dose to an infusion bag. Dilute SB12 or Soliris® to a final concentration of 5 mg/mL by addition to the infusion bag using sodium chloride 9 mg/mL (0.9%) solution for injection, sodium chloride 4.5 mg/mL (0.45%) solution for injection, or 5% dextrose in water, as the diluent. | Dilution should be performed in accordance with good particles practices rules, particularly for the respect of asepsis. Withdraw the total amount of SB12 or Soliris® from the vials using a sterile syringe. Transfer the recommended dose to an infusion bag. Dilute SB12 or Soliris® to a final concentration of 5 mg/mL by addition to the infusion bag using sodium chloride 9 mg/mL (0.9%) solution for injection, sodium chloride 4.5 mg/mL (0.45%) solution for injection, or 5% dextrose in water, as the diluent. | To correct editorial error |
| 5.2.5. Treatment Compliance and Investigation -al Product Accountabili -ty | () () At the completion or termination of the study, a final drug accountability review and reconciliation must be completed; any discrepancies must be investigated and their resolution must be documented. Unless otherwise notified, empty vials and vials with residual materials should be kept for inspection and accountability by the study monitor prior to their destruction or handled per local pharmacy SOP for clinical study drugs. () In case of expanded access of SB12 to subjects, the Investigator is responsible for maintaining the SB12 records which include information on amounts delivered, dispensed, and returned/destroyed; for ensuring proper storage conditions are maintained and documented including details of dates, quantities, batch numbers, expiry dates; ensuring the SB12 is only used as specified by the expanded access; for reconciling all SB12 | () () At the completion or termination of each part of the study, a final drug accountability review and reconciliation must be completed; any discrepancies must be investigated and their resolution must be documented. Unless otherwise notified, To avoid accidental unblinding, used drug kits (empty vials and, vials with residual materials, and cartons) should be kept for inspection promptly discarded after the infusion bag is prepared and accountability by the study monitor prior to their in accordance with the local destruction or handled per local pharmacy SOP/policies for clinical study drugs. () In case of expanded access of SB12 to subjects, the Investigator is responsible for maintaining the SB12 records which include information on amounts delivered, dispensed, and returned/destroyed; for ensuring proper storage | To reflect the changes due to 2-year extension period To revise according to latest pharmacy manual |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | received from the Sponsor. Further details will be provided in a guideline for expanded access. | conditions are maintained and documented including details of dates, quantities, batch numbers, expiry dates; ensuring the SB12 is only used as specified by the expanded access; for reconciling all SB12 received from the Sponsor. Further details will be provided in a guideline for expanded access. For the Extension Part, compliance will be assessed by the subject's source documents. All dosing information should be recorded in the subject's source documents. | |
| 5.3.<br>Concomitant<br>Medication<br>or Treatment | All medication including both prescription and non-prescription drugs, and any procedures undertaken during the study period (from the study informed consent has been signed to EOS/ET visit) should be recorded in the subject's source documents and eCRF. () | All medication including both prescription and non-prescription drugs, and any procedures undertaken during the study period (from the study informed consent has been signed to EOS/ET visit) between 4 weeks prior to Screening (except for immunosuppressant) and end of the Main Part should be recorded in the subject's source documents and eCRF. () | To reflect the changes due to 2-year extension period |
| 5.3.1.<br>Permitted<br>Concomitant<br>Medications<br>or Treatment | The following concomitant medications are allowed if on a stable dose (only for chronic administration) during the study treatment period (up to Week 52). However, for the subject's welfare, medications can be adjusted after discussion between the Investigator and medical monitor and/or Sponsor. () | The following concomitant medications are allowed if <b>given</b> on a stable dose (only for chronic administration) during the <b>study treatment period (up to Week 52) Main Part</b> . However, for the subject's welfare, medications can be adjusted after discussion between the Investigator and medical monitor and/or Sponsor. () | To reflect the changes due to 2-year extension period |
| 5.3.2.<br>Prohibited<br>Concomitant<br>Medications | Immunosuppressant except for cyclosporine is prohibited including but not limited to: () | Immunosuppressant except for cyclosporine is prohibited during the Main Part including but not limited to: () | To reflect the changes due to 2-year extension period |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| or Treatment | | | |
| 6.1.2.<br>Breakthroug<br>-h<br>Haemolysis | The Investigator and/or designee will record the breakthrough haemolysis in the source documents and eCRF during the study period. | The Investigator and/or designee will record the breakthrough haemolysis in the source documents and eCRF during the study period Main Part. | To reflect the changes due to 2-year extension period |
| 6.1.3.<br>Transfusions | () It is recommended that the transfusion would be performed within 48 hours of the haemoglobin assessment. Transfusion record will be collected from the signing of the informed consent until EOS (or 8 weeks after the last dose of study drug in case of ET). Anaemia-related signs or symptoms, haemoglobin value, number of units of pRBCs will be documented on the source documents and eCRF. | It is recommended that the transfusion would be performed within 48 hours of the haemoglobin assessment. The decision to give a transfusion may be based on either local or central laboratory haemoglobin values. Transfusion record will be collected from the signing of the informed consent until EOS end of the Main Part (or 8 weeks after the last dose of study drug in case of ET during the Main Part). Anaemia-related signs or symptoms, haemoglobin value, number of units of pRBCs will be documented on the source documents and eCRF. | To clarify the guide for transfusion To reflect the changes due to 2-year extension period |
| 6.1.4. Major<br>Adverse<br>Vascular<br>Events | The description of MAVEs, anatomical site, method of diagnosis, date of diagnosis, and outcome will be recorded in the source documents and eCRF as medical history and AEs throughout the study period. | The description of MAVEs, anatomical site, method of diagnosis, date of diagnosis, and outcome will be recorded in the source documents and eCRF as medical history and AEs throughout the study period during the Main Part. | To reflect the changes due to 2-year extension period |
| | The MAVE is defined as following; • Thrombophlebitis/deep vein thrombosis, pulmonary embolus, cerebrovascular accident, myocardial infarction, transient ischemic attack, unstable angina, renal vein thrombosis, mesenteric vein thrombosis, | The MAVE is defined as following; Thrombophlebitis/deep vein thrombosis, pulmonary embolus, cerebrovascular accident cerebral arterial/venous occlusion, myocardial infarction, transient ischemic attack, unstable angina, renal vein thrombosis, mesenteric vein thrombosis, portal vein | To update MAVE definition |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | portal vein thrombosis (Budd-Chiari syndrome), acute mesenteric ischaemia, etc. | thrombosis (Budd-Chiari syndrome), acute mesenteric ischaemia, etc. | |
| 6.1.5.<br>Paroxysmal<br>Nocturnal<br>Haemolgobi-<br>nuria-related<br>Symptoms | The PNH-related symptom questionnaire will be completed by subjects. The questionnaire will be provided to subjects before IP administration at the visits specified in Table 1 and Table 2; at Screening, Weeks 0 (Day 1), 4, 14, 26, 30, 40, and 52. () | The PNH-related symptom questionnaire will be completed by subjects. The questionnaire will be provided to should be completed by subjects before IP administration at the visits specified in Table 1 and Table 2; at Screening, Weeks 0 (Day 1), 4, 14, 26, 30, 40, and 52. () | To clarify the study procedure |
| 6.2.1.<br>Adverse<br>Events | All AEs will be recorded from the timing of the signed informed consent until EOS or 8 weeks after the last dose of study drug in case of ET. Further description on monitoring and reporting of AEs is presented in Section 8. | All AEs will be recorded from the timing of the signed-<br>informed consent until EOS or 8 weeks after the last dose of<br>study drug in case of ET. Further description on monitoring<br>and reporting of AEs is presented in according to Section 8. | To reduce<br>redundant wording<br>and simplify the<br>paragraph |
| 6.2.2.<br>Clinical<br>Laboratory<br>Evaluations | () If other laboratory tests not listed below are performed as per local practice and found to be abnormal, it is recommended that the Investigator uses their best clinical judgement to determine if the abnormal values would affect subjects' safety while participating in the study. It is highly recommended to test the abnormal parameter by central laboratory as well, if available. () | () If other laboratory tests not listed below are performed as per local practice and found to be abnormal, it is recommended that the Investigator uses their best clinical judgement to determine if the abnormal values would affect subjects' safety while participating in the study. It is highly recommended to test the abnormal parameter by central laboratory as well, if available. () | To clarify the study procedure |
| Table 5 | <ul> <li>WBC count</li> <li>RBC count</li> <li>Haemoglobi</li> </ul> | Haematology - WBC count - RBC count - RBC count - Mean - corpuscular - haemoglobin | To add several haematology parameters |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | n Haematocrit Platelet count Differential WBC count Nucleated RBC | Haemoglobin Haematocrit Haematocrit Platelet count Differential WBC count Nucleated RBC Mean corpuscular haemoglobin concentration (MCHC) Mean corpuscular volume (MCV) Mean platelet volume (MPV) Red cell distribution width (RDW) | |
| Table 5<br>Footnote | <sup>1</sup> Pregnancy test will performed for women of childbearing potential (serum or urine). Serum pregnancy test will be performed at Screening and EOS and urine pregnancy test will be performed at other applicable visits. | <sup>1</sup> Pregnancy test will <b>be</b> performed for women of childbearing potential (serum or urine). Serum pregnancy test will be performed at Screening and EOS 8 weeks after the last dose of study drug in case of ET during the Main Part and urine pregnancy test will be performed at other applicable visits before study drug administration. | To reflect the changes due to 2-year extension period and clarify the timeframe |
| 6.3.1.<br>Pharmacokin<br>-etic<br>Assessments | () The Sponsor or its designated representative will store PK samples after the end of the clinical study for several years in order to have the possibility to repeat the assay already performed (e.g., re-analysis requested by regulatory authorities or failure of first analysis [see Section 10.4]). | () The Sponsor or its designated representative will store PK samples after the end of the clinical study for several maximum 15 years in order to have the possibility to repeat the assay already performed (e.g., re-analysis requested by | To clarify the sample storage period |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | | regulatory authorities or failure of first analysis [see Section 10.4]). | |
| 6.3.2.<br>Immunogeni<br>-city<br>assessments | () Blood samples should be collected at the same day of study drug administration except for EOS/ET. Subjects' samples may be used for immunogenicity testing assay method development and/or method validation. () The Sponsor or its designated representative will store immunogenicity samples after the end of clinical study for several years in order to have the possibility to repeat the assay already performed (e.g., re-analysis requested by regulatory authorities or failure of first analysis [see Section 10.4]). | () Blood samples should be collected at the same day of study drug administration except for <b>EOS/</b> ET <b>visit</b> . Subjects' samples may be used for immunogenicity testing assay method development and/or method validation. () The Sponsor or its designated representative will store immunogenicity samples after the end of <b>the</b> clinical study for <b>several maximum 15</b> years in order to have the possibility to repeat the assay already performed (e.g., re-analysis requested by regulatory authorities or failure of first analysis [see Section 10.4]). | To reflect the changes due to 2-year extension period To clarify the sample storage period |
| 6.3.3. Pharmacody -namic Assessments | Complement activity will be measured by the validated method by the Sponsor or its designated representative. If the IP administration is delayed for any reasons after blood sample for PD is collected, blood sample for PD analysis should be repeated on actual dosing day and be used for anlaysis. In all cases, the exact date and time of the PD sampling and IP administration must be carefully recorded in the source documents and eCRF. Detail instructions of handling, storage, and shipment for PD samples are described in the laboratory manual. The Sponsor or its designated representative will store PD samples after the end of the clinical study for several years in order to have the possibility to repeat the assay already performed (e.g., re-analysis requested by regulatory authorities or failure of first analysis [see Section 10.4]). | Complement activity will be measured within the secured sample stability period by the validated method by the Sponsor or its designated representative. If the IP administration is delayed for any reasons after blood sample for PD is collected, blood sample for PD analysis should be repeated on actual dosing day and be used for anlaysis analysis. In all cases, the exact date and time of the PD sampling and IP administration must be carefully recorded in the source documents and eCRF. Detail instructions of handling, storage, and shipment for PD samples are described in the laboratory manual. The Sponsor or its designated representative will store PD samples after the end of the clinical study for several maximum 15 years in order to have the possibility to repeat the | To reflect agency comments To clarify the sample storage period |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | | assay already performed (e.g., re-analysis requested by regulatory authorities or failure of first analysis [see Section 10.4]). | |
| 6.3.4. Pharmacogenetic Assessments | () Genetic variants in C5 is associated with poor response to eculizumab since C5 mutation causes the structural change in binding site of eculizumab, resulting in less suppression of complement-mediated haemolysis. These blood samples can be used for extraction and analysis of DNA in order to investigate the mutational status of the subjects including, but not limited to C5 protein. The analysis will be performed during or after the study for subjects who present poor response to study drug, or only if scientifically appropriate and data required. () | () Genetic variants in C5 is associated with poor response to eculizumab since C5 mutation causes the structural change in binding site of eculizumab, resulting in less suppression of complement-mediated haemolysis. These blood samples can be used for extraction and analysis of DNA in order to investigate the mutational status of the subjects including, but not limited to C5 protein. The analysis will be performed during or after the study for subjects who present poor response to study drug, or only if scientifically appropriate and data required. () The Sponsor or its designated representative will store pharmacogenetic samples after the end of the clinical study for maximum 15 years in order to have the possibility to repeat the assay already performed (e.g., re-analysis requested by regulatory authorities or failure of first analysis [see Section 10.4]). | To add the sample storage period and clarify the meaning |
| 7.1. Study<br>Flow and<br>Visit<br>Schedule | During this study, efficacy, safety, PK, immunogenicity, and PD assessments will be performed. The complete schedule of activities is outlined in Table 1 and Table 2. | During this study, efficacy, safety, PK, immunogenicity, and PD assessments will be performed. The complete schedule of activities is outlined in Table 1, and Table 2, and Table 3 | To reflect the changes due to 2-year extension period |
| 7.1.1.1.<br>Screening<br>Visit (D–63<br>to D–22) | Review of laboratory results Haematology: Haemoglobin, haematocrit, RBC count, total WBC count including differential count, platelet count, and nucleated RBC | <ul> <li>Review of laboratory results</li> <li>Haematology: Haemoglobin, haematocrit, RBC count, total WBC count including differential count, platelet count, and nucleated RBC, MCH, MCHC, MCV, MPV, and RDW</li> </ul> | To add several<br>haematology<br>parameters |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| 7.1.1.2.<br>Vaccination<br>for Neisseria<br>meningitidis | To reduce the risk of meningococcal infection, all subjects must be vaccinated against Neisseria meningitidis prior to or on Day 1 in accordance with current local guidelines or Soliris® SmPC. Vaccines against serogroups A, C, Y, W135, and B where available, are recommended in preventing the commonly pathogenic meningococcal serogroups. In case subjects were vaccinated against meningococcal infection within 3 years prior to Day 1, which is properly documented, vaccination for this study could be omitted. For the information including formulation, preparation, and storage of vaccine, refer to the prescribing information in SmPC of vaccine. | To reduce the risk of meningococcal infection, all subjects must be vaccinated against Neisseria meningitidis prior to or on Day 1 in accordance with current local guidelines or Soliris® SmPC. Vaccines against serogroups A, C, Y, W135, and B where available, are recommended in preventing the commonly pathogenic meningococcal serogroups. In case subjects were vaccinated against meningococcal infection within 3 years prior to Day 1, which is properly documented, vaccination for this study could be omitted. For the information including formulation, preparation, and storage of vaccine, refer to the prescribing information in SmPC of vaccine. Subjects must be revaccinated later during the study if local guidelines indicate to do so. | To add guide for re-vaccination |
| 7.1.3.<br>Randomised<br>Treatment<br>Period | 7.1.3. Treatment Period All procedures and assessments will be performed at the visits specified in Table 1 and Table 2. Samples for laboratory assessments will be collected before IP administration on same day or up to 2 days prior, unless otherwise specified. Laboratory assessments will be performed at central laboratory. | 7.1.3. Randomised Treatment Period The Investigator should check if the subject does not meet the discontinuation criteria before the initiation of study drug at Day 1. All procedures and assessments will be performed at the visits specified in Table 1 and Table 2, Samples for laboratory assessments will | To reflect the changes due to 2-year extension period and clarify the eligibility reconfirmation process |
| | Detail instructions of collecting, processing, storing, and shipping for blood samples are described in the laboratory manual. Laboratory reports will be available to the Investigator in a timely manner for clinical management of subjects during treatment period. | be collected and before IP administration on same day or up to 2 days prior, unless otherwise specified. Laboratory assessments will be performed at central laboratory. Detail instructions of collecting, processing, storing, and shipping for blood samples are described in the laboratory | |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | () | manual. Laboratory reports will be available to the Investigator in a timely manner for clinical management of subjects during randomised treatment period. () | |
| 7.1.3.1.<br>Randomised<br>Treatment<br>Period 1<br>(before<br>Cross-over) | <ul> <li>7.1.3.1. Treatment Period 1 (before Cross-over)</li> <li>AEs, concomitant medications, MAVEs, and transfusion record will be assessed and recorded throughout the study period.</li> </ul> | <ul> <li>7.1.3.1. Randomised Treatment Period 1 (before Cross-over)</li> <li>AEs, concomitant medications, MAVEs, and transfusion record will be assessed and recorded throughout the study period.</li> </ul> | To reflect the changes due to 2-year extension period |
| 7.1.3.2. Visit<br>16 (Week<br>26/Day 183) | Each subject will cross-over from the treatment initially assigned to another treatment at Visit 16 (Week 26) and IPs will be given until Visit 29 (Week 52). () | Each subject will cross-over from the treatment initially assigned to another treatment at Visit 16 (Week 26) and IPs will be given until Visit 29 28 (Week 52 50). () | To reflect the changes due to 2-year extension period |
| 7.1.3.3. Randomised Treatment Period 2 (after Crossover) | <ul> <li>7.1.3.3. Treatment Period 2 (after Cross-over)</li> <li>AEs, concomitant medications, MAVEs, and transfusion record will be assessed and recorded throughout the study period.</li> </ul> | <ul> <li>7.1.3.3. Randomised Treatment Period 2 (after Cross-over)</li> <li>AEs, concomitant medications, MAVEs, and transfusion record will be assessed and recorded throughout the study period.</li> </ul> | To reflect the changes due to 2-year extension period |
| 7.1.3.4.<br>Early<br>Termination<br>Visit | 7.1.3.4. End of Study/Early Termination Visit (Week 60/Day 421) EOS visit and ET visit is defined as 8 weeks (± 7 days) after the last dose of study drug. | 7.1.3.4. End of Study/Early Termination Visit (Week 60/Day 421) EOS visit and ET visit is defined as 8 weeks (± 7 days) after the last dose of study drug during the randomised treatment period. This includes when the subject does not enroll into the extension period (i.e., discontinue at Week 52 without study drug administration). | To reflect the changes due to 2-year extension period |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| 7.1.4.<br>Unscheduled<br>Visits | If a sign or symptom of breakthrough haemolysis is suspected, an unscheduled visit should be occurred and samples should be collected for LDH, PK, and PD assessment for central laboratory at that time. Additionally, other unscheduled visits are permitted at the discretion of the Investigator. Any tests, procedures, or assessments performed at the unscheduled visits must be recorded in the source documents and eCRF. | If a sign or symptom of breakthrough haemolysis is suspected during randomised treatment period, an unscheduled visit should be occurred and samples should be collected for LDH, PK, and PD assessment for central laboratory at that time. Additionally, other unscheduled visits are permitted at the discretion of the Investigator. Any tests, procedures, or assessments performed at the unscheduled visits must be recorded in the source documents and eCRF. | To reflect the changes due to 2-year extension period |
| 7.1.5.<br>Extension<br>Period | N/A | After the randomised treatment period, all subjects who have completed the Main Part will enter the extension period and receive SB12 from Week 52 for 2 years. • SB12 administrations by IV infusion for 35 ± 10 minutes (900 mg every 14 ± 2 days) | To reflect the changes due to 2-year extension period |
| | | • SAEs will be assessed and recorded. Discontinuation of study treatment can be decided at the discretion of the Investigator or by subject's consent withdrawal. Specific study procedures are not required for subjects who have discontinued prematurely. SAEs must be collected until 8 weeks (± 7 days) from the last dose of study | |
| 7.2.1. Subject Discontinuat ion from Study Treatment | The study treatment must be discontinued for a subject in the event of the following: • Consent withdrawal by subject - () • Pregnancy () | drug (Section 8.2.2). The study treatment must be discontinued for a subject in the event of the following: • Consent withdrawal by subject - () • Pregnancy () | To add/revise the discontinuation criteria |
| | Other complement inhibitor use The Investigator should discuss with the medical monitor prior to | • Unblinding the study treatment to the Investigator or subject (i.e., breaking the double-blind). | |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | discontinuing a subject's study treatment in case of the following criteria, but not limited to: Conditions or intercurrent illness that preclude compliance with the protocol in terms of their safety or well-being Lack of efficacy (e.g., C5 gene polymorphism) Note: () Lack of subject's compliance (e.g., repeated delay in study treatment and lost to follow-up) Note: () Investigator discretion or other reasons | <ul> <li>Other complement inhibitor use</li> <li>The During the Main Part, the Investigator should discuss with the medical monitor prior to discontinuing a subject's study treatment in case of the following criteria, but not limited to: <ul> <li>Conditions or intercurrent illness that preclude compliance with the protocol in terms of their safety or well-being</li> <li>Lack of efficacy (e.g., C5 gene polymorphism)</li> <li>Note: ()</li> </ul> </li> <li>Unacceptable toxicity including meningococcal infection or anaphylaxis</li> <li>Serious protocol deviations including ILack of subject's compliance (e.g., repeated delay in study treatment and lost to follow-up) that preclude continuation fot the study</li> <li>Note: ()</li> <li>Investigator discretion or other reasons</li> </ul> | |
| 7.2.1. Subject Discontinuat ion from Study Treatment | Discontinuation from study treatment does not mean discontinuation from the study, and remaining study procedures should be completed as indicated by the study protocol. Only subjects who discontinue from the study at any time post-Day 1 (after the initiation of study drug) will be required to have an ET visit. The data to be collected at the 8 weeks after the last dose of study drug are described in the Section 7.1.3.4. Every effort will be employed to keep subjects who discontinued from study treatment to undertake the scheduled ET visit procedures. | For the Extension Part, discontinuation of study treatment can be decided at the discretion of the Investigator or by subject's consent withdrawal. Discontinuation from study treatment does not mean immediate discontinuation from the study, and remaining study procedures should be completed as indicated by the study protocol. Only subjects Subjects who discontinue from the study at any time post-Day 1 (after the initiation of study drug) will be required to have an ET visit. The data to be collected at the 8 weeks after | To reflect the changes due to 2-year extension period |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | Any subject who discontinues SB12 or Soliris® should be monitored for at least 8 weeks after last study drug to detect serious haemolysis and other reactions. If serious haemolysis occurs after SB12 or Soliris® discontinuation, consider the following procedures and/or treatments: • Blood transfusion (pRBCs) or exchange transfusion if the PNH RBCs are > 50% of the total RBCs by flow cytometry • Anticoagulation • Corticosteroids • Complement inhibitors According to the Investigator's medical judgement, if complement inhibitor should be administered again due to serious haemolysis and other reactions which occur within 8 weeks after completion of the study treatment with SB12 or Soliris®, the Investigator should discuss with Sponsor for an expanded access of SB12 to such subjects. Accordingly, the Sponsor will provide SB12 to those subjects as an expanded access up to 1 year period, where applicable, in accordance with relevant local regulations and/or law. | the last dose of study drug are described in the Section 7.1.3.4. Every effort will be employed to keep subjects who discontinued from study treatment to undertake the scheduled ET visit procedures. For the Extension Part, specific study procedures are not required for subjects who have discontinued the study treatment prematurely and the subject will discontinue from the study once the study treatment is permanently discontinued. SAEs must be collected until 8 weeks (± 7 days) from the last dose of study drug in such cases (Section 8.2.2). Once study treatment is discontinued during the Extension Part, it is recommended to inform the Sponsor, if occurs. () Any subject who discontinues SB12 or Soliris® should be monitored for at least 8 weeks after last dose of study drug to detect serious haemolysis and other reactions. If serious haemolysis occurs after SB12 or Soliris® discontinuation, consider the following procedures and/or treatments: • Blood transfusion (pRBCs) or exchange transfusion if the PNH RBCs are > 50% of the total RBCs by flow cytometry • Anticoagulation • Corticosteroids • Complement inhibitors According to the Investigator's medical judgement, if complement inhibitor should be administered again due to serious haemolysis and other reactions which occur within 8 weeks after completion of the study treatment with SB12 or | |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | | Soliris <sup>®</sup> , the Investigator should discuss with Sponsor for an expanded access of SB12 to such subjects. Accordingly, the Sponsor will provide SB12 to those subjects as an expanded access up to 1 year period, where applicable, in accordance with relevant local regulations and/or law. | |
| 8.1.1. Definition of Adverse Event | () All AEs during the period of observation (as specified in Section 8.1.2) including the events that occurred prior to administration of an IP should be reported as an AE in the AE section of the eCRF. () | () All AEs during the period of observation (as specified in Section 8.1.2) including the events that occurred prior to administration of an IP should be reported as an AE in the AE section of the eCRF. () | To reflect the changes due to 2-year extension period |
| 8.1.1.1.<br>Clinically<br>Significant<br>Abnormality | () If the clinically significant laboratory or other abnormality from safety assessment is not a sign of a disease or syndrome, the abnormality itself should be reported as an AE in the eCRF. If the abnormality can be characterised by a precise clinical term, the clinical term should be reported as the AE. For example, an elevated serum potassium level of 7.0 mEq/L should be reported as 'hyperkalaemia.' Observations of the same clinically significant abnormality from visit to visit should not be repeatedly reported as AEs in the eCRF, unless their severity, seriousness, or aetiology changes. | () If the clinically significant laboratory or other abnormality from safety assessment is not a sign of a disease or syndrome, the abnormality itself should be reported as an AE in the eCRF. If the abnormality can be characterised by a precise clinical term, the clinical term should be reported as the AE. For example, an elevated serum potassium level of 7.0 mEq/L should be reported as 'hyperkalaemia,'. Observations of the same clinically significant abnormality from visit to visit should not be repeatedly reported as AEs in the eCRF, unless their severity, seriousness, or aetiology changes. | To reflect the changes due to 2-year extension period |
| 8.1.2. Period<br>of<br>Observation<br>for Adverse<br>Events | AEs will be reported from the time of signing the ICF until EOS visit or ET visit. However, SAEs must be collected until 10.5 weeks from the last dose of study drug (five half-lives of the study drug). SAEs that occurred after EOS visit or ET visit must be reported to the Sponsor or its designated representative using the paper SAE report form at least within 24 hours of the Investigator | AEs will be reported from the time of signing the ICF until EOS visit end of the Main Part (or ET visit of the Main Part). Only SAEs will be collected during the Extension Part from start of study treatment at Week 52. However, SAEs must be collected until 10.5 weeks from the last dose of study drug (five half lives of the study drug). SAEs that occurred after EOS visit or ET visit must be | To reflect the changes in AE/SAE reporting period due to 2-year extension period |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | becoming aware of the event (see Section 8.2.2). Unresolved AEs during the study period should be followed up until the EOS and recorded in the eCRF. The Investigator should observe the AEs for appropriate medical care of the subject until AE resolution or stabilisation. If the subject has an ongoing SAE at the EOS, these cases will be followed until event resolution or stabilisation (see Section 8.2.2). | reported to the Sponsor or its designated representative using the paper SAE report form at least within 24 hours of the Investigator becoming aware of the event (see according to Section 8.2.2). Unresolved AEs during the study period Main Part should be followed up until end of the EOS Main Part and recorded in the eCRF. The Investigator should observe the AEs for appropriate medical care of the subject until AE resolution or stabilisation. If the subject has an ongoing SAE at 8 weeks after the last dose of study drug EOS, these cases will be followed until event resolution or stabilisation (see Section 8.2.2). | |
| 8.1.3.<br>Reporting<br>Adverse<br>Events | () If the subject who received the additional SB12 provision according to Section 7.2.1 has an AE, it must be reported to the Sponsor or its designated representative using the paper AE report form. If the AE is classified as an SAE, it must be reported to Sponsor or its designated representative using the paper SAE report form at least within 24 hours of the Investigator becoming aware of the event (see Section 8.2.2). | () If the subject who received the additional SB12 provision according to Section 7.2.1 has an AE, it must be reported to the Sponsor or its designated representative using the paper AE report form. If the AE is classified as an SAE, it must be reported to Sponsor or its designated representative using the paper SAE report form at least within 24 hours of the Investigator becoming aware of the event (see Section 8.2.2). | To reflect the changes in AE reporting due to 2-year extension period |
| 8.1.7.<br>Withdrawal<br>due to<br>Adverse<br>Events | Subject withdrawal from the study due to an AE should be distinguished from withdrawal due to personal reasons and recorded in the source documents and appropriate eCRF section. Subjects withdrawn due to an AE should be followed up until the time point specified in the protocol. When a subject withdraws from the study due to an SAE, the SAE must be reported and followed in accordance with the requirements outlined in Section 8.2.2. | Subject withdrawal from the study due to an AE should be distinguished from withdrawal due to personal reasons and recorded in the source documents and appropriate eCRF section. Subjects withdrawn due to an AE should be followed up until the time point specified in the protocol Section 7.2.1. When a subject withdraws from the study due to an SAE, the SAE must be reported and followed in accordance with the requirements outlined in Section 8.2.2. | To specify the reference section |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | () | () | |
| 8.2.2.<br>Reporting<br>Serious<br>Adverse<br>Events | SAEs must be collected until 10.5 weeks from the last dose of study drug (five half-lives of the study drug). SAEs that occurred at or before EOS visit or ET visit must be reported to the Sponsor or its designated representative via eCRF SAE report form at least within 24 hours of the Investigator becoming aware of the event. SAEs that occurred after EOS visit or ET visit must be reported to the Sponsor or its designated representative using the paper SAE report form at least within 24 hours of the Investigator becoming aware of the event. SAEs that occurred from the subject who received the additional SB12 must be reported to the Sponsor or its designated representative using the paper SAE report form at least within 24 hours of the Investigator becoming aware of the event. () The Investigator is obligated to pursue and provide information to the Sponsor on all SAEs in accordance with the timeframes for reporting specified above. In addition, an Investigator may be requested by the Sponsor to obtain specific additional follow-up information in an expedited fashion. This information may be more detailed than that captured on eCRF. In general, this will include a description of the SAE, which should be provided in sufficient detail so as to allow for a complete medical assessment of the case and | SAEs must be collected until 10.5 8 weeks (± 7 days) from the last dose of study drug (five half-lives of the study drug). SAEs that occurred at or before EOS visit until end of the Main Part (or ET visit of the Main Part) must be reported to the Sponsor or its designated representative via eCRF SAE report form at least within 24 hours of the Investigator becoming aware of the event. SAEs that occurred after EOS visit or ET visit end of the Main Part must be reported to the Sponsor or its designated representative using the paper SAE report form at least within 24 hours of the Investigator becoming aware of the event. SAEs that occurred from the subject who received the additional SB12 must be reported to the Sponsor or its designated representative using the paper SAE report form at least within 24 hours of the Investigator becoming aware of the event. () The Investigator is obligated to pursue and provide information to the Sponsor on all SAEs in accordance with the timeframes for reporting specified above. In addition, an Investigator may be requested by the Sponsor to obtain specific additional follow-up information in an expedited fashion. This information may be more detailed than that eaptured on eCRF. In general, this will include a description of the SAE, which should be provided in sufficient detail so as | To align the SAE reporting period with the safety follow-up oeriod (8 weeks) To reflect the changes in SAE reporting due to 2-year extension period |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | independent determination of possible causality. Information on other possible causes of the event, such as concomitant medications and illnesses must be provided. In the case of a subject death, a summary of available autopsy findings must be submitted as soon as possible to the Sponsor or its designated representative. () | to allow for a complete medical assessment of the case and independent determination of possible causality. Information on other possible causes of the event, such as concomitant medications and illnesses must be provided. In the case of a subject death, a summary of available autopsy findings must be submitted as soon as possible to the Sponsor or its designated representative. () | |
| 8.3.1. Meningococ -cal Infection | Due to its mechanism of action, the use of SB12 or Soliris® increases the subject's susceptibility to meningococcal infection (Neisseria meningitidis). These subjects might be at risk of disease by serogroups (particularly Y, W135, and X), although meningococcal disease due to any serogroup may occur. To reduce the risk of infection, all subjects will be vaccinated against Neisseria meningitidis prior to or on Day 1. However, vaccination may not be sufficient to prevent meningococcal infection. Consideration should be given to current local guidelines and/or the discretion of the Investigator on the appropriate use of antibacterial agents. Cases of serious or fatal meningococcal infections have been reported in Soliris®-treated patients. All subjects should be monitored for early signs of meningococcal infection, evaluated immediately if infection is suspected, and treated with appropriate antibiotics if necessary. () Subjects should be informed of these signs and symptoms and steps taken to seek medical care immediately. The Investigator must discuss the benefits and risks of SB12 or Soliris® treatment with subjects and provide them with medical | Due to its mechanism of action, the use of SB12 or Soliris® increases the subject's susceptibility to meningococcal infection (Neisseria meningitidis). These subjects might be at risk of disease by serogroups (particularly Y, W135, and X), although meningococcal disease due to any serogroup may occur. To reduce the risk of infection, all subjects will be vaccinated against Neisseria meningitidis prior to or on Day 1. Subjects must be revaccinated later during the study if local guidelines indicate to do so. However, vaccination may not be sufficient to prevent meningococcal infection. Consideration should be given to current local guidelines and/or the discretion of the Investigator on the appropriate use of antibacterial agents. Cases of serious or fatal meningococcal infections have been reported in Soliris®-treated patients. All subjects should be monitored for early signs of meningococcal infection, evaluated immediately if infection is suspected, and treated with appropriate antibiotics if necessary. () Subjects should be informed of these signs and symptoms and steps taken to seek medical care immediately. Subjects who are undergoing treatment for serious meningococcal | To add guide for re-vaccination To clarify the paragraph based on the regulatory document |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | instructions. | infections should discontinue SB12 or Soliris® treatment, and the The Investigator must discuss the benefits and risks of SB12 or Soliris® treatment with subjects and provide them with medical instructions. | |
| 8.3.3.<br>Infusion-<br>related<br>Reaction | Administration of SB12 or Soliris® may result in infusion reactions or immunogenicity that could cause allergic or hypersensitivity reactions (including anaphylaxis), though immune reactions within 48 hours of Soliris® administration did not differ from placebo arm in PNH, aHUS, refractory gMG, and other studies conducted with Soliris®. In clinical trials no PNH, aHUS, or refractory gMG patients experienced an infusion reaction which required discontinuation of Soliris®. | Administration of SB12 or Soliris® may result in infusion reactions or immunogenicity that could cause allergic or hypersensitivity reactions (including anaphylaxis), though immune reactions within 48 hours of Soliris® administration did not differ from placebo arm in PNH, aHUS, refractory gMG, NMOSD, and other studies conducted with Soliris®. In clinical trials no PNH, aHUS, or refractory gMG, or NMOSD patients experienced an infusion reaction which required discontinuation of Soliris®. | To refer the latest<br>version of<br>regulatory<br>document |
| 8.5.<br>Emergency<br>Unblinding<br>of Assigned<br>Treatment | () If IWRS is not working at emergency situation, Investigator can contact the Sponsor representative to unblind the treatment. Still, the Sponsor representative is not entitled to stall or reject unblinding and provides treatment code to the Investigator in a manual way. | () If IWRS is not working at emergency situation, Investigator can contact the Sponsor representative to unblind the treatment. Still, the Sponsor representative is not entitled to stall or reject unblinding and provides treatment code to the Investigator in a manual way. | Deleted as the process is no longer applicable. IWRS problems can be solved within IWRS framework. |
| 8.6.<br>Independent<br>Data and<br>Safety<br>Monitoring<br>Board | An independent DSMB will be assigned for this study. The DSMB will consist of external experts (i.e., haematologists, clinical pharmacologists, and biostatisticians) and will review the safety and tolerability data from the study at pre-specified intervals. The details of the safety data and time points for review will be described in the DSMB charter and in the DSMB statistical analysis plan (SAP). | An independent DSMB will be assigned for this study. The DSMB will consist of external experts (i.e., e.g., haematologists, clinical pharmacologists, and biostatisticians) and will review the safety and tolerability data from the study at pre-specified intervals. The details of the safety data and time points for review will be described in the DSMB charter and in the DSMB statistical analysis plan (SAP). | To clarify the<br>DSMB activities<br>and safety<br>monitoring process |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | In addition, an ongoing blinded review of AEs, including clinical laboratory data will be regularly and continuously undertaken by the Sponsor medical monitor. | In addition, an ongoing blinded review of AEs, including clinical laboratory data will be regularly and continuously undertaken by the Sponsor medical monitor <b>and</b> pharmacovigilance team. | |
| 9. Statistical<br>Methods and<br>Data<br>Analysis | Further information on the statistical methods for this study will be provided in the SAP, which will be finalised prior to the database lock for reporting the final clinical study report (CSR). Statistical analysis and reporting will be performed as follows: | Further information on the statistical methods for this study will be provided in the SAP, which will be finalised prior to the database lock for reporting the <b>final</b> clinical study report (CSR). Statistical analysis and reporting will be performed as follows: | To reflect the changes due to 2-year extension period |
| | • Interim safety analysis for independent DSMB meeting: | • Interim safety analysis for independent DSMB meeting: | |
| | A DSMB SAP, describing the methodology and presentation of results and access to results will be prepared as a separate document and included in the DSMB charter. The safety reports for the DSMB data review meetings will be prepared according to the DSMB SAP. | A DSMB SAP, describing the methodology and presentation of results and access to results will be prepared as a separate document <b>and included in the DSMB charter</b> . The safety reports for the DSMB data review meetings will be prepared according to the DSMB SAP. | |
| | The statistical analysis will be performed by an independent statistical reporting team and the results will be communicated to the DSMB directly by an independent unblind statistician. | The statistical analysis will be performed by an independent statistical reporting team and the results will be communicated to the DSMB directly by an independent unblind statistician. | |
| | • Final CSR: | • Final Main Part CSR: | |
| | The final analysis will take place after the last subject completes the procedures at Week 60 or the corresponding visit. All study data will be analysed and reported for final CSR. | The <b>final</b> analysis will take place after the last subject completes the procedures at Week <b>60 52</b> or the corresponding visit. All study data will be analysed and reported for <b>final</b> the <b>Main Part</b> CSR. | |
| | | • Extension Part CSR: | |
| | | A separate SAP for analyses of 2-year extension period will be prepared describing the methodology and | |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | | presentation of results. The analysis will take place after<br>the last subject completes the procedures of 2-year<br>extension period. | |
| 9.1.<br>Statistical<br>Hypotheses | or those who are in favour of the AUEC of LDH, the treatment effect will be measured by AUEC of LDH between two different time points in each period, from Week 14 to Week 26 and from Week 40 to Week 52. The equivalence will be declared if the 90% confidence interval (CI) of the ratio between treatment effects is entirely contained within the predefined equivalence margin of [0.77, 1.29]. for those who are in favour of the LDH level at a single time point, equivalence will be declared if the 95% CI of the difference between treatments in LDH level at Week 26 is entirely contained within the pre-defined equivalence margin of [-1.2 × ULN, 1.2 × ULN] where ULN of LDH to be specified in the central laboratory specification for this study. | for those who are in favour of the time-adjusted AUEC of LDH, the treatment effect will be measured by time-adjusted AUEC of LDH between two different time points in each period, from Week 14 to Week 26 and from Week 40 to Week 52. The equivalence will be declared if the 90% confidence interval (CI) of the ratio between treatment effects is entirely contained within the pre-defined equivalence margin of [0.77, 1.29]. for those who are in favour of the LDH level at a single time point, equivalence will be declared if the 95% CI of the difference between treatments in LDH level at Week 26 is entirely contained within the pre-defined equivalence margin of [-1.2 × ULN, 1.2 × ULN] where ULN of LDH to be specified in the central laboratory specification for this study. If normal range of LDH is gender specific, the smaller/smallest ULN will be used for the equivalence margin; otherwise ULN is not gender specific, unified ULN will be used for the equivalence margin. | To clarify the primary endpoint and reflect the local amendment |
| 9.2. Analysis<br>Sets | The following sets will be used for the analyses performed in the study: | The following sets will be used for the analyses performed in the study: | To reflect the changes in analysis set due to 2-year |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | <ul> <li>()</li> <li>Safety Set (SAF) consists of all subjects who receive at least one IP during the study period. Subjects will be analysed according to the treatment received.</li> <li>PK Analysis Set (PKS) consists of all subjects in the SAF who have at least one PK sample analysed.</li> <li>PD Analysis Set (PDS) consists of all subjects in the SAF who have at least one PD sample analysed.</li> </ul> | <ul> <li>()</li> <li>Safety Set for the Main Part (SAF1) consists of all subjects who receive at least one IP during the study randomised treatment period. Subjects will be analysed according to the treatment received.</li> <li>Safety Set for the Extension Part (SAF2) consists of all subjects who receive at least one IP during the extension period</li> <li>PK Analysis Set (PKS) consists of all subjects in the SAF1 who have at least one PK sample analysed.</li> <li>PD Analysis Set (PDS) consists of all subjects in the SAF1 who have at least one PD sample analysed.</li> </ul> | extension period |
| 9.4. Analysis of the Primary Objectives | who are in favour of the AUEC of LDH, the primary efficacy analysis will be performed for the PPS-AUEC using a linear mixed model with treatment, subject, sequence, and period as fixed effects and subject nested within sequence as a random effect. The analysis will be performed with loge-transformed AUEC of LDH estimating the difference in least squares means and its 90% CI, and back transformation of those values will provide the ratio of geometric means and 90% CI. The equivalence will be declared if the two-sided 90% CI of the ratio of geometric means in AUEC of LDH between SB12 and Soliris® lies within the pre-defined equivalence margin of [0.77, 1.29]. | for those who are in favour of the <b>time-adjusted</b> AUEC of LDH, the primary efficacy analysis will be performed for the PPS-AUEC using a linear mixed model with treatment, <b>subject</b> , sequence, <b>period</b> , and <b>period gender</b> as fixed effects, and subject nested within sequence as a random effect. The analysis will be performed with loge-transformed <b>time-adjusted</b> AUEC of LDH estimating the difference in least squares means and its 90% CI, and back transformation of those values will provide the ratio of geometric means and 90% CI. The equivalence will be declared if the two-sided 90% CI of the ratio of geometric means in <b>time-adjusted</b> AUEC of LDH between SB12 and Soliris® lies within the pre-defined equivalence margin of [0.77, 1.29]. | To clarify the efficacy analysis and reflect the local amendment |

Samsung Bioepis -  Information

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| | efficacy analysis will be performed for the PPS-single using a linear mixed model with treatment as a fixed effect. The analysis will be performed with log <sub>e</sub> -transformed LDH at Week 26 estimating the difference in least squares means and its 95% CI, and the delta method will be used to provide the mean difference and 95% CI in original scale. The equivalence will be declared if the two-sided 95% CI of the mean difference in LDH level at Week 26 between SB12 and Soliris <sup>®</sup> lies within the pre-defined equivalence margin of [-1.2 × ULN, 1.2 × ULN] where ULN of LDH to be specified in the central laboratory specification for this study. | for those who are in favour of the LDH level at a single time point, the primary efficacy analysis will be performed for the PPS-single using a linear mixed model with treatment, and gender as a fixed effect. The analysis will be performed with loge-transformed LDH at Week 26 estimating the difference in least squares means and its 95% CI, and the delta method will be used to provide the mean difference and 95% CI in original scale. The equivalence will be declared if the two-sided 95% CI of the mean difference in LDH level at Week 26 between SB12 and Soliris® lies within the pre-defined equivalence margin of [-1.2 × ULN, 1.2 × ULN] where ULN of LDH to be specified in the central laboratory specification for this study. | |
| 9.5.1.<br>Efficacy<br>Variable<br>Analyses | As a secondary efficacy endpoint, number of units of pRBCs transfused will be analysed using Wilcoxon rank-sum test for each period. And mean LDH profile will be presented over time. | As a secondary efficacy endpoint, number of units of pRBCs transfused during the Main Part will be analysed using Wilcoxon rank-sum test for each period. And mean LDH profile during the Main Part will be presented over time. | To reflect the changes due to 2-year extension period |
| 9.5.2. Safety<br>Analyses for<br>the Main<br>Part | 9.5.2. Safety Analyses () All TEAEs and SAEs will be summarised respectively by count and percentage of subjects experiencing events by system organ class, preferred term, treatment sequence, and period. SAEs leading to IP discontinuation and TEAEs by causality and severity will be summarised similarly. All AEs including those pre-existing before the initiation of study drug will be listed by subject. In addition, infection-related AEs including meningococcal | 9.5.2. Safety Analyses for the Main Part () All TEAEs and SAEs reported during the randomised treatment period will be summarised respectively by count and percentage of subjects experiencing events by system organ class, preferred term, treatment sequence, and period. SAEs leading to IP discontinuation and TEAEs by causality and severity will be summarised similarly. All AEs including those pre-existing before the initiation of study drug will be listed by subject. | To reflect the changes due to 2-year extension period |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| 9.5.3. Safety<br>Analyses for | infection and other systemic infection, and IRRs will also be summarised. Duration of exposure to IP and number of IV infusion will be summarised by treatment sequence and period with descriptive statistics for the SAF. Prior and concomitant medications, and significant non-drug therapies will be summarised by treatment sequence and period with count and percentage. () All safety analyses will be performed using the SAF. | In addition, infection-related AEs including meningococcal infection and other systemic infection, and IRRs reported during the randomised treatment period will also be summarised. Duration of exposure to IP and number of IV infusion during the randomised treatment period will be summarised by treatment sequence and period with descriptive statistics for the SAF1. Prior and concomitant medications, and significant non-drug therapies will be summarised by treatment sequence and period with count and percentage. () All safety analyses will be performed using the SAF1. | To reflect the changes due to 2- |
| the Extension Part | | All reported terms for SAEs will be coded using MedDRA®. SAEs reported during the Extension Part will be summarised and listed for the SAF2. Duration of exposure to IP and number of IV infusion during the Extension Part will be summarised with descriptive statistics for the SAF2. | year extension<br>period |
| 9.5.5.<br>Immunogeni<br>city<br>Analyses | () Immunogenicity analyses will be performed using the SAF. | () Immunogenicity analyses will be performed using the SAF1. | To reflect the<br>changes due to 2-<br>year extension<br>period |
| 9.6. Sample<br>Size | () For calculation of the equivalence margin for AUEC of LDH, | () For calculation of the equivalence margin for time-adjusted | To clarify the primary endpoint |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| Calculation | mean and coefficient of variation (%CV) were referred from TRIUMPH study. The mean (%CV) of AUEC of LDH at Week 26 is 81140.0 U/L × day (142.45%) and 429874.1 U/L × day (33.49%) for eculizumab and non-eculizumab arms, respectively. From the results in the reference study, mean ratio of AUEC of LDH is estimated to be 0.19 with a 90% CI [0.1308, 0.2724]. The upper limit of the equivalence margin is calculated as where it preserves at least of eculizumab treatment effect over the placebo, but the equivalence margin will be [0.77, 1.29] for the comparison with the 90% CI of mean ratio of AUEC of LDH. | AUEC of LDH, mean and coefficient of variation (%CV) were referred from TRIUMPH study. The mean (%CV) of AUEC of LDH at Week 26 is 81140.0 U/L × day (142.45%) and 429874.1 U/L × day (33.49%) for eculizumab and non-eculizumab arms, respectively. From the results in the reference study, mean ratio of <b>time-adjusted</b> AUEC of LDH is estimated to be 0.19 with a 90% CI [0.1308, 0.2724]. The upper limit of the equivalence margin is calculated as at least of eculizumab treatment effect over the placebo, but the equivalence margin will be [0.77, 1.29] for the comparison with the 90% CI of mean ratio of AUEC of LDH. | |
| 10.2<br>Monitoring | () Monitors will also perform source data verification by comparing entries in the eCRF with corresponding source data and informing the Investigator of any errors or omissions. Monitors will verify adherence to the protocol at the investigational site. All PDs will be reported to the Sponsor via the monitoring visit reports. Monitors will arrange for the supply of IP and ensure appropriate storage conditions are maintained. Monitoring visits will be conducted at regular intervals according to ICH-GCP. The monitor will provide written reports to the Sponsor on each occasion they make contact with the Investigator regardless of whether it is by phone or in person. | () () Monitors will also perform source data verification by comparing entries in the eCRF with corresponding source data and informing the Investigator of any errors or omissions for the Main Part and IP infusion date/time at Week 52. Monitors will verify adherence to the protocol at the investigational site. All PDs will be reported to the Sponsor via the monitoring visit reports. Monitors will arrange for the supply of IP and ensure appropriate storage conditions are maintained. Monitoring visits will be conducted at regular intervals according to ICH-GCP. The monitor will provide written reports to the Sponsor on each occasion they make contact with the Investigator regardless of whether it is by phone or in person () | To reflect the changes due to 2-year extension period |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| 10.5.<br>Database<br>Management<br>and Coding | Data generated within this clinical study will be handled according to the relevant SOPs of the data management and biostatistics departments of the Sponsor (or an appropriate company designated by the Sponsor to perform these activities). Subject data will be captured in an eCRF and reviewed by the monitor in order to check adherence to the protocol and to detect any data inconsistency or discrepancy. () | Data generated within this clinical study will be handled according to the relevant SOPs of the data management and biostatistics departments of the Sponsor (or an appropriate company designated by the Sponsor to perform these activities). Subject data will be captured in an eCRF and reviewed by the monitor in order to check adherence to the protocol and to detect any data inconsistency or discrepancy. The eCRF will be used only during the Main Part and IP infusion date/time at Week 52. | To reflect the changes due to 2-year extension period |
| 10.6. Quality<br>Control and<br>Quality<br>Assurance | During the conduct of the study, the Sponsor or its agent will conduct periodic monitoring visits to ensure that the protocol and ICH-GCP are being followed. The monitors may review source documents to confirm that the data recorded in the eCRF are accurate. The Investigator and institution will allow the domestic and foreign regulatory authorities, the Sponsor's monitors and auditors' direct access to source documents to perform this verification. The investigational site may be subject to review by the IRB/IEC, and/or to quality assurance audits performed by the Sponsor, and/or to inspection by appropriate regulatory authorities. It is important that the Investigators and their relevant personnel are available during the monitoring visit and possible audits or inspections and that sufficient time is devoted to the process. | During the conduct of the study, the Sponsor or its agent will conduct periodic monitoring visits to ensure that the protocol and ICH-GCP are being followed. The monitors may review source documents to confirm that the data recorded in the eCRF are accurate. The Investigator and institution will allow the domestic and foreign regulatory authorities, the Sponsor's monitors and auditors' direct access to source documents to perform this verification. The investigational site may be subject to review by the IRB/IEC, and/or to quality assurance audits performed by the Sponsor, and/or to inspection by appropriate regulatory authorities. It is important that the Investigators and their relevant personnel are available during the monitoring visit, and possible audits and/or inspections regulatory inspection(s) and that sufficient time is devoted to the process. | To reflect the changes due to 2-year extension period |
| 10.7.<br>Protocol<br>Deviation | () PDs will be reviewed and confirmed prior to database lock to decide which subjects and/or subject data will be excluded from certain analyses. Decisions regarding the exclusion of subjects and/or subject data from analyses will be documented and approved prior to database lock. | PDs will be reviewed and confirmed prior to database lock for the Main Part to decide which subjects and/or subject data will be excluded from certain analyses. Decisions regarding the exclusion of subjects and/or subject data from analyses will be documented and approved prior to database lock for the Main Part. | To reflect the<br>changes due to 2-<br>year extension<br>period |

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| 13. References | [10] Soliris® EPAR – Product Information. EMA (Oct 24, 2018). Retrieved Dec 11, 2018 from https://www.ema.europa.eu/documents/product-information/soliris-epar-product-information_en.pdf | [10] Soliris® EPAR – Product Information. EMA (Oct 24, 2018 Sep 04, 2019). Retrieved Dec 11, 2018 Sep 09, 2019 from https://www.ema.europa.eu/documents/product-information/soliris-epar-product-information_en.pdf | To refer the latest<br>version of<br>regulatory<br>document |
| 13. References | [21] Soliris® Prescribing Information. FDA (Jul 25, 2018). Retrieved Oct 04, 2018 from https://www.accessdata.fda.gov/drugsatfda docs/label/2018/125166s047s048lbl.pdf | [21] Soliris® Prescribing Information. FDA (Jul 25, 2018 Jun 27, 2019). Retrieved Oct 04, 2018 Jul 09, 2019 from https://www.accessdata.fda.gov/drugsatfda_docs/label/2018/125166s047s048lbl.pdf https://www.accessdata.fda.gov/drugsatfda_docs/label/2019/125166s431lbledt.pdf | To refer the latest<br>version of<br>regulatory<br>document |
| Protocol<br>Signature<br>Pages | Sponsor Representative Name: | Sponsor Representative Name: | Administrative change |
| Protocol<br>Signature<br>Pages | Declaration of the Global Principal/Coordinating Investigator () Global Principal/Coordinating Investigator | Declaration of the Global Principal/Coordinating Investigator () Global Principal/Coordinating Investigator | To use the terminology as defined by GCP |

Amendment 4: Version 5.0, Aug 21, 2020

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| SYNOPSIS<br>Planned<br>Study Period | After Screening, the duration of study participation will be 52-week randomised treatment period and an extension period of up to 2 years. | After Screening, the duration of study participation will be 58 weeks per subject including 52 week randomised treatment period and an extension period of up to 2 years. 50 weeks of treatment and 8 weeks of post-treatment follow-up. After completion of study treatment, subjects may be entered into an extended supply of up to 2 years. | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| SYNOPSIS<br>Study<br>Design | This multicentre Phase III study is composed of the Main Part and Extension Part. The Main Part is a randomised, double-blind period to compare the efficacy, safety, pharmacokinetics, and immunogenicity between SB12 and Soliris® in subjects with PNH. The Extension Part is an open-label, single-arm, 2-year extension period to provide SB12 in subjects with PNH for an extended duration under an ethical basis. For the Main Part, subjects will be randomised in a 1:1 ratio to treatment sequence I (SB12 to Soliris®) or treatment sequence II (Soliris® to SB12). Subjects who are randomised to initially receive SB12 will be switched to receive Soliris® and subjects who are randomised to initially receive SB12 at Week 26. End of the Main Part is defined as completion of pre-dose activities at Week 52. Subjects who complete the Main Part will enter the Extension Part. For the Extension Part, all subjects will receive SB12 for 2 years. | This multicentre Phase III study is composed of the Main Part and Extension Part. The Main Part is a randomised, Phase III, double-blind period, multicentre, cross-over study to compare the efficacy, safety, pharmacokinetics, and immunogenicity between SB12 and Soliris® in subjects with PNH. The Extension Part is an open label, single arm, 2 year extension period to provide SB12 in subjects with PNH for an extended duration under an ethical basis. For the Main Part, sSubjects will be randomised in a 1:1 ratio to treatment sequence I (SB12 to Soliris®) or treatment sequence II (Soliris® to SB12). Subjects who are randomised to initially receive SB12 will be switched to receive Soliris® and subjects who are randomised to initially receive SB12 at Week 26. End of the Main Part is defined as completion of pre-dose activities at Week 52. Subjects who complete the Main Part will enter the Extension Part. For the Extension Part, all subjects will receive SB12 for 2 years. After completion of activities at Week 52, an open-label extended supply of SB12 will be provided for up to 2 | To update study design/process in order to minimize the risk of COVID-19 pandemic |

| | | calendar years to subjects who have benefited from study<br>treatment and opt to participate in extended supply under<br>an ethical basis. | |
|---|---|---|---|
| SYNOPSIS<br>Eligibiltiy<br>Criteria | Main Eligibility Criteria: | Main Eligibility Criteria: | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| SYNOPSIS<br>Investigation<br>-al Products | • Dose regimen: 600 mg every 7 days for the first 4 weeks (initial phase) and 900 mg for the fifth week, followed by 900 mg every 14 ± 2 days, thereafter (maintenance phase). | • Dose regimen: 600 mg every 7 days for the first 4 weeks (initial phase) and 900 mg for the fifth week, followed by 900 mg every 14 ± 2 days, thereafter until Week 50 (maintenance phase). | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| SYNOPSIS<br>Main<br>Criteria for<br>Evaluation | Secondary endpoints Efficacy endpoints LDH profile during the Main Part Number of units of pRBCs transfused during the Main Part Safety endpoints () During the Extension Part, only SAEs will be collected. Immunogenicity endpoints Incidence of anti-drug antibodies (ADAs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and early termination (ET) | Secondary endpoints Efficacy endpoints LDH profile during the Main Part over time Number of units of pRBCs transfused during the Main Part throughout the study period Safety endpoints Curry During the Extension Part, only SAEs will be collected. Immunogenicity endpoints Incidence of anti-drug antibodies (ADAs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and early termination (ET) visit | To update study design/process in order to minimize the risk of COVID-19 pandemic |
| | <ul> <li>Incidence of neutralising antibodies (NAbs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and ET</li> </ul> | <ul> <li>Incidence of neutralising antibodies (NAbs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and ET visit</li> </ul> | |

| SYNOPSIS | Efficacy analyses | Efficacy analyses | To update study |
|---|---|---|---|
| Statistical<br>Methods | () | () | design/process in order to minimize |
| Methods | | | the risk of COVID- |
| | As a secondary efficacy endpoint, the number of units of | As a secondary efficacy endpoint, the number of units of | 19 pandemic |
| | pRBCs transfused during the Main Part will be analysed using | pRBCs transfused during the Main Part will be summarised | 1 |
| | Wilcoxon rank-sum test for each period. And mean LDH profile during the Main Part will be presented over time. | descriptively by treatment sequence and treatment sequence within period and will be analysed using Wilcoxon rank-sum | To clarify the |
| | during the Main Part will be presented over time. | test for each period. And mean LDH profile during the Main | efficacy/safety |
| | Safety analyses | Part will be presented over time. | analysis |
| | Safety analyses will be performed in the Safety Set for the Main Part (SAF1) and Safety Set for the Extension Part (SAF2). | Safety analyses | |
| | | Safety analyses will be performed in the Safety Set (SAF). for- | |
| | () | the Main Part (SAF1) and Safety Set for the Extension Part | |
| | All AE data reported during the Main Part will be summarised | (SAF2). | |
| | by count and percentage of subjects experiencing events by | All AE data reported during the Main Part will be | |
| | system organ class, preferred term, treatment sequence, and | summarised by count and percentage of subjects experiencing | |
| | period for the SAF1. SAEs leading to IP discontinuation and treatment-emergent AEs (TEAEs) by causality and severity will | events by system organ class, preferred term, treatment | |
| | be summarised similarly. () | sequence, and period for the SAF1. SAEs TEAEs leading to | |
| | • | IP discontinuation and treatment-emergent AEs (TEAEs) by | |
| | Changes in vital signs and clinical laboratory parameters will be | causality and severity will be summarised similarly. () | |
| | summarised descriptively by treatment sequence, period, and | Changes in vital signs and clinical laboratory parameters will be | |
| | time point for the SAF1. () | summarised descriptively by treatment sequence, period, and | |
| | All SAEs reported during the Extension Part will be | time point for the SAF1 visit. () | |
| | summarised by count and percentage of subjects experiencing | All SAEs reported during the Extension Part will be | |
| | events by system organ class and preferred term for the SAF2. | summarised by count and percentage of subjects | |
| | PK analyses | experiencing events by system organ class and preferred | |
| | | term for the SAF2. | |
| | PK analysis will be performed for the PK Analysis Set (PKS). | PK analyses | |
| | C <sub>trough</sub> will be summarised descriptively by treatment sequence, | 1 K anaryses | |
| | period, and time point. | | |

| | Immunogenicity analyses The immunogenicity analyses will be performed for the SAF1. ADA and NAb results will be summarised with count and percentage by treatment sequence, period, and time point. The incidence of overall ADA will be summarised by treatment sequence and period. PD analyses | PK analysis will be performed for the PK Analysis Set (PKS). C <sub>trough</sub> will be summarised descriptively by treatment sequence, period, and time point visit. Immunogenicity analyses The immunogenicity analyses will be performed for the SAF4. ADA and NAb results will be summarised with count and percentage by treatment sequence, period, and time point visit. The incidence of overall ADA will be summarised by treatment | |
|---|---|---|---|
| | PD analysis will be performed for the PD Analysis Set (PDS). The absolute value and change from baseline in terminal complement activities will be summarised by treatment sequence, period, and time point. | sequence and period. PD analyses PD analysis will be performed for the PD Analysis Set (PDS). The absolute value and change from baseline in terminal complement activities will be summarised by treatment sequence, period, and time point visit. | |
| Figure 1 | Sequence I (n=25) Sequence I (n=25) Sequence I (n=25) Period 1 ALEC <sup>d</sup> Period 2 AUEC <sup>d</sup> | Sequence (n=25) Soliris | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| Figure 1<br>Footnote | <ul> <li>d. From Week 4, 900 mg of SB12 or Soliris® every 14 ± 2 days up to Week 50. During the Extension Part, SB12 will be given to all subjects.</li> <li>()</li> <li>f. Completion of pre-dose activities at Week 52 is defined as end of the Main Part.</li> <li>g. EOS is defined as the date of last subject's last visit in the Extension Part.</li> </ul> | <ul> <li>d. From Week 4, 900 mg of SB12 or Soliris® every 14 ± 2 days up to Week 50. During the Extension Part, SB12 will be given to all subjects.</li> <li>()</li> <li>f. Completion of pre-dose activities at Week 52 is defined as end of the Main Part. After completion of activities at Week 52, an open-label extended supply of SB12 will be provided for up to 2 calendar years to subjects who have benefited from </li> </ul> | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |

| | | study treatment and opt to participate in extended supply under an ethical basis. g. EOS is defined as the date of last subject's last visit in the Extension Part. either completion of safety follow-up at Week 58 or completion of ET visit (8 weeks after the last dose of SB12 or Soliris®), which may be up to Week 56. | |
|---|---|---|---|
| Table 1 | Table 1. Schedule of Activities (Main Part: Period 1, before Cross-over) | Table 1. Schedule of Activities (Main Part: Period 1, before Cross-over) | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| Table 1<br>Footnote | 7. Females of childbearing potential only. Serum pregnancy test at Screening and 8 weeks after the last dose of study drug in case of early termination (ET) during the Main Part; urine pregnancy test at other applicable visits before study drug administration. | 7. Females of childbearing potential only. Serum pregnancy test at Screening and 8 weeks after the last dose of study drug in case of early termination (ET) during the Main-Part; urine pregnancy test at other applicable visits before study drug administration. | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| | () | () | |
| | 14. Blood sample for immunogenicity assay will be taken prior to dosing at Weeks 0, 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and ET. Blood samples should be collected at the same day of study drug administration except for ET visit. If the administration of IPs is delayed for any reasons after pre-dose blood sampling for immunogenicity assay, blood sample should be re-collected on actual dosing day and be used for analysis. | 14. Blood sample for immunogenicity assay will be taken prior to dosing at Weeks 0, 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and ET visit. Blood samples should be collected at the same day of study drug administration except for ET visit. If the administration of IPs is delayed for any reasons after pre-dose blood sampling for immunogenicity assay, blood sample should be re-collected on actual dosing day and be used for analysis. | |
| | () | () | |
| | 19. Adverse events (AEs) will be collected from the time of signing the informed consent until end of the Main Part (or | 19. Adverse events (AEs) will be collected from the time of signing the informed consent until <b>end of the Main Part</b> | |

| | signing the informed consent until end of the Main Part (or 8 weeks after the last dose of study drug in case of ET during the Main Part). | | (or 8 weeks after the late ET during the Main Part of the | within 4 weeks pri<br>ant, 8 weeks prio<br>all be recorded and<br>orded until end of<br>est dose of study<br>art) EOS.<br>be collected from<br>asent until end of<br>est dose of study | ior to Screening r to Screening for d concomitant fethe Main Part drug in case of the time of fethe Main Part | |
|---|---|---|---|---|---|---|
| Table 2 | Table 2. Schedule of Activities (Main Part: Period 2, after Cross-over) | | Table 2. Schedule of Activiti Tollow-up/ET, after Cross-c | ` | eriod 2 and Safety | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| Table 2 | Assessments | Study Period | Assessments | Study | Period | To update study |
| | Study Visit<br>Week | ET <sup>21</sup><br>8 (±1) weeks after the last | Study Visit | Safety<br>Follow-up <sup>21</sup> | ET <sup>22</sup> | design/process in order to minimize the risk of COVID- |
| | Day (± Visit Window) | dose of study d | Week | 58 | 8 (±1) weeks | 19 pandemic |
| | 243 (= 1350 1134011) | rug | Day (± Visit Window) | 407 (±7) | after the last<br>dose of study<br>drug | 28 F.M. |
| | | | Adverse events <sup>17</sup> | Contin | nuously | |
| | | | Previous and concomitant medications <sup>18</sup> | Contin | nuously | |
| | | | Thrombosis record (MAVEs) | Contin | nuously | |

| | | Transfusion record (date and number of Continuously pRBCs) <sup>19</sup> | |
|---|---|---|---|
| Table 2<br>Footnote | ET = Early Termination; () 4. Females of childbearing potential only. Serum pregnancy test at Screening and 8 weeks after the last dose of study drug in case of ET during the Main Part; urine pregnancy test at other applicable visits before study drug administration. | ET = Early Termination; () 4. Females of childbearing potential only. Serum pregnancy test at Screening and 8 weeks after the last dose of study drug in case of ET during the Main Part; urine pregnancy test at other applicable visits before study drug administration. To update design/proor order to mit the risk of 19 pandem | cess in inimize COVID- |
| | <ul> <li>()</li> <li>11. Blood sample for immunogenicity assay will be taken prior to dosing at Weeks 0, 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and ET. Blood samples should be collected at the same day of study drug administration except for ET visit. If the administration of IPs is delayed for any reasons after pre-dose blood sampling for immunogenicity assay, blood sample should be re-collected on actual dosing day and be used for analysis.</li> </ul> | () 11. Blood sample for immunogenicity assay will be taken prior to dosing at Weeks 0, 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and ET visit. Blood samples should be collected at the same day of study drug administration except for ET visit. If the administration of IPs is delayed for any reasons after pre-dose blood sampling for immunogenicity assay, blood sample should be re-collected on actual dosing day and be used for analysis. | |
| | <ul> <li>()</li> <li>17. AEs will be collected from the time of signing the informed consent until end of the Main Part (or 8 weeks after the last dose of study drug in case of ET during the Main Part).</li> <li>18. Concomitant medications will be recorded until end of the Main Part (or 8 weeks after the last dose of study drug in case of ET during the Main Part).</li> <li>19. Transfusion record will be collected from the time of</li> </ul> | <ul> <li>()</li> <li>17. AEs will be collected from the time of signing the informed consent until end of the Main Part (or 8 weeks after the last dose of study drug in case of ET during the Main Part) EOS.</li> <li>18. Concomitant medications will be recorded until end of the Main Part (or 8 weeks after the last dose of study drug in case of ET during the Main Part) EOS.</li> </ul> | |
| | signing the informed consent until end of the Main Part (or | 19. Transfusion record will be collected from the time of signing the informed consent until end of the Main Part | |
| | <ul> <li>8 weeks after the last dose of study drug in case of ET during the Main Part).</li> <li>20. End of the Main Part is defined as completion of pre-dose activities at Week 52.</li> <li>21. ET visit is defined as 8 weeks after the last dose of SB12 or Soliris®, which may be up to Week 58.</li> </ul> | (or 8 weeks after the last dose of study drug in case of ET during the Main Part) EOS. 20. End of the Main Part is defined as completion of predose activities at Week 52. After completion of activities at Week 52, an open-label extended supply of SB12 will be provided for up to 2 calendar years to subjects who have benefited from study treatment and opt to participate in extended supply under an ethical basis. The Week 52 activities must be completed prior to initiation of extended supply. Subjects who are eligible to participate should provide separate informed consent prior to enter an extended supply of SB12. | |
|---|---|---|---|
| | | 21. ET visit is defined as 8 weeks after the last dose of SB12 or Soliris®, which may be up to Week 58. Safety follow-up will be done at Week 58 for subjects who complete the study treatments until Week 50, regardless whether subject receives extended supply of SB12 or not. These activities will be conducted either by visit or by phone call on subjects' preference. | |
| | | 22. ET visit is defined as 8 weeks after the last dose of SB12 or Soliris®, which may be up to Week 56. Subjects who discontinue from the study at any time post-Day 1 (after the initiation of study drug) before completion of last study treatment at Week 50 will be required to have an ET visit. | |
| Table 3 | Table 7. Schedule of Activities (Extension Part: 2-year Extension Period) | Table 8. Schedule of Activities (Extension Part: 2-year Extension Period) | To update study<br>design/process in<br>order to minimize<br>the risk of COVID- |

| | Assessment | | | Study | Period | | | Assessment | | | Study | Period | | | 19 pandemic |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Week | 52 | 54 | | 152 | 154 | End<br>of<br>the<br>Exte<br>nsio<br>n<br>Part | Week | 52 | 54 | | 152 | 154 | End- of- the- Exte nsio n- Part 3 | |
| | SB12<br>administrati<br>on <sup>1</sup> | ✓ | ✓ | | ~ | ✓ | | SB12-<br>administrati | <b>≠</b> | 4 | <del></del> | 4 | 4 | | |
| | Serious<br>adverse<br>events <sup>2</sup> | | I | Contin | uously | | | Serious - adverse - events <sup>2</sup> | | ı | Contir | nuously | | | |
| | From Wee IV infusio Only SAE from start End of the last dose on not require Main Part. | n for 35<br>s will be<br>of study<br>Extensi<br>f SB12.<br>e any spo | ± 10 mi<br>e collect<br>treatme<br>ion Part<br>Premate | nutes for<br>ed during<br>ent at We<br>is define<br>urely dis | r all subject the Extends of the Ext | ects. tension reeks aft | Part er the ets do | From Wee IV infusio Only SAE from start End of the last dose of not require Main Part | n for 35 s will be of study Extension SB12. c any sp | ± 10 mi<br>collect<br>treatme<br>ion Part<br>Premat | inutes for<br>ed during<br>ent at Wo<br>is define<br>urely dis | r all subgethe Exceed 52. Seed as 8 westinue | jects.<br>tension :<br>vecks aft<br>ed subject | Part— er the— ets do— | |
| LIST OF<br>ABBREVIA | N/A<br>SAF1 | N/A<br>Safety | Set for | the Maii | n Part | | | COVID-19 DSUR | | | Disease<br>Safety | | Renort | | To revise/add abbreviations |
| -TIONS | SAF2 | • | | the Exte | | ırt | | IgG | | inoglob | · | - paut | - report | | according to updated contents |
| | | | | | | | | PC | | ict Com | - | sto Dow | · ut | | |
| | | | | | | | | PSUR | Perio | dic Safe | ety Upda | ite Repo | ort | | |

| | | SAF1 Safety Set for the Main Part | |
|---|---|---|---|
| | | SAF2 Safety Set for the Extension Part | |
| LIST OF<br>STUDY<br>STAFF | Clinical Project Manager | Clinical Project — | Administrative change |
| | Clinical Development Assistant Statistician | Clinical Research Physician | |
| | Project Safety Lead | Clinical Development Assistant Research Scientist | |
| | | Statistician | |
| | | Project Safety Lead | |
| 1.2.<br>Overview of<br>SB12 | () SB12 and Soliris® have identical primary structure and the active substance for both products is eculizumab, a humanised monoclonal antibody (IgG2/4 kappa immunoglobulin) that binds to the human C5 complement protein with high affinity. Binding to this protein blocks its cleavage into C5a and C5b, thereby inhibiting terminal complement-mediated intravascular haemolysis. | () SB12 and Soliris® have identical primary structure and the active substance for both products is eculizumab, a humanised monoclonal antibody (immunoglobulin G[IgG]2/4 kappa immunoglobulin) that binds to the human C5 complement protein with high affinity. Binding to this protein blocks its cleavage into C5a and C5b, thereby inhibiting terminal complement-mediated intravascular haemolysis. | To refer the latest information |

| | () According to the guideline International Conference on Harmonisation Q6B, characterisation of a biological therapeutic must involve its physicochemical properties, biological activities, purity, impurities, and quantity. () | () According to the guideline International Conference on Council for Harmonisation (ICH) Q6B, characterisation of a biological therapeutic must involve its physicochemical properties, biological activities, purity, impurities, and quantity. () | |
|---|---|---|---|
| 1.5.1.<br>Known<br>Potential<br>Risks | According to Soliris® Summary of Product Characteristics (SmPC) [10], supportive safety data were collected from 30 completed and one ongoing clinical studies that included 1,503 patients exposed to eculizumab in complement-mediated disease populations, including PNH, aHUS, refractory gMG and NMOSD. The most common adverse reaction was headache (occurred mostly in the initial phase) and of all meningococcal infections the most frequently reported serious adverse reaction was meningococcal sepsis. | According to Soliris® Summary of Product Characteristics (SmPC) [10], supportive safety data were collected from 30 31 completed and one ongoing clinical studies that included 1,503 patients exposed to eculizumab in complement-mediated disease populations, including PNH, aHUS, refractory gMG and NMOSD. The most common adverse reaction was headache (occurred mostly in the initial phase) and of all meningococcal infections—the most frequently reported serious adverse reaction was meningococcal sepsis. | To refer the latest<br>version of<br>regulatory<br>document |
| 2.2.2.<br>Secondary<br>Endpoints | Secondary endpoints Efficacy endpoints LDH profile during the Main Part Number of units of pRBCs transfused during the Main Part Safety endpoints () During the Extension Part, only SAEs will be collected. Immunogenicity endpoints Incidence of anti-drug antibodies (ADAs) at Weeks 0 | Secondary endpoints Efficacy endpoints LDH profile during the Main Part over time Number of units of pRBCs transfused during the Main Part throughout the study period Safety endpoints Curing the Extension Part, only SAEs will be collected. Immunogenicity endpoints Incidence of anti-drug antibodies (ADAs) at Weeks 0 | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| | (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and early termination (ET) | (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and early termination (ET) <b>visit</b> | |

| | • Incidence of neutralising antibodies (NAbs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and ET | • Incidence of neutralising antibodies (NAbs) at Weeks 0 (Day 1), 2, 4, 6, 10, 14, 18, 22, 26, 28, 30, 32, 36, 40, 44, 48, 52, and ET <b>visit</b> | |
|---|---|---|---|
| 3.1.<br>Overview of<br>Study | This multicentre Phase III study is composed of the Main Part and Extension Part. | This multicentre Phase III study is composed of the Main Part and Extension Part. | To update study design/process in order to minimize |
| Design | The Main Part is a randomised, double-blind period to compare | The Main Part is a randomised, Phase III, double-blind period, | the risk of COVID |
| | the efficacy, safety, pharmacokinetics, and immunogenicity | multicentre, cross-over study to compare the efficacy, safety, | 19 pandemic |
| | between SB12 and Soliris® in subjects with PNH. The Extension | pharmacokinetics, and immunogenicity between SB12 and | |
| | Part is an open-label, single-arm, 2-year extension period to | Soliris® in subjects with PNH. The Extension Part is an open- | |
| | provide SB12 in subjects with PNH for an extended duration | label, single-arm, 2-year extension period to provide SB12 in | |
| | under an ethical basis. | subjects with PNH for an extended duration under an ethical | |
| | Cubicata will be mandamized in a 1.1 matic to treatment accusance | <del>basis.</del> | |
| | Subjects will be randomised in a 1:1 ratio to treatment sequence | C-1.i-4i111did-id | |
| | I (SB12 to Soliris®) or treatment sequence II (Soliris® to SB12). | Subjects will be randomised in a 1:1 ratio to treatment sequence | |
| | Subjects randomly assigned to treatment with SB12 or Soliris® | I (SB12 to Soliris®) or treatment sequence II (Soliris® to SB12). | |
| | will receive 600 mg of eculizumab IV every week for first 4 | Subjects randomly assigned to treatment with SB12 or Soliris® | |
| | weeks (initial phase) and 900 mg for the fifth week, followed by | will receive 600 mg of eculizumab IV every week for first 4 | |
| | 900 mg every 2 weeks thereafter. Subjects who are randomised | weeks (initial phase) and 900 mg for the fifth week, followed by | |
| | to initially receive SB12 will be switched to receive Soliris® and | 900 mg every 2 weeks thereafter. Subjects who are randomised | |
| | subjects who are randomised to initially receive Soliris® will be | to initially receive SB12 will be switched to receive Soliris® and | |
| | switched to receive SB12 at Week 26. SB12 or Soliris® will be | subjects who are randomised to initially receive Soliris® will be | |
| | given until Week 50. End of the Main Part is defined as | switched to receive SB12 at Week 26. SB12 or Soliris® will be | |
| | completion of pre-dose activities at Week 52. Subjects who | given until Week 50. End of the Main Part is defined as | |
| | complete the Main Part will enter the Extension Part. | completion of pre-dose activities at Week 52. Subjects who | |
| | For the Extension Part, all subjects will receive SB12 for 2 years. | complete the Main Part will enter the Extension Part. | |
| | Details of assessment that will be conducted and treatment that | For the Extension Part, all subjects will receive SB12 for 2 years. | |
| | will be administered are presented in, Table 1, Table 2, and Table | <del>years.</del> | |
| | 3. The last assessment for the Main Part will be performed at pre- | Details of assessment that will be conducted and treatment that | |
| | dose of Week 52 or 8 weeks after the last dose of SB12 or Soliris® | will be administered are presented in, Table 1 and Table 2, and | |
| | in case of ET during the Main Part. The last assessment for the | Table 3. The last assessment for the Main Part will be | |
| | Extension Part will be performed at 8 weeks after the last dose of | performed at pre-dose of Week 52 58 or 8 weeks after the last | |

| | SB12. | dose of SB12 or Soliris® in case of ET during the Main Part. The last assessment for the Extension Part will beperformed at 8 weeks after the last dose of SB12. After completion of activities at Week 52, an open-label extended supply of SB12 will be provided for up to 2 calendar years to subjects who have benefited from study treatment and opt to participate in extended supply under an ethical basis. | |
|---|---|---|---|
| 3.3. Duration of Study Participation | After Screening, the duration of study participation will be 52-week randomised treatment period and an extension period of up to 2 years. | After Screening, the duration of study participation will be 58 weeks per subject including 52-week randomised treatment period and an extension period of up to 2 years. 50 weeks of treatment and 8 weeks of post-treatment follow-up. After completion of study treatment, subjects may be entered into an extended supply of up to 2 years. | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| 3.5. End of Study Definition | A subject is considered to have completed the each part of study if he or she has completed all study treatment including the last visit or the last scheduled procedure shown in Table 2 and Table 3. The end of the Main Part is defined as completion of pre-dose activities at Week 52 for subjects. The end of the Extension Part is defined as 8 weeks after the last dose of SB12. The end of study (EOS) is defined as the date of last subject's last visit in the Extension Part. | A subject is considered to have completed the each part of study if he or she has completed all study treatment including and the last visit or the last scheduled procedure shown in Table 2 and Table 3. The end of the Main Part end of study (EOS) is defined as completion of pre-dose activities safety follow-up at Week 52 for subjects. The end of the Extension Part is defined as 58 or completion of ET visit (8 weeks after the last dose of SB12 or Soliris®). The end of this clinical study is defined as completion of the last subject's EOS. The end of study (EOS) is defined as the date of last subject's last visit in the Extension Part. | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| 4.4. Screen<br>Failures and<br>Re-screening | N/A | During Coronavirus Disease 2019 (COVID-19) pandemic circumstances, eligibility may not be confirmed at Screening due to unexpected COVID-19 related restrictions. These cases may fall into screen failures due to out of 42 days screening window or consent withdrawal related with COVID-19 concern, etc. These will be considered as | To implement<br>recommendations<br>belonging to DDLs<br>issued to address<br>COVID-19<br>pandemic |

| | | technical issue so that re-screening is applicable after COVID-19 related restrictions are relieved. | |
|---|---|---|---|
| 5.1.1. Dosing and Treatment Schedule | Dosing and treatment schedule of SB12 or Soliris® should be kept as follows: • 600 mg every 7 ± 2 days for the first 4 weeks, followed by • 900 mg for the fifth dose 7 ± 2 days later, then • 900 mg every 14 ± 2 days thereafter () The subject receiving SB12 or Soliris® therapy may require dosing interval adjustment within the recommended 14 ± 2 days dosing schedule during the maintenance period (up to every 12 days) when it is deemed necessary at the discretion of the Investigator; e.g., two consecutive events of elevated LDH ≥ 2 × ULN combined with sign or symptom of intravascular haemolysis after prior LDH reduction to < 1.5 × ULN on treatment. For subjects whose dosing interval is adjusted to 12 days in Period 1 of the Main Part, it is recommended that the dosing interval be switched back to 14 days after switching IP at Week 26. Once the above event has occurred, the Investigator should inform the medical monitor and/or Sponsor immediately during the Main Part, but in the Extension Part, the event can be managed at the discretion of the Investigator. | SB12 or Soliris® will be administered up to Week 50 (a total of 28 administrations of IP) unless they are early discontinued from study treatment. Dosing and treatment schedule of SB12 or Soliris® should be kept as follows: • 600 mg every 7 ± 2 days for the first 4 weeks, followed by • 900 mg for the fifth dose 7 ± 2 days later, then • 900 mg every 14 ± 2 days thereafter () The subject receiving SB12 or Soliris® therapy may require dosing interval adjustment within the recommended 14 ± 2 days dosing schedule during the maintenance period (up to every 12 days) when it is deemed necessary at the discretion of the Investigator; e.g., two consecutive events of elevated LDH ≥ 2 × ULN combined with sign or symptom of intravascular haemolysis after prior LDH reduction to < 1.5 × ULN on treatment. If a 12 or 13 day dosing interval conflicts with administrative schedules (e.g., holidays or weekends) but a shortened dosing interval is considered necessary for safety of subject, consultation with medical monitor (or Sponsor) is recommended. For subjects whose dosing interval is adjusted to 12 days in Period 1 of the Main Part, it is recommended that the dosing interval be switched back to 14 days after switching IP at Week 26. Once the above event has occurred, the Investigator should inform the medical monitor and/or Sponsor immediately during the Main Part, but in the Extension | To update study design/process in order to minimize the risk of COVID-19 pandemic To add clarification of dosing interval adjustement to address DSMB feedback |

| | | Part, the event can be managed at the discretion of the Investigator. | |
|---|---|---|---|
| 5.1.3.<br>Blinding | The Main Part of this study is double-blinded. Subjects, Investigators, and other study personnel will remain blinded to the treatment sequence assignment until end of the Main Part after randomisation. () | The Main Part of tThis study is double-blinded. Subjects, Investigators, and other study personnel will remain blinded to the treatment sequence assignment until end of the Main Part throughout the study period after randomisation. () | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| 5.2.1.<br>Identify of<br>Investigation<br>-al Product | The IPs will be supplied to investigational site in one carton containing a single vial. These IP vials will be packed and labelled in a double-blinded manner for the Main Part. For the Extension Part, SB12 will also be supplied to investigational site in one carton containing a single vial. These SB12 vials will be packed and labelled using open label for the Extension Part. () | The IPs will be supplied to investigational site in one carton containing a single vial. These IP vials will be packed and labelled in a double-blinded manner for the Main Part. For the Extension Part, SB12 will also be supplied to investigational site in one carton containing a single vial. These SB12 vials will be packed and labelled using open label for the Extension Part clinical use. () | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| 5.2.2.<br>Formulation,<br>Packaging,<br>and<br>Labelling | Packaging and labelling of SB12 or Soliris® will follow standard operating procedure (SOP) of the manufacturing site and regulatory requirements in each country, as well as will be in accordance with International Council for Harmonisation (ICH)-Good Clinical Practice (GCP). SB12 or Soliris® will be pre-packaged and labelled in a double-blinded form for the Main Part. For the Extension Part, SB12 will be packaged and labelled using open label. () | () Packaging and labelling of SB12 or Soliris® will follow standard operating procedure (SOP) of the manufacturing site and regulatory requirements in each country, as well as will be in accordance with International Council for Harmonisation—(ICH)—Good Clinical Practice (GCP). SB12 or Soliris® will be pre-packaged and labelled in a double-blinded form for the—Main Part. For the Extension Part, SB12 will be packaged—and labelled using open label. () | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| 5.2.5. Treatment Compliance and Investigation -al Product | () At the completion or termination of each part of the study, a final drug accountability review and reconciliation must be completed; any discrepancies must be investigated and their | () At the completion or termination of each part of the study, a final drug accountability review and reconciliation must be completed; any discrepancies must be investigated and their | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |

| Accountabili | resolution must be documented. | resolution must be documented. | |
|---|---|---|---|
| -ty | () For the Extension Part, compliance will be assessed by the subject's source documents. All dosing information should be recorded in the subject's source documents. | () For the Extension Part, compliance will be assessed by the subject's source documents. All dosing information should be recorded in the subject's source documents. | |
| 5.3.<br>Concomitant<br>Medication<br>or Treatment | All medication including both prescription and non-prescription drugs, and any procedures undertaken between 4 weeks prior to Screening (except for immunosuppressant) and end of the Main Part should be recorded in the subject's source documents and eCRF. () | All medication including both prescription and non-prescription drugs, and any procedures undertaken between 4 weeks prior to Screening (except for immunosuppressant) and end of the Main Part EOS should be recorded in the subject's source documents and eCRF. () | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| 5.3.1. Permitted Concomitant Medications or Treatment | The following concomitant medications are allowed if given on a stable dose (only for chronic administration) during the Main Part. However, for the subject's welfare, medications can be adjusted after discussion between the Investigator and medical monitor and/or Sponsor. | The following concomitant medications are allowed if given on a stable dose (only for chronic administration) during the Main Part study period. However, for the subject's welfare, medications can be adjusted after under discussion between the Investigator and medical monitor and/or Sponsor. | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| | () | () | To clarify the meaning regarding permitted medications dose adjustement for subjects' welfare |
| 5.3.2.<br>Prohibited<br>Concomitant<br>Medications<br>or Treatment | Immunosuppressant except for cyclosporine is prohibited during the Main Part including but not limited to: () | Immunosuppressant except for cyclosporine is prohibited during the Main Part study period from randomisation including but not limited to: () | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |

| 6.1.2.<br>Breakthroug<br>-h<br>Haemolysis | The Investigator and/or designee will record the breakthrough haemolysis in the source documents and eCRF during the Main Part. () | The Investigator and/or designee will record the breakthrough haemolysis in the source documents and eCRF during the Main Part study period. () | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
|---|---|---|---|
| 6.1.3.<br>Transfusions | () Transfusion record will be collected from the signing of the informed consent until end of the Main Part (or 8 weeks after the last dose of study drug in case of ET during the Main Part). Anaemia-related signs or symptoms, haemoglobin value, number of units of pRBCs will be documented on the source documents and eCRF. | Transfusion record will be collected from the signing of the informed consent until end of the Main Part (or 8 weeks after the last dose of study drug in case of ET during the Main Part) EOS. Anaemia-related signs or symptoms, haemoglobin value, number of units of pRBCs will be documented on the source documents and eCRF. | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| 6.1.4. Major<br>Adverse<br>Vascular<br>Events | The description of MAVEs, anatomical site, method of diagnosis, date of diagnosis, and outcome will be recorded in the source documents and eCRF as AEs during the Main Part. () | The description of MAVEs, anatomical site, method of diagnosis, date of diagnosis, and outcome will be recorded in the source documents and eCRF as AEs during the <b>Main Part study period</b> . () | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| 6.2.2.<br>Clinical<br>Laboratory<br>Evaluations | N/A | During COVID-19 pandemic circumstances, it may be unable to get central laboratory values in time due to COVID-19 related restrictions. For those cases, local laboratory will be allowed in addition to central laboratory for scheduled visit after randomisation until COVID-19 restrictions are relieved under discussion with Sponsor. | To implement<br>recommendations<br>belonging to DDLs<br>issued to address<br>COVID-19<br>pandemic |
| Table 4 Footnote | <sup>1</sup> Pregnancy test will be performed for women of childbearing potential (serum or urine). Serum pregnancy test will be performed at Screening and 8 weeks after the last dose of study drug in case of ET during the Main Part and urine pregnancy test will be performed at other applicable visits before study drug administration. | <sup>1</sup> Pregnancy test will be performed for women of childbearing potential (serum or urine). Serum pregnancy test will be performed at Screening and 8 weeks after the last dose of study drug in case of ET <b>during the Main Part</b> and urine pregnancy test will be performed at other applicable visits before study drug administration. | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |

| 6.3.2.<br>Immunogeni<br>-city<br>assessments | () Blood samples should be collected at the same day of study drug administration except for ET visit. () () | () Blood samples should be collected at the same day of study drug administration except for ET visit. () () | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
|---|---|---|---|
| 7.1. Study<br>Flow and<br>Visit<br>Schedule | During this study, efficacy, safety, PK, immunogenicity, and PD assessments will be performed. The complete schedule of activities is outlined in Table 1, Table 2, and Table 3. | During this study, efficacy, safety, PK, immunogenicity, and PD assessments will be performed. The complete schedule of activities is outlined in Table 1, and Table 2, and Table 3. | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| 7.1.2.<br>Randomisati<br>-on | N/A | During COVID-19 pandemic circumstances, Day 1 (1st dosing) may not be started within 21 days of randomisation due to unexpected COVID-19 related restrictions. In such cases, the subject will be monitored for safety per Investigator's discretion. Day 1 will be started after the COVID-19 related restrictions are relieved. | To implement<br>recommendations<br>belonging to DDLs<br>issued to address<br>COVID-19<br>pandemic |
| 7.1.3.<br>Treatment<br>Period | 7.1.3. Randomised Treatment Period () Laboratory assessments will be performed at central laboratory. Detail instructions of collecting, processing, storing, and shipping for blood samples are described in the laboratory manual. Laboratory reports will be available to the Investigator in a timely manner for clinical management of subjects during randomised treatment period. () | 7.1.3. Randomised Treatment Period () Laboratory assessments will be performed at central laboratory. Detail instructions of collecting, processing, storing, and shipping for blood samples are described in the laboratory manual. Laboratory reports will be available to the Investigator in a timely manner for clinical management of subjects during randomised treatment period. () | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| 7.1.3.1.<br>Randomised<br>Treatment<br>Period 1<br>(before | 7.1.3.1. Randomised Treatment Period 1 (before Cross-over) | 7.1.3.1. Randomised Treatment Period 1 (before Cross-over) | To update study<br>design/process in<br>order to minimize<br>the risk of COVID- |

| Cross-over) | | | 19 pandemic |
|---|---|---|---|
| 7.1.3.3. Randomised Treatment Period 2 (after Crossover) | 7.1.3.3. Randomised Treatment Period 2 (after Cross-over) | 7.1.3.3. Randomised Treatment Period 2 (after Cross-over) | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| 7.1.3.4.<br>Early<br>Termination<br>Visit | N/A | <ul> <li>7.1.3.4. Safety Follow-up (Week 58/Day 407)</li> <li>Safety follow-up will be done at Week 58 (± 7 days) which is 8 weeks after the last dose of SB12 or Soliris® for subjects who complete the study treatments until Week 50, regardless whether subject receives extended supply of SB12 or not to ensure subject's safety. These activities will be conducted either by visit or by phone call based on subjects' preference.</li> <li>AEs, concomitant medications, MAVEs, and transfusion record will be assessed and recorded.</li> </ul> | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| 7.1.3.5.<br>Early<br>Termination<br>Visit | 7.1.3.4. Early Termination Visit ET visit is defined as 8 weeks (± 7 days) after the last dose of study drug during the randomised treatment period. This includes when the subject does not enroll into the extension period (i.e., discontinue at Week 52 without study drug administration). () | 7.1.3.4. 7.1.3.5. Early Termination Visit ET visit is defined as 8 weeks (± 7 days) after the last dose of study drug SB12 or Soliris® during the randomised treatment period. This includes when the subject does not enroll into the extension period (i.e., discontinue at Week 52 without study drug administration). () | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| 7.1.4.<br>Unscheduled<br>Visits | If a sign or symptom of breakthrough haemolysis is suspected during randomised treatment period, an unscheduled visit should be occurred and samples should be collected for LDH, PK, and | If a sign or symptom of breakthrough haemolysis is suspected during randomised treatment period, an unscheduled visit | To update study<br>design/process in<br>order to minimize<br>the risk of COVID- |

| PD assessment for central laboratory at that time. () | should be occurred and samples should be collected for LDH, PK, and PD assessment for central laboratory at that time. () | 19 pandemic |
|---|---|---|
| <ul> <li>7.1.5. Extension Period</li> <li>After the randomised treatment period, all subjects who have completed the Main Part will enter the extension period and receive SB12 from Week 52 for 2 years.</li> <li>SB12 administrations by IV infusion for 35 ± 10 minutes (900 mg every 14 ± 2 days)</li> <li>SAEs will be assessed and recorded.</li> </ul> | 7.1.5. Extension Period After the randomised treatment period, all subjects who have completed the Main Part will enter the extension period and receive SB12 from Week 52 for 2 years. * SB12 administrations by IV infusion for 35 ± 10 minutes (900 mg every 14 ± 2 days) * SAEs will be assessed and recorded. | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| Discontinuation of study treatment can be decided at the discretion of the Investigator or by subject's consent withdrawal. Specific study procedures are not required for subjects who have discontinued prematurely. SAEs must be collected until 8 weeks (± 7 days) from the last dose of study drug (Section 8.2.2). | Discontinuation of study treatment can be decided at the discretion of the Investigator or by subject's consent withdrawal. Specific study procedures are not required for subjects who have discontinued prematurely. SAEs must be collected until 8 weeks (± 7 days) from the last dose of study drug (Section 8.2.2). | |
| () During the Main Part, the Investigator should discuss with the medical monitor prior to discontinuing a subject's study treatment in case of the following criteria, but not limited to: () For the Extension Part, discontinuation of study treatment can be | During the Main Part, tThe Investigator should discuss with the medical monitor prior to discontinuing a subject's study treatment in case of the following criteria, but not limited to: () For the Extension Part, discontinuation of study treatment | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| decided at the discretion of the Investigator or by subject's consent withdrawal. Discontinuation from study treatment does not mean immediate discontinuation from the study, and remaining study procedures | can be decided at the discretion of the Investigator or by subject's consent withdrawal. Discontinuation from study treatment does not mean immediate discontinuation from the study, and remaining study procedures | |
| | 7.1.5. Extension Period After the randomised treatment period, all subjects who have completed the Main Part will enter the extension period and receive SB12 from Week 52 for 2 years. • SB12 administrations by IV infusion for 35 ± 10 minutes (900 mg every 14 ± 2 days) • SAEs will be assessed and recorded. Discontinuation of study treatment can be decided at the discretion of the Investigator or by subject's consent withdrawal. Specific study procedures are not required for subjects who have discontinued prematurely. SAEs must be collected until 8 weeks (± 7 days) from the last dose of study drug (Section 8.2.2). () During the Main Part, the Investigator should discuss with the medical monitor prior to discontinuing a subject's study treatment in case of the following criteria, but not limited to: () For the Extension Part, discontinuation of study treatment can be decided at the discretion of the Investigator or by subject's consent withdrawal. Discontinuation from study treatment does not mean immediate | 7.1.5. Extension Period After the randomised treatment period, all subjects who have completed the Main Part will enter the extension period and receive SB12 from Week 52 for 2 years. • SB12 administrations by IV infusion for 35 ± 10 minutes (900 mg every 14 ± 2 days) • SAEs will be assessed and recorded. Discontinuation of study treatment can be decided at the discretion of the Investigator or by subject's consent withdrawal. Specific study procedures are not required for subjects who have discontinued prematurely. SAEs must be collected until 8 weeks (± 7 days) from the last dose of study drug (Section 8.2.2). () During the Main Part, the Investigator should discuss with the medical monitor prior to discontinuing a subject's study treatment in case of the following criteria, but not limited to: () For the Extension Part, discontinuation of study treatment does not mean immediate discontinuation from study treatment does not mean immediate discontinuation from the study, and remaining study procedures |

| 8.1.2. Period of Observation for Adverse Events | who discontinue from the study at any time post-Day 1 (after the initiation of study drug) will be required to have an ET visit. The data to be collected at the 8 weeks after the last dose of study drug are described in the Section 7.1.3.4. Every effort will be employed to keep subjects who discontinued from study treatment to undertake the scheduled ET visit procedures. For the Extension Part, specific study procedures are not required for subjects who have discontinued the study treatment prematurely and the subject will discontinue from the study once the study treatment is permanently discontinued. SAEs must be collected until 8 weeks (± 7 days) from the last dose of study drug in such cases (Section 8.2.2). Once study treatment is discontinued during the Extension Part, it is recommended to inform the Sponsor, if occurs. () AEs will be reported from the time of signing the ICF until end of the Main Part (or ET visit of the Main Part). Only SAEs will be collected during the Extension Part from start of study treatment at Week 52. () Unresolved AEs during the Main Part should be followed up until end of the Main Part and recorded. The Investigator should observe the AEs for appropriate medical care of the subject until AE resolution or stabilisation. If the subject has an ongoing SAE at 8 weeks after the last dose | who discontinue from the study at any time post-Day 1 (after the initiation of study drug) before completion of last study treatment at Week 50 will be required to have an ET visit. The data to be collected at the 8 weeks after the last dose of study drug are described in the Section 7.1.3.4 7.1.3.5. Every effort will be employed to keep subjects who discontinued from study treatment to undertake the scheduled ET visit procedures. For the Extension Part, specific study procedures are not required for subjects who have discontinued the study treatment prematurely and the subject will discontinue from the study once the study treatment is permanently discontinued. SAEs must be collected until 8 weeks (± 7 days) from the last dose of study drug in such cases (Section 8.2.2). Once study treatment is discontinued during the Extension Part, it is recommended to inform the Sponsor, if occurs. () AEs will be reported from the time of signing the ICF until end of the Main Part (or ET visit of the Main Part). Only SAEs will be collected during the Extension Part from start of study treatment at Week 52 EOS. () Unresolved AEs during the Main Part and recorded EOS. The Investigator should observe the AEs for appropriate medical care of the subject until AE resolution or stabilisation. If the subject has an ongoing SAE at 8 weeks after the last dose | To update study design/process in order to minimize the risk of COVID-19 pandemic |
|---|---|---|---|
| | · | | |

| 8.2.2.<br>Reporting<br>Serious<br>Adverse<br>Events | SAEs that occurred until end of the Main Part (or ET visit of the Main Part) must be reported to the Sponsor or its designated representative via eCRF SAE report form at least within 24 hours of the Investigator becoming aware of the event. SAEs that occurred after end of the Main Part must be reported to the Sponsor or its designated representative using the paper | SAEs that occurred until end of the Main Part (at or ET visit of the Main Part) before EOS must be reported to the Sponsor or its designated representative via eCRF SAE report form at least within 24 hours of the Investigator becoming aware of the event. SAEs that occurred after end of the Main Part EOS must be reported to the Sponsor or its designated representative using | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
|---|---|---|---|
| | SAE report form at least within 24 hours of the Investigator becoming aware of the event. () | the paper SAE report form at least within 24 hours of the Investigator becoming aware of the event. () | |
| 9. Statistical<br>Methods and<br>Data<br>Analysis | Statistical analysis and reporting will be performed as follows: () Main Part CSR: | Statistical analysis and reporting will be performed as follows: () Main Part CSR: | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| | The analysis will take place after the last subject completes<br>the procedures at Week 52 or the corresponding visit. All<br>study data will be analysed and reported for the Main Part<br>CSR. | The analysis will take place after the last subject completes the procedures at Week <b>52 58</b> or the corresponding visit. All study data will be analysed and reported for <b>the Main Part</b> CSR. | |
| | • Extension Part CSR: | • Extension Part CSR: | |
| | A separate SAP for analyses of 2-year extension period will be prepared describing the methodology and presentation of results. The analysis will take place after the last subject completes the procedures of 2-year extension period. | A separate SAP for analyses of 2 year extension period will be prepared describing the methodology and presentation of results. The analysis will take place after the last subject completes the procedures of 2 year extension period. | |

| 9.2. Analysis<br>Sets | The following sets will be used for the analyses performed in the study: | The following sets will be used for the analyses performed in the study: | To update study design/process in order to minimize |
|---|---|---|---|
| | • () | • () | the risk of COVID-<br>19 pandemic |
| | • Safety Set for the Main Part (SAF1) consists of all subjects who receive at least one IP during the randomised treatment period. Subjects will be analysed according to the treatment received. | • Safety Set for the Main Part (SAF1) consists of all subjects who receive at least one IP during the randomised treatment study period. Subjects will be analysed according to the treatment received. | |
| | • Safety Set for the Extension Part (SAF2) consists of all subjects who receive at least one IP during the extension period. | <ul> <li>Safety Set for the Extension Part (SAF2) consists of all<br/>subjects who receive at least one IP during the extension<br/>period.</li> </ul> | |
| | • PK Analysis Set (PKS) consists of all subjects in the SAF1 who have at least one PK sample analysed. | • PK Analysis Set (PKS) consists of all subjects in the SAF1 who have at least one PK sample analysed. | |
| | PD Analysis Set (PDS) consists of all subjects in the SAF1 who have at least one PD sample analysed. | • PD Analysis Set (PDS) consists of all subjects in the SAF1 who have at least one PD sample analysed. | |
| 9.5.1.<br>Efficacy<br>Variable<br>Analyses | As a secondary efficacy endpoint, number of units of pRBCs transfused during the Main Part will be analysed using Wilcoxon rank-sum test for each period. And mean LDH profile during the Main Part will be presented over time. | As a secondary efficacy endpoint, number of units of pRBCs transfused during the Main Part will be summarised descriptively by treatment sequence and treatment sequence within period and will be analysed using Wilcoxon rank-sum test for each period. And mean LDH profile during the Main Part will be presented over time. | To update study design/process in order to minimize the risk of COVID-19 pandemic To clarify the efficacy/safety analysis |
| 9.5.2. Safety<br>Analyses | 9.5.2. Safety Analyses for the Main Part | 9.5.2. Safety Analyses for the Main Part | To update study design/process in |
| 7 11141 3003 | () | () | order to minimize<br>the risk of COVID- |
| | All TEAEs and SAEs reported during the randomised treatment | All TEAEs and SAEs reported during the randomised | and link of CO (ID |

| | period will be summarised respectively by count and percentage | treatment period will be summarised respectively by count and | 19 pandemic |
|---|---|---|---|
| | of subjects experiencing events by system organ class, preferred | percentage of subjects experiencing events by system organ | ry punaenne |
| | term, treatment sequence, and period. SAEs leading to IP | class, preferred term <del>, treatment sequence, and period</del> . SAEs | To clarify the |
| | discontinuation and TEAEs by causality and severity will be | <b>TEAEs</b> leading to IP discontinuation and TEAEs by causality | efficacy/safety |
| | summarised similarly. All AEs including those pre-existing | and severity will be summarised similarly. All AEs including | analysis |
| | before the initiation of study drug will be listed by subject. | those pre-existing before the initiation of study drug will be listed | - |
| | before the initiation of study drug will be listed by subject. | by subject. | |
| | In addition, infection-related AEs including meningococcal | by subject. | |
| | infection and other systemic infection, and IRRs reported during | In addition, infection-related AEs including meningococcal | |
| | the randomised treatment period will also be summarised. | infection and other systemic infection, and IRRs reported | |
| | | during the randomised treatment period will also be | |
| | Duration of exposure to IP and number of IV infusion during the | summarised. | |
| | randomised treatment period will be summarised by treatment | | |
| | sequence and period with descriptive statistics for the SAF1. | Duration of exposure to IP and number of IV infusion during the | |
| | Prior and concomitant medications, and significant non-drug | randomised treatment period will be summarised by treatment | |
| | therapies will be summarised by treatment sequence and period | sequence and within period with descriptive statistics for the | |
| | with count and percentage. | SAF4. Prior and concomitant medications, and significant non- | |
| | Changes in vital signs and clinical laboratory parameters will be | drug therapies will be summarised by treatment sequence and | |
| | summarised descriptively by treatment sequence, period, and | period with count and percentage. | |
| | time point. Other safety variables will be summarised unless | Changes in vital signs and clinical laboratory parameters will be | |
| | otherwise specified, and all safety variables will be listed. | summarised descriptively by treatment sequence, period, and | |
| | otherwise specified, and an safety variables will be fisted. | time point visit. Other safety variables will be summarised | |
| | All safety analyses will be performed using the SAF1. | unless otherwise specified, and all safety variables will be listed. | |
| | | aniess otherwise specified, and an safety variables will be listed. | |
| | | All safety analyses will be performed using the SAF1. | |
| 9.5.3. Safety | 9.5.3. Safety Analyses for the Extension Part | 9.5.3. Safety Analyses for the Extension Part | To update study |
| Analyses for | All nomented towns for CAEs will be soled voice MJDD A.® | All reported terms for CAEs will be soded using MadDDA® | design/process in |
| the | All reported terms for SAEs will be coded using MedDRA®. | All reported terms for SAEs will be coded using MedDRA®. | order to minimize |
| Extension | SAEs reported during the Extension Part will be summarised and listed for the SAF2. | SAEs reported during the Extension Part will be summarised and listed for the SAF2. | the risk of COVID- |
| Part | ilsted for the SAF2. | and nated for the SAF 2. | 19 pandemic |
| | Duration of exposure to IP and number of IV infusion during | Duration of exposure to IP and number of IV infusion | |
| | the Extension Part will be summarised with descriptive statistics | during the Extension Part will be summarised with | |
| | for the SAF2. | descriptive statistics for the SAF2. | |

| 9.5.4.<br>Immunogeni<br>-city<br>Analyses | ADA and NAb results (e.g., 'positive' or 'negative') will be summarised with count and percentage by treatment sequence, period, and time point. In addition, incidence of overall ADA will be summarised by treatment sequence and period. Immunogenicity analyses will be performed using the SAF1. | ADA and NAb results (e.g., 'positive' or 'negative') will be summarised with count and percentage by treatment sequence, period, and time point visit. In addition, incidence of overall ADA will be summarised by treatment sequence and period. Immunogenicity analyses will be performed using the SAF1. | To clarify the efficacy/safety analysis |
|---|---|---|---|
| 9.5.5.<br>Pharmacody<br>-namic<br>Analyses | PD analysis will be performed for the PDS. The absolute values, and change from baseline in terminal complement activities will be summarised by treatment sequence, period, and time point. | PD analysis will be performed for the PDS. The absolute values, and change from baseline in terminal complement activities will be summarised by treatment sequence, period, and time point visit. () | To clarify the efficacy/safety analysis |
| 10.2<br>Monitoring | () Monitors will also perform source data verification by comparing entries in the eCRF with corresponding source data and informing the Investigator of any errors or omissions for the Main Part and IP infusion date/time at Week 52. () () | () Monitors will also perform source data verification by comparing entries in the eCRF with corresponding source data and informing the Investigator of any errors or omissions for the Main Part and IP infusion date/time at Week 52. () () | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| Database Management and Coding | <ul><li>() The eCRF will be used only during the Main Part and IP infusion date/time at Week 52.</li><li>()</li></ul> | () The eCRF will be used only during the Main Part and IP infusion date/time at Week 52. () | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |
| 10.7.<br>Protocol<br>Deviation | PDs will be reviewed and confirmed prior to database lock for the Main Part to decide which subjects and/or subject data will be excluded from certain analyses. Decisions regarding the exclusion of subjects and/or subject data from analyses will be documented and approved prior to database lock for the Main Part. | PDs will be reviewed and confirmed prior to database lock for the Main Part to decide which subjects and/or subject data will be excluded from certain analyses. Decisions regarding the exclusion of subjects and/or subject data from analyses will be documented and approved prior to database lock for the Main Part. | To update study<br>design/process in<br>order to minimize<br>the risk of COVID-<br>19 pandemic |

| 12 E / 1 1 | N/A | 1117 | T 1 1 |
|---|---|---|---|
| 13. Extended | N/A After completion of activities at Week 52, an open supplies that the supplies a supp | | To update study |
| Supply | extended supply of SB12 will be provided for up to 2 | | design/process in |
| | years starting from Week 52 to subjects who have I | , | order to minimize |
| | from study treatment and opt to participate in | LAICHUCU | the risk of COVID- |
| | supply under an ethical basis. | 1 | 19 pandemic |
| | Before entering an extended supply, the Investig | | |
| | review the subject status including reduction of PNI | | |
| | activity, such as improvement of symptoms or la | | |
| | parameters, during eculizumab treatment to decide | | |
| | subject will benefit from participation in extended | | |
| | Once subjects are considered to benefit from | | |
| | supply, subjects will be asked if he/she would like to | o receive | |
| | an extended supply. For receiving an extended | supply, | |
| | subjects should agree with signing ICF for extende | d supply | |
| | and with required activities including refraining | ng from | |
| | pregnancy, maintaining a highly effective contr | aceptive | |
| | method, and receiving meningococcal vaccina | tion (if | |
| | required by local regulations) to ensure subject | ` | |
| | during extended supply. | • | |
| | During extended supply, Investigators will treat subj | | |
| | 900 mg of SB12 every $14 \pm 2$ days for up to 2 years | ears (104 | |
| | weeks). SB12 will be packaged and labelled using of | oen label | |
| | and dispensed through the IWRS. Investigators | should | |
| | ensure the compliance and accountability of SB12 do | iring the | |
| | course of extended supply. Any PC must be rep | orted to | |
| | Sponsor. | | |
| | SAEs that occur during this phase must be reported | | |
| | Sponsor, which will be reported to regulatory author | | |
| | the Sponsor according to local/national requirem | ents via | |
| | expedited reporting and periodic reporting | such as | |
| | Development Safety Update Report (DSUR) or | Periodic | |

Safety Update Report (PSUR). Pregnancy should also be reported until 5 months after the last SB12 treatment. Other particular activities will not be imposed and no data collection or reporting will occur for extended supply.

Discontinuation of study treatment can be decided if unacceptable toxicity, pregnancy, other complement inhibitor use or lack of efficacy occurs, or at the discretion of the Investigator or by subject's consent withdrawal. Specific study procedures are not required for subjects who have discontinued prematurely except for SAEs reporting and pregnancy reporting.

During the period of extended supply, the Investigator and the Sponsor will follow all local laws and regulations relating to contact with and approvals from the IRB/IEC. The Investigator is responsible for ensuring that the study is conducted according to the signed Investigator statement, the study protocol and applicable regulations; for protecting the rights, safety, and welfare of subjects under the Investigator's care; and for the control of drugs under investigation.

The Investigators must maintain essential study documents until at least 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or at least 2 years after the formal discontinuation of clinical development of the IP or 15 years from completion of the extended supply, if applicable.

Investigational sites participation may be discontinued if the Sponsor, Investigator or IRB/IEC consider necessary. Extended supply may be terminated by the Sponsor if medically or ethically indicated, and in such cases will be

| | | promptly notified to the Investigator. In any case, health authorities and IRB/IEC will be informed for the action in accordance with applicable regulations | |
|---|---|---|---|
| 14. | [10] Soliris® EPAR – Product Information. EMA (Sep 04, | [10] Soliris® EPAR – Product Information. EMA (Sep 04, 2019) | To refer the latest |
| References | 2019). Retrieved Sep 09, 2019 from | Jul 01, 2020). Retrieved <del>Sep 09, 2019</del> Jul 13, 2020 from | version of |
| | https://www.ema.europa.eu/documents/product- | https://www.ema.europa.eu/documents/product- | regulatory |
| | information/soliris-epar-product-information_en.pdf | information/soliris-epar-product-information_en.pdf | document |

Amendment 5: Version 6.0, Nov 27, 2020

| Section<br>Affected | Original Content | Amended/New Content | Rationale |
|---|---|---|---|
| SYNOPSIS<br>Study<br>Design | This is a randomised, Phase III, double-blind, multicentre, cross-over study to compare the efficacy, safety, pharmacokinetics, and immunogenicity between SB12 and Soliris® in subjects with PNH. | This is a randomised, Phase III, double-blind, multicentre, cross-over study to compare the efficacy, safety, pharmacokinetics, and immunogenicity between SB12 and Soliris® in subjects with PNH. | To update study<br>design/process in<br>order to address a<br>special<br>circumstances of a |
| | Subjects will be randomised in a 1:1 ratio to treatment sequence I (SB12 to Soliris®) or treatment sequence II (Soliris® to SB12). Subjects who are randomised to initially receive SB12 will be switched to receive Soliris® and subjects who are randomised to initially receive Soliris® will be switched to receive SB12 at Week 26. | Subjects will be randomised in a 1:1 ratio to treatment sequence I (SB12 to Soliris®) or treatment sequence II (Soliris® to SB12). Subjects who are randomised to initially receive SB12 will be switched to receive Soliris® and subjects who are randomised to initially receive Soliris® will be switched to receive SB12 at Week 26. | shortage of the comparator |
| | After completion of activities at Week 52, an open-label extended supply of SB12 will be provided for up to 2 calendar years to subjects who have benefited from study treatment and opt to participate in extended supply under an ethical basis. | In special circumstances of a shortage of the comparator, to ensure continuity of study treatment for the duration of study, the Sponsor will provide SB12 instead of Soliris® in a blinded manner. | |
| | | After completion of activities at Week 52, an open-label extended supply of SB12 will be provided for up to 2 calendar years to subjects who have benefited from study treatment and opt to participate in extended supply under an ethical basis. | |
| SYNOPSIS<br>Statistical<br>Methods | Analysis sets for efficacy analyses Modified Full Analysis Set (M-FAS) consists of all randomised subjects who do not have positive result of pharmacogenetic analysis (C5 gene polymorphism). However, subjects who do not have any efficacy assessment result after randomisation and do not receive IP during the study period will be excluded from this analysis set. Following the intent-to-treat principle, subjects | Analysis sets for efficacy analyses Modified Full Analysis Set (M-FAS) consists of all randomised subjects who do not have positive result of pharmacogenetic analysis (C5 gene polymorphism). However, subjects who do not have any efficacy assessment result after randomisation and do not receive IP during the study period will be excluded from this analysis set. Following the intent-to-treat principle, subjects | To update study<br>design/process in<br>order to address a<br>special<br>circumstances of a<br>shortage of the<br>comparator |

will be analysed according to the treatment sequence they are assigned to at randomisation.

Per-Protocol Set for AUEC of LDH (PPS-AUEC) consists of all M-FAS subjects who have sufficient LDH assessments for AUEC calculation without any major protocol deviations (PDs) that have impact on efficacy assessment. Subjects excluded from the primary analysis will be pre-defined on a case-by-case basis prior to unblinding the treatment sequence assignment for analyses.

Per-Protocol Set for LDH at a single time point (PPS-single) consists of all M-FAS subjects who have LDH assessment at Week 26 without any major PDs that have impact on efficacy assessment. Subjects excluded from the primary analysis will be pre-defined on a case-by-case basis prior to unblinding the treatment sequence assignment for analyses.

(...)

## Safety analyses

Safety analyses will be performed in the Safety Set (SAF).

All reported terms for AEs will be coded using Medical Dictionary for Regulatory Activities (MedDRA®). AEs will be collected and classified according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0.

All AE data will be summarised by count and percentage of subjects experiencing events by system organ class, preferred term. TEAEs leading to IP discontinuation and treatment-emergent AEs (TEAEs) by causality and severity will be summarised similarly. Infection-related AEs including

will be analysed according to the treatment sequence they are assigned to at randomisation.

Per-Protocol Set for AUEC of LDH (PPS-AUEC) consists of all M-FAS subjects who have sufficient LDH assessments for AUEC calculation without any major protocol deviations (PDs) that have impact on efficacy assessment. Subjects excluded from the primary analysis will be pre-defined on a case-by-case basis prior to unblinding the treatment sequence assignment for analyses. In addition, subjects who received different treatment from the randomised treatment sequence due to a shortage of the comparator will be excluded from this analysis set.

Per-Protocol Set for LDH at a single time point (PPS-single) consists of all M-FAS subjects who have LDH assessment at Week 26 without any major PDs that have impact on efficacy assessment. Subjects excluded from the primary analysis will be pre-defined on a case-by-case basis prior to unblinding the treatment sequence assignment for analyses. In addition, subjects who received different treatment in Period 1 from the randomised treatment sequence due to a shortage of the comparator will be excluded from this analysis set.

 $(\ldots)$ 

## Safety analyses

Safety analyses will be performed in the Safety Set (SAF).

All reported terms for AEs will be coded using Medical Dictionary for Regulatory Activities (MedDRA®). AEs will be collected and classified according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0.

| | meningococcal infection and other systemic infection, and IRRs will also be summarised. Changes in vital signs and clinical laboratory parameters will be summarised descriptively by treatment sequence and visit. Other safety variables will be summarised unless otherwise specified. | All AE data will be summarised by count and percentage of subjects experiencing events by system organ class, preferred term. TEAEs leading to IP discontinuation and treatment-emergent AEs (TEAEs) by causality and severity will be summarised similarly. Infection-related AEs including meningococcal infection and other systemic infection, and IRRs will also be summarised. Changes in vital signs and clinical laboratory parameters will be summarised descriptively by treatment sequence and visit. Other safety variables will be summarised unless otherwise specified. Additional analyses will be performed for the subjects who received different treatment from the randomised treatment sequence due to a shortage of the comparator if needed. For example, AEs and concomitant medications will be analysed based on the actual switched treatment. | |
|---|---|---|---|
| Figure 1 | Sequence (n-25) Soliris | Sequence (n-25) <sup>b</sup> SB12 Soliris <sup>2</sup> | To update study design/process in order to address a special circumstances of a shortage of the comparator |
| Figure 1<br>Footnote | N/A | During the treatment period, in special circumstances of a shortage of the comparator, to ensure continuity of study treatment for the duration of study, the Sponsor will provide SB12 instead of Soliris® in a blinded manner. | To update study design/process in order to address a special circumstances of a shortage of the comparator |

| LIST OF<br>STUDY<br>STAFF | Clinical Project Manager | Clinical Project Manager | Administrative change |
|---|---|---|---|
| | Clinical Development Lead Clinical Research Physician Clinical Research Scientist | Clinical Development Lead Clinical Research Physician Clinical Research Scientist | |
| 1.5.1.<br>Known<br>Potential<br>Risks | Considering the mechanism of action of eculizumab, () All subjects will be monitored for early signs of meningococcal infection, evaluated immediately if infection is suspected, and treated with appropriate antibiotics if necessary. In order to ensure the safety of subjects who participate in the study, () | Considering the mechanism of action of eculizumab, () All subjects will be monitored for early signs of meningococcal infection, evaluated immediately if infection is suspected, and treated with appropriate antibiotics if necessary. According to the study design, the switch of IP (cross-over) occurs during the study. The potential negative impact from this IP switch is considered to be minimal given similarity and comparability of SB12 to Soliris® and low antibody responses in Soliris® (3.4%) similar to that of placebo (4.8%) in placebo controlled studies in subjects with PNH [10]. In order to ensure the safety of subjects who participate in the study, () | To update risk assessment in order to address a special circumstances of a shortage of the comparator |

| 3.1.<br>Overview of<br>Study<br>Design | This is a randomised, Phase III, double-blind, multicentre, crossover study to compare the efficacy, safety, pharmacokinetics, and immunogenicity between SB12 and Soliris® in subjects with PNH. Subjects will be randomised in a 1:1 ratio to treatment sequence I (SB12 to Soliris®) or treatment sequence II (Soliris® to SB12). Subjects randomly assigned to treatment with SB12 or Soliris® will receive 600 mg of eculizumab IV every week for first 4 weeks (initial phase) and 900 mg for the fifth week, followed by 900 mg every 2 weeks thereafter. Subjects who are randomised to initially receive SB12 will be switched to receive Soliris® and subjects who are randomised to initially receive SB12 at Week 26. SB12 or Soliris® will be given until Week 50. | This is a randomised, Phase III, double-blind, multicentre, crossover study to compare the efficacy, safety, pharmacokinetics, and immunogenicity between SB12 and Soliris® in subjects with PNH. Subjects will be randomised in a 1:1 ratio to treatment sequence I (SB12 to Soliris®) or treatment sequence II (Soliris® to SB12). Subjects randomly assigned to treatment with SB12 or Soliris® will receive 600 mg of eculizumab IV every week for first 4 weeks (initial phase) and 900 mg for the fifth week, followed by 900 mg every 2 weeks thereafter. Subjects who are randomised to initially receive SB12 will be switched to receive Soliris® and subjects who are randomised to initially receive SB12 at Week 26. SB12 or Soliris® will be switched to receive SB12 at Week 26. SB12 or Soliris® will be given until Week 50. However, in special circumtances of a shortage of the comparator, to ensure continuity of study treatment for the duration of study, the Sponsor will provide SB12 instead of Soliris® in a blinded manner. | To update study design/process in order to address a special circumstances of a shortage of the comparator |
|---|---|---|---|
| 5.1.1. Dosing and Treatment Schedule | () The subject receiving SB12 or Soliris® therapy may require dosing interval adjustment within the recommended 14 ± 2 days dosing schedule during the maintenance period (up to every 12 days) when it is deemed necessary at the discretion of the Investigator; e.g., two consecutive events of elevated LDH ≥ 2 × ULN combined with sign or symptom of intravascular haemolysis after prior LDH reduction to < 1.5 × ULN on treatment. If a 12 or 13 day dosing interval conflicts with administrative schedules (e.g., holidays or weekends) but a shortened dosing interval is considered necessary for safety of subject, consultation with medical monitor (or Sponsor) is recommended. For subjects whose dosing interval is adjusted to 12 days in Period 1, it is recommended that the dosing interval be | () The subject receiving SB12 or Soliris® therapy may require dosing interval adjustment within the recommended 14 ± 2 days dosing schedule during the maintenance period (up to every 12 days) when it is deemed necessary at the discretion of the Investigator; e.g., two consecutive events of elevated LDH ≥ 2 × ULN combined with sign or symptom of intravascular haemolysis after prior LDH reduction to < 1.5 × ULN on treatment. If a 12 or 13 day dosing interval conflicts with administrative schedules (e.g., holidays or weekends) but a shortened dosing interval is considered necessary for safety of subject, consultation with medical monitor (or Sponsor) is recommended. For subjects whose dosing interval is adjusted to 12 days in Period 1, it is recommended that the dosing interval be | To update study design/process in order to address a special circumstances of a shortage of the comparator |

| | switched back to 14 days after switching IP at Week 26. Once the above event has occurred, the Investigator should inform the medical monitor and/or Sponsor immediately. | switched back to 14 days after switching IP at Week 26. Once the above event has occurred, the Investigator should inform the medical monitor and/or Sponsor immediately. In special circumstances of a shortage of the comparator, to ensure continuity of study treatment for the duration of study, the Sponsor will provide SB12 instead of Soliris® in a blinded manner. Rules for allocation of remaining comparators during the comparator shortage situation will | |
|---|---|---|---|
| | | be prespecified prior to execution of the potential change of IP assignment from Soliris® to SB12 in a blinded manner. This is to avoid the risk of unblinding and potential bias. | |
| 7.1.3.<br>Treatment<br>Period | The Investigator will evaluate the assessment results and manage subjects based on the medicinal judgement and/or knowledge. | The Investigator will evaluate the assessment results and manage subjects based on the medicinal judgement and/or knowledge. In special circumstances of a shortage of the comparator, to ensure continuity of study treatment for the duration of study, the Sponsor will provide SB12 instead of Soliris® in a blinded manner. Investigators and subjects will be informed prior to the execution of the potential change of IP assignment. Subjects willing to continue the study treatment after knowing that they may receive SB12 instead of Soliris® in a blinded manner during the study, should have their agreement both documented in the source document and an ICF. If the Investigators or subjects do not agree to the potential change of IP assignment, then subjects may withdraw from the study and be closely monitored for at least 8 weeks after last dose of study drug. | To update study design/process in order to address a special circumstances of a shortage of the comparator |
| 8.3.3.<br>Infusion-<br>related<br>Reactions | Administration of SB12 or Soliris® may result in infusion reactions or immunogenicity that could cause allergic or hypersensitivity reactions (including anaphylaxis), though immune reactions within 48 hours of Soliris® administration did not differ from placebo arm in PNH, aHUS, refractory | Administration of SB12 or Soliris® may result in infusion reactions or immunogenicity that could cause allergic or hypersensitivity reactions (including anaphylaxis), though immune reactions within 48 hours of Soliris® administration did not differ from placebo arm in PNH, | To refer the latest<br>version of<br>regulatory<br>document |

Samsung Bioepis -  Information

| | gMG, NMOSD, and other studies conducted with Soliris <sup>®</sup> . In clinical trials no PNH, aHUS, refractory gMG, or NMOSD patients experienced an infusion reaction which required discontinuation of Soliris <sup>®</sup> . () | aHUS, refractory gMG, NMOSD, and other studies conducted with Soliris. In clinical trials, 1 (0.9%) gMG patient experienced an infusion reaction which required discontinuation of Soliris. The PNH, aHUS, refractory gMG, or NMOSD patients experienced an infusion reaction which required discontinuation of Soliris in clinical trials. | |
|---|---|---|---|
| 9.2. Analysis<br>Sets | <ul> <li>The following sets will be used for the analyses performed in the study:</li> <li>()</li> <li>Per-Protocol Set for AUEC of LDH (PPS-AUEC) consists of all M-FAS subjects who have sufficient LDH assessments for AUEC calculation without any major PDs that have impact on efficacy assessment. Subjects excluded from the primary analysis will be pre-defined on a case-by-case basis prior to unblinding the treatment sequence assignment for analyses.</li> <li>Per-Protocol Set for LDH at a single time point (PPS-single) consists of all M-FAS subjects who have LDH assessment at Week 26 without any major PDs that have impact on efficacy assessment. Subjects excluded from the primary analysis will be pre-defined on a case-by-case basis prior to unblinding the treatment sequence assignment for analyses.</li> <li>()</li> </ul> | <ul> <li>The following sets will be used for the analyses performed in the study:</li> <li>()</li> <li>Per-Protocol Set for AUEC of LDH (PPS-AUEC) consists of all M-FAS subjects who have sufficient LDH assessments for AUEC calculation without any major PDs that have impact on efficacy assessment. Subjects excluded from the primary analysis will be pre-defined on a case-by-case basis prior to unblinding the treatment sequence assignment for analyses. In addition, subjects who received different treatment from the randomised treatment sequence due to a shortage of the comparator will be excluded from this analysis set.</li> <li>Per-Protocol Set for LDH at a single time point (PPS-single) consists of all M-FAS subjects who have LDH assessment at Week 26 without any major PDs that have impact on efficacy assessment. Subjects excluded from the primary analysis will be pre-defined on a case-by-case basis prior to unblinding the treatment sequence assignment for analyses. In addition, subjects who received different treatment in Period 1 from the randomised treatment sequence due to a shortage of the comparator will be excluded from</li> </ul> | To update study design/process in order to address a special circumstances of a shortage of the comparator |

| | | this analysis set. | |
|---|---|---|---|
| | | () | |
| 9.5.2. Safety<br>Analyses | () | () | To update study design/process in |
| | All safety analyses will be performed using the SAF. | All safety analyses will be performed using the SAF. Additional analyses will be performed for the subjects who received different treatment from the randomised treatment sequence due to a shortage of the comparator if needed. For example, AEs and concomitant medications will be analysed based on the actual switched treatment. | order to address a<br>special<br>circumstances of a<br>shortage of the<br>comparator |
| 14.<br>References | [21] Soliris® Prescribing Information. FDA (Jun 27, 2019). Retrieved Jul 09, 2019 from <a href="https://www.accessdata.fda.gov/drugsatfda_docs/label/2019/125">https://www.accessdata.fda.gov/drugsatfda_docs/label/2019/125</a> <a href="https://www.accessdata.fda.gov/drugsatfda_docs/label/2019/125">https://www.accessdata.fda.gov/drugsatfda_docs/label/2019/<a href="https://www.accessdata.fda.gov/drugsatfda_docs/label/2019/125">https://www.accessdata.fda.gov/drugsatfda_docs/label/2019/125</a> <a href="https://www.accessdata.fda.gov/drugsatfda_docs/label/2019/125">https://www.accessdata.fda.gov/drugsatfda_docs/label/2019/125</a> <a href="https://www.accessdata.fda.gov/drugsatfda_docs/label/2019/125">https://www.accessdata.fda.gov/drugsatfda_docs/label/2019/125</a> <a 125166s434lbl.pdf"="" 2020="" drugsatfda_docs="" href="https://www.accessdata.fda&lt;/td&gt;&lt;td&gt;[21] Soliris® Prescribing Information. FDA (Jun 27, 2019 Nov 20, 2020). Retrieved Jul 09, 2019 Nov 26, 2020 from &lt;a href=" https:="" label="" www.accessdata.fda.gov="">https://www.accessdata.fda.gov/drugsatfda_docs/label/2020/125166s434lbl.pdf</a></a> | To refer the latest<br>version of<br>regulatory<br>document | |